

## STATISTICAL ANALYSIS PLAN

A single centre, open label, pilot phase Ib study to investigate blood stage malaria infection after Direct Venous Inoculation of cryopreserved Plasmodium falciparum (NF54 strain) Sporozoites (PfSPZ-DVI) in malaria naïve healthy adult volunteers

**Protocol:** MMV\_PfSPZ-DVI Blood Stage\_19\_01

**SGS LS number:** BE-80-1914715

Development phase: Ib

**Sponsor:** Medicines for Malaria Venture (MMV)

**SAP version number:** Final 1.0

**SAP version date:** 11FEB2021



## **SIGNATURE PAGE**

| Name and function | Date<br>(ddMMMyyyy) | Signature |
|---|---|---|
| SGS LS author(s) and rev | viewer(s): | |
| Daniel Izquierdo<br>Juncàs, Biostatistician | 11FEB2021 | DocuSigned by: Daniel Izquierdo Juncas Signer Name: Daniel Izquierdo Juncas Signing Reason: I am the author of this document Signing Time: 11-Feb-2021 16:11 CET 690E658303D54613A9EC59ED7BAE2148 |
| Bastiaan Jansen,<br>Biostatistical<br>Coordinator | 11FEB2021 | DocuSigned by: bastiaan Jansen Signer Name: bastiaan Jansen Signing Reason: I approve this document Signing Time: 11-Feb-2021 16:22 CET 15ADFC6D3E734686B167F978EA41202B |
| Sponsor's approval: | | |
| The approver agrees the statistical analysis plan. | statistical analysis w | ill be performed according to this |
| Farouk Chughlay, Project and Medical Director | | DocuSigned by: Signer Name: Farouk Chughlay Signing Reason: I approve this document Signing Time: 11-Feb-2021 07:54 PST 6A2C1E232AEB48DFA6A544CF570BF27F |
| Myriam El Gaaloul<br>Director, Clinical<br>Sciences | | DocuSigned by: Myriam El Gaaloul Signer Name: Myriam El Gaaloul Signing Reason: I approve this document Signing Time: 13-Feb-2021 01:24 PST C2CA71F33AA843DAB327CC3B36DFB37C |



## PROTOCOL HISTORY

| Protocol: | | |
|---|---|---|
| Version or ID | Date (ddMMMyyyy) | Impact of the changes on the statistical analysis |
| Final 1.0 | 17DEC2019 | NAP |
| Final 2.0 | 27JAN2020 | Including substantial amendment 1: no impact on the statistical analysis. |
| Final 3.0 | 24JUN2020 | Including substantial amendment 2: no impact on the statistical analysis. |

This statistical analysis plan (SAP) only considers the last version of the protocol, and of the protocol amendments, as listed above.



## LIST OF ABBREVIATIONS

ADaM analysis data model

AE adverse event

ALP alkaline phosphatase
ALT alanine transaminase

aPTT activated partial thromboplastin time

AST aspartate transaminase

β-HCG β-human chorionic gonadotropin

BMI body mass index
bpm beats per minute
CI confidence interval
CMV cytomegalovirus
CRF case report form
CRP C-reactive protein

DBP diastolic blood pressure
DVI direct venous inoculation

DY relative day

EBV Epstein Barr Virus ECG electrocardiogram

eGFR estimated glomerular filtration rate

EOS end of study

FSH follicle stimulating hormone
GGT gamma-glutamyl transferase
HbsAg hepatitis B surface antigen

HCV hepatitis C virus

HIV human immunodeficiency virus

HR heart rate

ICF informed consent form

ICH International Council for Harmonisation

IgM immunoglobulin M

INR international normalised ratio

LDH lactate dehydrogenase

log10PRR48 log10 parasite reduction ratio per 48 h



log10PRR48,max maximum log10 parasite reduction ratio per 48 h

MCH mean corpuscular haemoglobin

MCHC mean corpuscular haemoglobin concentration

MCV mean corpuscular volume

MedDRA Medical Dictionary for Regulatory Activities

NAP not applicable

NCE new chemical entities

PC50 parasite clearance half-life

PC99 predicted time to reach parasite clearance of 99%

PCR polymerase chain reaction

PD pharmacodynamic

PfSPZ P. falciparum sporozoites

PfSPZ-DVI inoculation of P. falciparum sporozoites through direct venous

Challenge inoculation

PMR parasite multiplication rate

PMR48 parasite multiplication rate standardised to 48 h

PMRLC parasite multiplication rate per life cycle (if not 48 h)

PRR parasite reduction ratio

PT prothrombin time

QTc corrected QT interval

QTcB Bazett's corrected QT interval
QTcF Fridericia's corrected QT interval

RBC red blood cell

rRT-PCR real-time reverse transcription polymerase chain reaction

SAP statistical analysis plan

SAF safety analysis set

SARS-CoV-2 severe acute respiratory syndrome coronavirus 2

SBP systolic blood pressure

SCR all screened subject's analysis set

SD standard deviation

SE standard error

SGS LS SGS Life Sciences

SOP standard operating procedure

STAT statistics



TLF tables, listings and figures

ULN upper limit of normal

varATS the acidic terminal segment in Plasmodium falciparum var

genes

VIS volunteer infection study

VS vital signs

WBC white blood cell

WHO World Health Organisation

WI work instruction



## **DEFINITION OF TERMS**

baseline An initial measurement of a condition that is taken at an early time

point and used for comparison over time to look for changes. The

study specific definition is in section 5.2.2.

case report form (CRF)

A printed, optical, or electronic document designed to record protocol required information to be reported to the sponsor for each

trial subject.

display Analysis table, figure or listing

phase Interval of time in the planned conduct of a study associated with a

specific purpose: for example, screening, treatment, follow-up.

round half up tiebreaking rule Convention to round values ending with 5 to positive infinity. The round half up rule is implemented in the SAS® ROUND function.

Examples:

| <b>Database value</b> | Rounded value |
|-----------------------|---------------|
| -1.35 | -1.3 |
| -1.25 | -1.2 |
| 1.25 | 1.3 |
| 1.35 | 1.4 |

significant digit All digits of a number used to express it to the required degree of accuracy, starting from the first non-zero digit.

postbaselineemergent abnormality Any post-baseline abnormality that was not present at baseline (e.g. haemoglobin normal at baseline and grade 1 post-baseline; glucose low at baseline and high post-baseline.

MMV\_PfSPZ-DVI Blood Stage\_19\_01

Final 1.0 of 11FEB2021

## TABLE OF CONTENTS

| _ | | 2 |
|---|---|---|
| | • | <i>7</i> 3 |
| | | tions4 |
| | | ms |
| Tab | | ts8<br>on11 |
| 1.1 | • | bjectives |
| 1.2<br>1.3 | • | esign |
| | • | ed sample size |
| 1.4 | | nisation and blinding |
| 1.5 | | analysis |
| 1.6 | | re |
| 1.7 | | on model |
| 2. | | lynamic analyses14 |
| 2.1 | | codynamics |
| | 2.1.1 | Available data14 |
| | 2.1.2 | Endpoints and derivation rules |
| | 2.1.3 | Inferential statistics |
| | 2.1.3.1 | Secondary endpoints: |
| | 2.1.3.2 | Exploratory endpoints: |
| | 2.1.4 | Presentation of results |
| 3. | - | yses20 |
| 3.1 | Adverse | e events |
| | 3.1.1 | Available data |
| | 3.1.2 | Derivation rules |
| | 3.1.3 | Presentation of results |
| 3.2 | Clinical | laboratory evaluation |
| | 3.2.1 | 3.2.1 Available data |
| | 3.2.2 | 3.2.2 Derivation rules |
| | 3.2.3 | 3.2.3 Presentation of results |
| 3.3 | .3 Vital signs22 | |
| | 3.3.1 | Available data24 |
| | 3.3.2 | Derivation rules |
| | 3.3.3 | 3.3.3 Presentation of results |



## Statistical Analysis Plan

MMV\_PfSPZ-DVI Blood Stage\_19\_01

Final 1.0 of 11FEB2021

| 3.4 | Electro | cardiograms | 25 |
|-----|------------|--------------------------------------------|----|
| | 3.4.1 | Available data | 25 |
| | 3.4.2 | Derivation rules | 25 |
| | 3.4.3 | Presentation of results | 25 |
| 3.5 | Malaria | a clinical score | 26 |
| | 3.5.1 | Available data | 26 |
| | 3.5.2 | Derivation rules | 26 |
| | 3.5.3 | Presentation of results | 26 |
| 3.6 | Physica | al examinations | 27 |
| 4. | General ch | haracteristics analyses | 28 |
| 4.1 | Subject | t disposition | 28 |
| 4.2 | Protoco | ol deviations and eligibility | 28 |
| 4.3 | Demog | graphic and other baseline characteristics | 28 |
| | 4.3.1 | Available data | 28 |
| | 4.3.2 | Derivation rules | 29 |
| | 4.3.3 | Presentation of results | 29 |
| 4.4 | Medica | al history and concomitant diseases | 29 |
| | 4.4.1 | Available data | 29 |
| | 4.4.2 | Derivation rules | 29 |
| | 4.4.3 | Presentation of results | 30 |
| 4.5 | Prior a | nd concomitant therapies | 30 |
| | 4.5.1 | Available data | 30 |
| | 4.5.2 | Derivation rules | 30 |
| | 4.5.3 | Presentation of results | 30 |
| 4.6 | Exposu | re to challenge agent | 30 |
| | 4.6.1 | Available data | 30 |
| | 4.6.2 | Derivation rules | 31 |
| | 4.6.3 | Presentation of results | 31 |
| 5. | General m | nethodology | 32 |
| 5.1 | Analys | is sets | 32 |
| | 5.1.1 | Analysis sets | 32 |
| | 5.1.2 | As planned versus as actual analysis | 32 |
| 5.2 | Phases | and time points | 32 |
| | 5.2.1 | Phases | 32 |



## Statistical Analysis Plan

MMV\_PfSPZ-DVI Blood Stage\_19\_01

Final 1.0 of 11FEB2021

| | 5.2.2 | Baseline and change from baseline | 33 |
|---|---|---|---|
| | 5.2.3 | Relative day | 33 |
| | 5.2.4 | Analysis visits | 33 |
| | 5.2.5 | Worst-case | 34 |
| 5.3 | Imputat | ion and rounding rules | 34 |
| | 5.3.1 | Missing values | 34 |
| | 5.3.2 | Handling partially or completely missing dates in calculations. | 34 |
| | 5.3.3 | Values below or above a threshold | 34 |
| | 5.3.4 | Rounding of derived variables | 35 |
| | 5.3.5 | Outliers | 35 |
| 5.4 | Presenta | ation of results | 35 |
| | 5.4.1 | Calculation of descriptive statistics and percentages | 35 |
| | 5.4.2 | Presentation of treatments | 36 |
| | 5.4.3 | Ordering in tables, figures and listings | 36 |
| 6. | Changes to | the planned analysis | 37 |
| 6.1 | Change | s not covered by protocol amendments before database lock | 37 |
| 6.2 | Change | s not covered by protocol amendments after database lock | 37 |
| 6.3 | Change | s to the final statistical analysis plan | 37 |
| 7. | References | | 38 |
| 8. | List of tabl | es, listings and figures | 39 |
| 8.1 | Tables . | | 39 |
| 8.2 | Listings | 3 | 41 |
| 8.3 | Figures | | 42 |
| 9. | Appendice | s | 44 |
| 9.1 | SAS co | de | 44 |
| 9.2 | Schedu | le of assessments | 45 |



## 1. INTRODUCTION

This SAP describes the final statistical analysis to be performed for the MMV\_PfSPZ-DVI Blood Stage\_19\_01 (BE-80-1914715) study.

This SAP covers the pharmacodynamic (PD), safety, and general characteristics parts of the statistical analysis. It specifies the analysis displays to be presented and describes the methods and procedures in a more elaborated way than in the statistical methods section of the protocol. The parasite transcriptomics analysis is not in the scope of this SAP but will be described by the Institute of Tropical Medicine and reported separately.

The statistical analysis will process and present the results following the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) standards, in particular the ICH-E3, ICH-E6, and ICH-E9 guidelines.

## 1.1 STUDY OBJECTIVES

According to the protocol, the primary objectives of this study are:

- To evaluate the safety and tolerability associated with blood-stage malaria infection in naïve healthy participants after PfSPZ-DVI Challenge.
- To characterise key stages in the blood-stage parasite growth profile in malaria infection in naïve healthy participants after PfSPZ-DVI Challenge.

According to the protocol, the secondary objectives of this study are:

- To determine the safety and tolerability of Riamet® in blood-stage malaria infection in naïve healthy participants after PfSPZ-DVI Challenge.
- To characterise the blood-stage parasite profile in malaria infection in naïve healthy participants after PfSPZ-DVI Challenge before Riamet® administration.
- To characterise the blood-stage parasite clearance profile of Riamet® in malaria infection in naïve healthy participants after PfSPZ-DVI Challenge.

According to the protocol, the exploratory objective of this study is to characterise the individual variability of blood-stage parasite profile.

## 1.2 STUDY DESIGN

This is a single-centre, open-label, Phase Ib study designed to assess if intravenous bolus injection of approximately 3200 P. falciparum (NF54 strain) sporozoites can be safely administered to achieve blood-stage parasitaemia with a kinetics/PCR profile that will allow for the future characterisation of antimalarial blood-stage activity of NCEs in a relatively small number of participants during early drug development.

Up to 16 healthy, malaria-naïve males and females, aged 18-55 years, will be enrolled in a maximum of 2 cohorts (up to 8 participants per cohort; a participant may be enrolled in one cohort only). Enrolment into the cohorts will proceed sequentially, with two target levels of parasitaemia previously achieved in healthy participants enrolled in malaria VIS at other study sites, i.e., 5000 parasites/mL blood in Cohort 1 and 10000 parasites/mL blood in Cohort 2.



Each participant will be admitted to the clinical unit in the morning of Day -1 and inoculated with approximately 3200 P. falciparum sporozoites (NF54 strain) by DVI on Day 1. Participants will be discharged 2 h post inoculation on Day 1 and will be monitored daily via phone call from Day 2 until Day 6 to solicit any AEs. Participants will come to the clinical unit daily from Day 7 until Day 9 and together with the malaria clinical score, the presence of parasites will be assessed once daily by a specific qPCR targeting the varATS (the acidic terminal segment in Plasmodium falciparum var genes) multigenic family; this to accurately describe parasite growth even in case PCR positivity, i.e., a qPCR outcome ≥250 parasites per mL blood, is confirmed this early (very low probability and with low densities). Participants will be confined to the clinical unit from Day 10 in the morning. qPCR will be performed and malaria clinical score assessed twice daily and participants will be administered registered antimalarial therapy, i.e., Riamet®, when the following criteria are met:

- 1. Cohort 1: ≥5000 parasites/mL blood or earlier if a participant has a malaria clinical score >6 or at Investigator's discretion.
- 2. Cohort 2: ≥10000 parasites/mL blood or earlier if a participant has a malaria clinical score >6 or at Investigator's discretion.

The registered 3-day antimalarial therapy regimen will be further administered and monitored. qPCR assessments of parasitaemia will be carried out at multiple time points (2, 6, 8, 12, 16, 24, 36, 48 and 72 h) following initiation of Riamet® and malaria clinical score will be assessed twice daily during confinement in the clinical unit. Safety and tolerability will be monitored during the whole study duration, specific assessments will be done at periodic pre-specified time points from Day 10 and for at least 72 h after initiating antimalarial therapy, i.e., during confinement in the clinical unit. If an intolerance or contraindication to Riamet® develops, Malarone® will be administered.

Upon parasite clearance (defined as a qPCR value below the limit of quantification of 50 parasites per mL blood after initiating antimalarial therapy) and at least 72 h after initiating antimalarial therapy (estimated to occur on or before Day 19 and on or before Day 22 for Cohort 1 and Cohort 2, respectively), and if clinically well, participants will be discharged from the clinical unit and will be followed up for safety assessments, clinical evaluation and malaria qPCR in the clinical unit at the EOS visit on Day 28.

All participants inoculated with PfSPZ-DVI Challenge will commence antimalarial therapy no later than Day 24 for both cohorts, regardless if they reach pre-defined cohort-specific PCR parasitaemia/malaria clinical score thresholds. Participants who start antimalarial therapy on Day 24 will only be discharged from confinement at the end of the EOS visit on Day 28.

The schedule of assessments is in appendix 9.2.

After evaluation of data from Cohort 1, the Safety Review Team decided to continue with Cohort 2 (8 participants) using a threshold of 5000 parasites/mL.



#### 1.3 EXPECTED SAMPLE SIZE

Up to 16 participants will be enrolled in 2 cohorts of 8 participants per cohort. In agreement with the Sponsor, additional participants may be recruited in each cohort, to replace discontinuations for non-safety reasons and achieve the required cohort size.

This is an exploratory study focusing on the methodology of malaria inoculation in healthy participants, thus no formal sample size calculation is performed.

## 1.4 RANDOMISATION AND BLINDING

Participants are not randomised. As participants are confirmed to be eligible for the study, they will be assigned a single unique identifier across the study and will be enrolled sequentially in one of the two cohorts.

All participants will be inoculated with PfSPZ-DVI Challenge and receive registered antimalarial therapy, i.e. Riamet® (Malarone® if an intolerance or contraindication to Riamet® develops).

As this is an open-label study, blinding is not applicable.

## 1.5 Interim analysis

No interim analyses are foreseen.

#### 1.6 SOFTWARE

SAS version 9.4 or later will be used for programming.

Monolix for modelling parasite growth.

#### 1.7 VALIDATION MODEL

SGS Life Sciences (SGS LS) – Clinical Research statistics (STAT) standard operating procedures (SOPs) and work instructions (WIs) as effective at the project start will be followed throughout the project, provided the applicable regulatory requirements are still met.

ADaMs and TLFs related to the time to first PCR positivity and time to parasitaemia of ≥5000 parasites per mL blood will be validated according to model C. All other tables/figures/listings follow validation model B (see SOP.STAT.020):

- Model B: review by an independent person
- Model C: review by an independent person and independent programming of the parameters indicated in this SAP



## 2. PHARMACODYNAMIC ANALYSES

### 2.1 PHARMACODYNAMICS

### 2.1.1 Available data

Parasitaemia is assessed by qPCR at the time points indicated in appendix 9.2.

## 2.1.2 Endpoints and derivation rules

The following primary endpoint parameters will be derived:

- Time to first PCR positivity in days: (datetime in seconds of first positive parasitaemia datetime in seconds of inoculation) / (24\*60\*60)
  - Positive parasitaemia is defined as qPCR outcome (MBTESTCD = PARADENS) ≥ 250 asexual parasites per mL.
  - o Subjects with absence of positive parasitaemia will be excluded.
- Parasitaemia at first PCR positivity defined as qPCR outcome ≥ 250 asexual parasites per mL
- Time to parasitaemia of ≥5000 parasites per mL blood in days: (datetime in seconds of first parasitaemia of ≥5000 parasites per mL blood datetime in seconds of inoculation) / (24\*60\*60)
  - In the absence of parasitaemia of ≥5000 parasites per mL blood, the duration will be censored. The censoring datetime will be set to the datetime of first administration of antimalarial treatment. If the date of antimalarial treatment is (partially) missing the censored duration will be set to 28 days.
- Parasitaemia at the first time of ≥5000 parasites per mL blood
- Time to first dose of treatment with Riamet®: (datetime of first dose of Riamet® datetime of inoculation) / (24\*60\*60)
- Parasitaemia at first dose of treatment with Riamet®

The following secondary endpoint parameter will be derived:

- Time to parasite clearance: (datetime of first PCR below the limit of quantification datetime of first dose of Riamet®) / (24\*60\*60)
  - PCR below the limit of quantification is defined as (MBTESTCD = PARADENS) < 50 asexual parasites per mL.

(Partially) missing times will be imputed as specified in section 5.3.2.

For the creation of the graphs of parasitaemia by time point, the individual subject assessments will be mapped as follows:

- Time from first PCR positivity (days) = (datetime of assessment datetime of first PCR positivity) / (24\*60\*60)
  - o (Partially) missing times will be imputed as specified in section 5.3.2.



#### 2.1.3 Inferential statistics

#### 2.1.3.1 SECONDARY ENDPOINTS:

Blood-stage parasite profile before treatment with Riamet®

To characterise the blood-stage parasite profile before treatment with Riamet® is initiated, first, a log-linear mixed effect model will be fitted to the measured parasitaemia (in count/mL, transformed on natural log scale) data prior to Riamet® administration. In this model, for each individual i:

$$\begin{cases} \frac{d \ log \ Parasitaemia_i}{dt} = GR_i \\ log Parasitaemia_{0,i} = log F_{inoc,i} + log P_{inoc} - log V_{blood} \end{cases}$$

where t is the time in hours since inoculation,  $GR_i$  is the individual parasitaemia growth rate (measured in 1/hour), Parasitaemia<sub>o,i</sub> is the individual parasitaemia at time of inoculation (t=0),  $F_{inoc,i}$  is the individual inoculum viability,  $P_{inoc}$  is the inoculum size, which is fixed to 3200 parasites, and  $V_{blood}$  is the blood volume (in mL units) which is fixed to 5000 mL for all individuals:

If the measured parasitaemia profile shows a cyclic behaviour due to synchronicity of the parasites and their sequestration during the late stages of their lifecycle, an attempt will be made to model this behaviour using the following extended version of the log-linear model:

$$\begin{cases} \frac{d\ log\ Parasitaemia_{i}}{dt} = GR_{i} \\ log\ Parasitaemia_{0,i} = logF_{inoc,i} + logP_{inoc} - logV_{blood} \\ logParasitaemia_{visible,i} = log\ Parasitaemia_{i} + log\left\{1 - 0.5F_{max,i}\left[1 - \cos\left(\frac{2\pi(t/24 - D_{t,i})}{P_{len,i}}\right)\right]\right\} \end{cases}$$

where  $Parasitaemia_{visible,i}$  denotes the measured parasitaemia,  $D_{t,i} = \phi_i P_{len,i}$ ,  $F_{max,i}$  denotes the individual maximum fraction of hidden parasites,  $P_{len,i}$  denotes the individual period length of the oscillation (in hours), and  $\phi_i$  denotes the individual oscillation phase.

Parameter estimation will be performed using Monolix (Antony, France: Lixoft SAS). By default, all of the model parameters described above will be estimated, including their inter-individual variability (IIV) distributions. If, due to limited data size, the relative standard error (RSE) of the estimates exceeds 40%, the modeler may decide to fix the IIV for some of the parameters to previous estimates based on pooled data from induced blood-stage malaria VIS studies. By default, the models should assume independence of the parameters in their uncertainty and IIV distributions. If, during the model exploration, indications appear of a strong correlation between specific pairs of parameters, both, in their uncertainty and/or IIV distributions, the modeler may attempt to explicitly estimate such parameter correlations. Data below the limit of quantification will be included in the dataset and flagged as censored observations.

The following parameters will be determined from the population fits of the data:



- Parasite growth rate expressed as the parasite multiplication rate (PMR) standardised to 48 h (PMR<sub>48</sub>), i.e., ratio of the parasite density at a specific time point to the parasite density 48 h earlier. Based on the population estimates for the GR parameter in the log-linear mixed effect model, PMR<sub>48</sub> will be reported in log10 units: , i.e.  $PMR_{48} = \frac{48GR}{\log(10)}$
- If cycles are observed and if their estimated period is not 48 h, parasite growth rate expressed as the PMR per life cycle (PMR<sub>LC</sub>). Based on the population estimates for the GR and  $P_{len}$  parameters in the extended loglinear mixed effect model, PMR<sub>LC</sub> will be reported in log10 units:  $PMR_{LC} = \frac{P_{len}GR}{\log(10)}$ .
- Predicted time to reach parasitaemia thresholds of first positive PCR,  $\geq$ 5000 parasites per mL blood for Cohorts 1 and 2. All these quantities should be calculated at the population level by solving for t the linear equations  $logX = logParasitaemia_0 + GR \times t$

where  $X \in \{250, 5000\}$  and  $\log_{10} Parasitaemia_0$  and GR are the population estimates for parasitaemia at time of inoculation and parasitaemia growth rates respectively.

To determine confidence intervals for the population mean, parameters will be sampled from uncertainty.

#### Blood-stage parasite clearance profile after treatment with Riamet®

To characterise the blood-stage parasite clearance profile of Riamet® in malaria infection in naïve healthy participants after PfSPZ-DVI challenge; a log-linear model will be fitted to the parasitaemia data observed from the administration of the treatment onwards.

For each participant *i*:

$$\log_{10} Parasitaemia_{ij} = \beta_{0,i} + \beta_{1,i}t_{ij} + \varepsilon_{ij}$$

Where  $t_{ij}$  is the time in hours since administration of antimalarial treatment,  $\beta_{0,i}$  and  $\beta_{1,i}$  are the participant's intercept and slope, respectively, and  $\varepsilon_{ij}$  the error terms. For each participant i,  $\beta_{0,i}$  is the  $\log_{10}(\text{Parasitaemia at initiation of antimalarial treatment})$  and  $-\beta_{1,i}$  is the clearance rate constant.

The following algorithm will be used to remove potential lag and/or tail phases of the parasitaemia clearance profile, in order to determine the optimal log-linear decay regression (Marquart et al, 2015 see section 7). The algorithm considers removing parasitaemia data points in an iterative process from both ends of the parasitaemia curve, i.e. a combination of removing values from the tail phase and removing values from the lag phase.

The optimal log-linear regression model for a participant is deemed an appropriate fit if the overall model p-value < 0.001.

Iteration process to determine the optimal log-linear decay curve:

For each participant:



- Step 1: Fit the full model fit a linear regression (as defined by the previous equation) to all *m* parasitaemia values of participant *i*
- Step 2: Fit two models:
  - $\circ$  Fit linear regression model to m-1 parasitaemia values, removing the first observation
  - $\circ$  Fit linear regression model to m-1 parasitaemia values, removing the last observation
- Step 3: Determine the best model of Step 2a and Step 2b, defined as the model corresponding to the minimum overall model p-value
- Step 4: Of the best model defined in Step 3, repeat Step 2 and Step 3 in an iterative process until a minimum of four observations remain.
- Step 5: Of the m-3 best models selected per iteration (including the full model [Step 1]), the optimal model is defined by the minimum overall model p-value.

The following parameters will be calculated from the estimates of the optimal linear regression model for participant i:

- log<sub>10</sub> parasite reduction ratio per 48 h (log<sub>10</sub>PRR<sub>48</sub>), i.e., ratio of the parasite density at a specific time point to the parasite density 48 h later and expressed in log<sub>10</sub>
  - $\circ \log_{10} PRR_{48_i} = -48\beta_{1,i}$
- Parasite clearance half-life (PC50), i.e., time taken for the parasite density to be reduced by 50% after the first dose administration of Riamet®

$$O PC50_i = \log_{10}(2) \left( \frac{48 hours}{\log_{10} PRR_{48i}} \right) = \frac{\log_{10}(2)}{-\beta_{1i}}$$

• Predicted time to reach parasite clearance of 99% (PC99) is calculated solving for *t* the linear equation

$$\log_{10} X = \hat{\beta}_{0,i} + \hat{\beta}_{1,i} \times t$$

where  $\hat{\beta}_{0,i}$  is the participant's estimated  $\log_{10}(\text{Parasitaemia at initiation of Riamet}\mathbb{R})$ ,  $\hat{\beta}_{1,i}$  the opposite of clearance rate constant, and X the Parasitaemia at initiation of Riamet $\mathbb{R}$  / 100. Thus:

$$PC99_i = \frac{\log_{10}(100)}{-\beta_{1,i}}$$

Note: when computing descriptive statistics per cohort and overall of the above estimated parameters, the summary statistics will be estimated by using the inverse-variance method to calculate the weighted average linear regression slope ( $\bar{\beta}_1$ ) and corresponding standard error [SE( $\bar{\beta}_1$ )] (Hartung et al, 2008 see section 7). Descriptive statistics are based only on the participants whose optimal regression model overall p-value < 0.001.

#### 2.1.3.2 EXPLORATORY ENDPOINTS:

To characterise the individual variability the results of modelling the blood-stage parasite profile with a log-linear or cyclic growth model whichever best describes the data (Section 2.1.3.1) will be used. Based on the individual parameter estimates from



the NLME model the inter-individual variability of the parasite growth rate and the predicted time to reach parasitaemia threshold of first positive PCR, ≥5000 parasites per mL blood for Cohorts 1 and 2 will be calculated according to corresponding equations from Section 2.1.3.1. In case that the IIV can be estimated for all parameters, prediction intervals for these variables will be determined based on 1000 samples of individual parameters from the estimated IIV.

### 2.1.4 Presentation of results

All parasitaemia tables, listings and figures will be presented for the PD set. As a sensitivity analysis the tables and figures will also be presented for the modified PD set. In this set subjects with a PCR assessment below the limit of quantification (<50 parasites per mL) after first PCR positivity (>250 parasites per mL) but before first antimalarial treatment administration will be excluded.

All parasitaemia data will be listed, including all derived parameters. The onset date of antimalarial treatment administration will be added to the listing.

## Primary endpoints:

Descriptive statistics (N, geometric mean, geometric SD, 95% CI, minimum, maximum) will be provided for the following primary endpoints per cohort and overall:

- Time to first PCR positivity
- Parasitaemia at first PCR positivity
- Parasitaemia at the time of ≥5000 parasites per mL blood
- Time to first dose of treatment with Riamet®
- Parasitaemia at first dose of treatment with Riamet®

Time to parasitaemia of ≥5000 parasites per mL blood will be analysed using Kaplan-Meier time to event analysis per cohort and overall. The number of events, number of censored observations, 25th percentile, median and 75th percentile with 95% CI will be presented.

The number and proportion of participants with presence of positive PCR and parasitaemia of ≥5000 parasites per mL blood between inoculation with PfSPZ-DVI Challenge and Day 28 will be summarised per cohort. Corresponding two-sided 90% Exact Clopper-Pearson confidence limits will be presented as well.

Parasitaemia actual values in the base-10 logarithmic scale will be summarised by means of descriptive statistics at each analysis visit. The visits will be grouped by analysis phase.

Graphs of the median actual values over time and spaghetti plots of the individual participants will be prepared for parasitaemia in the base-10 logarithmic scale. The median plot will be shown from the Day 7 assessment to the assessment 72 h following initiation of Riamet®. The spaghetti plots will be shown from the subject's first PCR positivity to parasite clearance. For the spaghetti plots, different plotting symbols will be used on the first assessment when antimalarial treatment was given.

For all time to event parameters, Kaplan-Meier plots per cohort and overall will be presented.



### Secondary endpoints:

#### Blood-stage parasite profile before treatment with Riamet®

Parameter estimates for fixed (mean parameter value) and random (inter-individual and residual variability) effects values will be tabulated including their standard error and shrinkage for the inter-individual variability.

To characterise the blood-stage parasite profile the mean, 90%-CI will be provided for:

- PMR<sub>48</sub>
- PMR<sub>LC</sub> (if cycles are observed and their estimated period is not 48 h)
- Predicted time to reach parasitaemia threshold of first positive PCR, ≥5000 parasites per mL blood for Cohorts 1 and 2

#### Blood-stage parasite clearance profile after treatment with Riamet®

The model estimates and derived parameters resulting from the optimal log-linear decay regression model of each subject will be tabulated.

To characterise the blood-stage parasite clearance profile of Riamet® descriptive statistics (N, geometric mean, geometric SD, 95% CI, minimum, maximum) will be provided for time to parasite clearance per cohort and overall.

The following cohort parameters will be estimated based on the weighted average slope and standard error of the subjects with the optimal regression model having a p-value <0.001. N, mean, 95% CI, minimum and maximum will be shown.

- log<sub>10</sub> parasite reduction ratio per 48 h (log<sub>10</sub>PRR<sub>48</sub>)
- Parasite clearance half-life (PC50)
- Predicted time to reach parasite clearance of 99% (PC99)

For each subject, the regression slope with 95% CI,  $log_{10}PRR_{48}$  with 95% CI and overall model p-value of all the fitted models leading to the selection of the optimal log-linear model will be listed. The optimal model of each subject will be flagged.

A Kaplan-Meier plot per cohort and overall will be presented for the time to parasite clearance.

#### Exploratory endpoints:

Summary statistics of all individual parameters (cohort 1 and cohort 2) of the log-linear growth model will be tabulated to show the inter-individual variability of the parasite growth rate of predicted time to reach parasitaemia threshold of first positive PCR, ≥5000 parasites per mL blood by geometric mean, standard deviation (including their 95% CI), and the range. In case that the IIV could be estimated for all parameters, the 90% prediction interval and the median will be reported.



## 3. SAFETY ANALYSES

### 3.1 ADVERSE EVENTS

### 3.1.1 Available data

Adverse events (AEs) are coded into system organ classes and preferred terms using the medical dictionary for regulatory activities (MedDRA). For each AE, start and stop date(time)s are collected as well as grade, severity, a seriousness flag, relatedness to PfSPZ inoculum, relatedness to Riamet®, relatedness to Malarone®, action taken towards PfSPZ inoculum, action taken towards Riamet®, action taken towards Malarone®, outcome and a flag for AEs of special interest.

To determine severity of Adverse Events, including the 14 signs/symptoms as part of the Malaria Clinical Score, we use the CTCAE grading scale grade 1 - 5.

## 3.1.2 Derivation rules

Based on their start date(time), AEs will be allocated to the phase during which they started. Each AE will therefore be reported in only one phase. Phases are defined in section 5.2.1. In case the AE start date(time) is incomplete or missing and the AE could consequently be allocated to more than one phase, a worst-case allocation will be done as detailed below:

- Screening phase vs. challenge phase: AE will be allocated to the challenge phase unless the available parts of the AE start or stop date(time) provide evidence for allocating to the screening phase.
- Challenge phase vs. rescue phase: AE will be allocated to the rescue phase unless the available parts of the AE start or stop date(time) provide evidence for allocating to the challenge phase.

A fatal AE is defined as an AE with outcome 'fatal'.

An AE for which the antimalarial treatment was discontinued is defined as an AE with action taken 'Permanently discontinued' towards Riamet® or Malarone®.

Treatment-relatedness will be assessed for PfSPZ inoculum, Riamet® and Malarone®. It will be dichotomised as follows in tables:

- Treatment-related: Related/Suspected or missing.
- Not treatment-related: Not related/Not suspected or Not Applicable.

AE onset and duration will be calculated as follows when start and stop dates are fully known:

- AE onset day / hour (vs. first PfSPZ Challenge administration) =
  - AE start date > date of first inoculation: AE start date date of first inoculation + 1 day
  - o AE start date < date of first inoculation: AE start date date of first inoculation
  - AE start date = date of first inoculation (AE start datetime datetime of first inoculation)/(60\*60)



- AE onset day / hour (vs. start of phase) =
  - o AE start date > analysis phase start date: AE start date − analysis phase start date + 1 day
  - $\circ$  AE start date = analysis phase start date (AE start datetime analysis phase start datetime)/(60\*60)
- AE duration (days) =
  - AE end date AE start date + 1 day
  - study discontinuation date AE start date + 1 day (when the AE start date is fully known but the AE is not resolved at the end of the study)
     In this case the duration will be presented as ">x days".

(Partially) missing times will be imputed as specified in section 5.3.2.

### 3.1.3 Presentation of results

Tables will present only AEs that start after the PfSPZ Challenge inoculation. Preinoculation AEs will only be listed. Unless stated otherwise, tables will not be shown by phase.

An overview table will show the number and percentage of subjects with at least one event and the number of events for the following:

- AEs
- Serious AEs
- Grade  $\geq$  3 AEs
- Fatal AEs
- AEs related to PfSPZ inoculum
- AEs related to antimalarial treatment
- AEs related to Riamet®
- AEs related to Malarone®
- Serious AEs related to PfSPZ inoculum
- AEs for which the study was discontinued
- AEs for which the antimalarial treatment was discontinued
- AEs for which Riamet® was discontinued
- AEs for which Malarone® was discontinued
- AEs of special interest
- AEs of special interest related to PfSPZ inoculum
- AEs of special interest related to antimalarial treatment

Summary tables by MedDRA system organ class and preferred term will show the number and percentage of subjects with at least one event. The table of AEs will additionally show the number of events.



Separate tables will be prepared for the following:

- AEs
- Serious AEs
- Grade > 3 AEs
- AEs related to PfSPZ inoculum
- AEs related to antimalarial treatment (overall, related to Riamet® and related to Malarone®)
- Serious AEs related to PfSPZ inoculum
- AEs for which the antimalarial treatment was discontinued (overall, Riamet® discontinued and Malarone® discontinued)
- AEs of special interest related to PfSPZ inoculum
- AEs of special interest related to antimalarial treatment (overall, related to Riamet® and related to Malarone®)

Additionally, a summary table by MedDRA preferred term will show the number and percentage of subjects with at least one event, by descending order of frequency (number of subjects with events in the total group).

All AEs, including pre-inoculation events will be listed. Separate listings will be prepared for serious AEs, AEs after antimalarial treatment administration, AEs for which the study was discontinued, AEs for which the antimalarial treatment was discontinued (Riamet® or Malarone®), fatal AEs and AEs for which another action is taken. A listing showing all coding information will be prepared as well.

### 3.2 CLINICAL LABORATORY EVALUATION

## 3.2.1 Available data

Per protocol, the following laboratory parameters are expected:

- Biochemistry: Liver biochemistry: albumin, AST, ALT, alkaline phosphatase (ALP), gamma glutamyl aminotransferase (GGT), total and direct bilirubin and total serum proteins; Biochemistry other than liver: sodium, potassium, chloride, bicarbonate, urate, inorganic phosphate, creatinine, estimated glomerular filtration rate (eGFR), glucose, lactate dehydrogenase (LDH), blood urea nitrogen (BUN) and creatine phosphokinase (CPK); C-reactive protein (CRP); High sensitive troponin T;
- Haematology: haemoglobin, haematocrit, RBC count, mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), mean corpuscular volume (MCV), white blood cell (WBC) count, platelet count, reticulocytes, neutrophils, eosinophils, basophils, lymphocytes and monocytes;
- Coagulation: prothrombin time (PT), international normalised ratio (INR), activated partial thromboplastin time (aPTT);
- Urinalysis: dipstick for glucose, protein, nitrite, pH and occult blood; microscopic examination for WBC, RBC and casts.



Normal ranges are available as provided by the laboratory. Based on the Regulatory Agency's recommendation, the Clinically Acceptable Ranges for Clinically Important Study Inclusion Laboratory Tests (including total and conjugated bilirubin) have been added in Attachment 4 of the protocol to guide inclusion/exclusion of study participants.

## 3.2.2 Derivation rules

The following abnormality categories will be defined:

- Low: value < lower limit of normal range
- Normal: lower limit of normal range ≤ value ≤ upper limit of normal range
- High: value > upper limit of normal range

#### Note:

- Classification will be done in standardised units, using non-imputed values and limits.
- For the worst-case analysis visit, as defined in section 5.2.5, an additional category low + high is defined in case there are both low and high values.
- If not straightforward how to categorise urinalysis results, a worst-case approach will be used. A value of '4 to 6' with normal range '0 to 5' will thus be classified as normal for predose assessments but as high for post-dose assessments.

Additionally, for liver enzymes, the following elevation categories will be defined:

- ALT or AST >3 x Upper Limit of Normal (ULN);
- ALT or AST >5 x ULN;
- ALT or AST >8 x ULN;
- ALT or AST >3 x ULN and total bilirubin >2 x ULN at the same time point, together with a conjugated bilirubin fraction (direct bilirubin / total bilirubin) > 35% (Potential Hy's law cases).

## 3.2.3 Presentation of results

The statistical analysis will present results in standardised units.

Continuous laboratory parameters will be summarised by means of descriptive statistics at each analysis visit. Actual values and changes from baseline will be tabulated. Categorical parameters will be listed only.

Laboratory abnormalities will be presented as cross-tabulations of the abnormality at each post-baseline analysis visit and at the worst-case analysis visit versus the baseline abnormality. Numbers of subjects with post-baseline-emergent abnormalities will also be shown.

Additionally, a frequency table showing the liver enzyme elevation categories for the highest post-inoculation values will be prepared.

All laboratory data will be listed, but only for subjects with any post-baseline abnormality or clinically significant value.



Spaghetti plots of the individual subjects' actual values over time will be prepared for liver biochemistry parameters, CRP and haemoglobin. For the spaghetti plots, the median will also be plotted.

#### 3.3 VITAL SIGNS

## 3.3.1 Available data

The following vital signs parameters are collected: supine heart rate, supine systolic (SBP) and diastolic blood pressure (DBP), oral body temperature and body weight.

### 3.3.2 Derivation rules

Abnormalities are defined in below table.

| | Heart rate (bpm) | SBP<br>(mmHg) | DBP<br>(mmHg) | Temperature (°C) | Weight (kg) |
|---|---|---|---|---|---|
| Low | <40 | <90 | <45 | <35.0 | < 50 |
| Normal | 40-100 | 90-150 | 45-90 | 35.0-37.5 | 50-120 |
| High | >100 | >150 | >90 | >37.5 | >120 |

Note: For the worst-case analysis visit, as defined in section 5.2.5, an additional category low + high is defined in case there are both low and high values.

For the figures, the median assessment of first antimalarial treatment administration will be calculated starting from the individual vital signs first assessments which follow the first administration. In case the median is found to be between two assessments the first of the two will be selected.

### 3.3.3 Presentation of results

Vital signs parameters will be summarised by means of descriptive statistics at each analysis visit. Actual values and changes from baseline will be tabulated.

Abnormalities will be presented as cross-tabulations of the abnormality at each post-baseline analysis visit versus the baseline abnormality and as cross-tabulations of the worst-case abnormality versus the baseline abnormality. Numbers of subjects with post-baseline-emergent abnormalities will also be shown.

All vital signs data will be listed, but only for subjects with any post-baseline abnormality or clinically significant value.

Spaghetti plots of the individual subjects' actual values over time will be prepared for heart rate and body temperature. For the spaghetti plots, the median will also be plotted. The median time to first antimalarial treatment administration will be shown.



#### 3.4 ELECTROCARDIOGRAMS

### 3.4.1 Available data

The following electrocardiogram (ECG) parameters will be collected: heart rate (HR), QRS interval, PR interval, QT interval and corrected QT interval (Bazett and Fridericia). Recordings will be performed in triplicate.

## 3.4.2 Derivation rules

Mean values of the triplicates will be calculated per time point and rounded as detailed in section 5.3.4. Throughout the analysis, including the derivation of baseline and abnormalities, the mean values will be used. Individual triplicate values will only be listed.

Abnormalities for HR, QRS, PR and QTc interval are defined in below table.

| | HR (bpm) | PR (ms) | QRS (ms) | QTc (ms) |
|--------|----------|---------|----------|----------------------------------|
| Low | <40 | <120 | - | - |
| Normal | 40-100 | 120-220 | ≤120 | ≤450 for males, ≤470 for females |
| High | >100 | >220 | >120 | >450 for males, >470 for females |

Note: For the worst-case analysis visit, as defined in section 5.2.5, an additional category low + high is defined in case there are both low and high values.

For QTc interval changes (ms), the following categories are defined:

- $\leq$  30 (normal)
- $>30; \le 60$
- >60

Note: The worst-case, as defined in section 5.2.5, is the highest value and associated change.

### 3.4.3 Presentation of results

Uncorrected QT interval will only be listed.

Continuous ECG parameters will be summarised by means of descriptive statistics at each analysis visit. Actual values and changes from baseline will be tabulated.

Abnormalities of the actual values will be presented as cross-tabulations of the abnormality at each post-baseline analysis visit, and at the worst-case analysis visit versus the baseline abnormality. Numbers of subjects with post-baseline-emergent abnormalities will also be shown.

Abnormalities of the QTc changes will be presented as tabulations of the change abnormality at each post-baseline analysis visit and at the worst-case analysis visit. Cumulative numbers of subjects with change abnormalities will also be shown.

All ECG data will be listed, but only for subjects with any post-baseline abnormality or clinically significant value or change.

Spaghetti plots of the individual subjects' actual values over time will be prepared for QTcF and QTcB. For the spaghetti plots, the median will also be plotted.



### 3.5 MALARIA CLINICAL SCORE

## 3.5.1 Available data

The following 14 signs/symptoms frequently associated with malaria will be graded using a 4-point scale (absent: 0; mild: 1; moderate: 2; severe: 3): headache, myalgia (muscle ache), arthralgia (joint ache), fatigue/lethargy, malaise (general discomfort/ uneasiness), chills/shivering/rigors, sweating/hot spells, anorexia, nausea, vomiting, abdominal discomfort, fever, tachycardia and hypotension.

## 3.5.2 Derivation rules

Malaria clinical score is calculated as the sum of all (14) malaria sign and symptoms scores (maximum score is 42). Missing individual scores will be imputed as detailed in section 5.3.1. The score will be rounded as detailed in section 5.3.4.

For malaria clinical score and individual signs and symptoms, a worst-case analysis visit, as defined in section 5.2.5 will be derived.

For the creation of the graphs of malaria clinical score and parasitaemia/C-reactive protein together, the individual subject assessments will be mapped as follows:

- Time from PfSPZ inoculation (days) = (datetime of assessment datetime of inoculation) / (24\*60\*60)
  - o (Partially) missing times will be imputed as specified in section 5.3.2.

For the figures, the median assessment of first antimalarial treatment administration will be calculated starting from the individual MCS first assessments which follow the first administration. In case the median is found to be between two assessments the first of the two will be selected.

## 3.5.3 Presentation of results

For the malaria clinical score, actual values and changes from baseline will be evaluated by means of descriptive statistics at each time point and at the worst-case analysis visit (by phase and overall).

Individual malaria signs and symptoms scores will be presented as frequency tabulations at the worst-case analysis visit (by phase and overall). Numbers and percentage of subjects with any post-baseline non-zero score will also be shown.

Malaria signs and symptoms and clinical score will be listed. The onset date of antimalarial treatment administration will be added to the listing.

Malaria clinical scores of more than 6 will be listed. The baseline score value, the corresponding parasitaemia values at those analysis visits and the onset date of antimalarial treatment administration will be added to the listing.

Spaghetti plots of the individual subjects' actual values over time will be prepared for malaria clinical score. For the spaghetti plots, the median will also be plotted and different plotting symbols will be used at the time point of first antimalarial treatment administration and at the time point of peak parasitaemia. The median time to first antimalarial treatment administration will be shown.

Spaghetti plots of the individual subjects' actual values over time will be prepared for malaria clinical score and parasitaemia together. These plots will be shown per cohort

| SGS | Statistical Analysis Plan | |
|---|---|---|
| MMV_PfSPZ-DVI Blood<br>Stage_19_01 | | Final 1.0 of 11FEB2021 |

and per individual subject. The same type of plot will be prepared for malaria clinical score and C-reactive protein together.

## 3.6 PHYSICAL EXAMINATIONS

Abnormal physical examination findings will be listed.



## 4. GENERAL CHARACTERISTICS ANALYSES

### 4.1 SUBJECT DISPOSITION

The following subject data will be tabulated:

- The number of subjects in each analysis set
- Dates of first signed informed consent, last visit and last contact (overall only)
- The number and percentage of subjects who completed or discontinued the study as documented on the study termination page and the number and percentage of subjects for each study discontinuation reason

All information collected in the CRF concerning allocation, study discontinuation, antimalarial treatment discontinuation and information on phases will be listed. The phases listing will also include the start and stop dates of antimalarial treatment administration.

## 4.2 PROTOCOL DEVIATIONS AND ELIGIBILITY

The number and percentage of subjects with major protocol deviations will be tabulated, overall and per class of deviation.

All available information concerning major protocol deviations, violations on eligibility criteria and subjects not inoculated with PfSPZ-DVI Challenge will be listed.

## 4.3 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

## 4.3.1 Available data

The following parameters will be available:

- Demographics: sex, age, race, ethnicity, height, body weight at screening, date of signing informed consent form (ICF), smoking habits
- Screening laboratory tests: Viral serology: hepatitis A IgM antibody,
  HbsAg, anti-HCV antibody, hepatitis D antibody (only in subjects positive
  for HbsAg), hepatitis E IgM antibody, CMV IgM antibody, EBV IgM
  antibody and HIV; Urine drug screen (amphetamines, barbiturates,
  benzodiazepines, cannabinoids, cocaine and opiates) and alcohol breath test.
  In all female participants, serum β-HCG at screening and at the EOS visit,
  urine β-HCG on Day-1 and FSH at screening. rRT-PCR test on
  nasopharyngeal swab to screen for infection with SARS-CoV-2 at screening
  and prior to confinement to the study site on Day 10
- Standing and supine heart rate, standing and supine systolic (SBP) and diastolic blood pressure (DBP)
- Beck depression inventory (question 9 suicidal thoughts and total score)



#### 4.3.2 Derivation rules

The following parameters will be derived:

Body mass index (BMI) at screening (kg/m²) = (body weight at screening (kg)) / (height (m))²

Note: The BMI will only be recalculated and rounded as detailed in section 5.3.4 when not available in the database.

- Smoking status:
  - o Non-smoker: SUOCCUR = N
  - o Ex-smoker: SUOCCUR = Y and non-missing smoking end date
  - Smoker: SUOCCUR = Y and missing smoking end date
- Orthostatic change = value in supine position value in standing position
- Beck depression inventory interpretation:
  - o 0-10: Normal
  - o 11-16: Mild mood disturbance
  - o 17-20: Borderline clinical depression
  - o 21-30: Clinical depression
  - o 31-40: Severe depression
  - >40: Extreme depression

### 4.3.3 Presentation of results

Demographics will be presented using descriptive statistics for age, height, body weight and BMI and frequency tabulations for sex, race, ethnicity and smoking status.

Orthostatic change and Beck depression inventory will be presented using descriptive statistics for the total score and frequency tabulations for interpretation.

All demographic data will be listed. Separate listings will also be created for smoking history, orthostatic changes, Beck depression inventory, screening laboratory tests, pregnancy tests (including EOS result) and rRT-PCR tests.

### 4.4 MEDICAL HISTORY AND CONCOMITANT DISEASES

### 4.4.1 Available data

Medical history and concomitant diseases findings are coded using the medical dictionary for regulatory activities (MedDRA) into system organ classes and preferred terms. For each finding, a start and stop date or ongoing flag is collected.

### 4.4.2 Derivation rules

The following parameters will be derived:

- Medical history finding: not ongoing at screening (MHENRTPT =BEFORE)
- Concomitant disease finding: still ongoing at screening (MHENRTPT = ONGOING)



#### 4.4.3 Presentation of results

Medical history and concomitant diseases will be tabulated separately. Each table will show:

- The number and percentage of subjects with and without findings
- The number and percentage of subjects with findings by system organ class and preferred term

All medical history and concomitant diseases data will be listed separately.

## 4.5 PRIOR AND CONCOMITANT THERAPIES

### 4.5.1 Available data

All therapies (excluding antimalarial treatment) are coded using WHO-DRUG. ATC selection is performed. ATC coding up to level 4 is available in the clinical database. For each therapy, a start date or prior flag and stop date or ongoing flag are collected.

For antimalarial treatment the start and end date(times) and the dose will be recorded.

### 4.5.2 Derivation rules

Based on their start and stop date(time), prior and concomitant therapies will be allocated to each phase during which they were administered. A therapy can therefore be reported in more than one phase.

Phases are defined in section 5.2.1. Therapies with (partially) missing dates will be allocated to each phase unless the available parts of the therapy start or stop date(time) provide evidence the therapy was not taken during that phase.

### 4.5.3 Presentation of results

The number and percentage of subjects with and without therapies and the number and percentage of subjects with therapies by ATC class (level 4) and generic term will be tabulated by phase and overall. Blank ATC levels, if any, will be shown as 'not available' in the tables.

A frequency table will be prepared showing the timing of antimalarial treatment administration (prior to day 24 / on day 24) and the generic name (Riamet® / Malarone®).

The number and percentage of subjects who completed or discontinued the antimalarial treatment as documented on the treatment termination page and the number and percentage of subjects for each discontinuation reason will be tabulated.

All prior and concomitant therapies data will be listed. A separate listing will be prepared for antimalarial treatment administration.

### 4.6 EXPOSURE TO CHALLENGE AGENT

### 4.6.1 Available data

For the challenge agent (PfSPZ-DVI) the administration date(time) and the dose will be recorded.

| SGS | Statistical Analysis Plan | |
|---|---|---|
| MMV_PfSPZ-DVI Blood<br>Stage_19_01 | | Final 1.0 of 11FEB2021 |

## 4.6.2 Derivation rules

Not applicable.

## 4.6.3 Presentation of results

All exposure to challenge agent data will be listed.

| SGS | Statistical Analysis Plan | |
|---|---|---|
| MMV_PfSPZ-DVI Blood<br>Stage_19_01 | | Final 1.0 of 11FEB2021 |

## 5. GENERAL METHODOLOGY

## 5.1 ANALYSIS SETS

## 5.1.1 Analysis sets

The following analysis sets will be considered in the statistical analysis:

All screened subjects set

subjects who signed an informed consent to participate

(SCR):

in this study

Safety analysis set

subjects who were *inoculated* with PfSPZ-DVI

*(SAF)*:

Challenge

PD analysis set:

subjects from the safety analysis set with at least one available PD data who received all Riamet® doses and who experienced no major protocol deviations with

relevant impact on PD data

Modified PD analysis

*set (m-PD):* 

subjects from the PD analysis set excluding subjects with a PCR assessment below the limit of quantification

(<50 parasites per mL) after first PCR positivity (>250 parasites per mL) but before first antimalarial treatment

administration

#### Notes:

- Having signed an informed consent is defined as having a complete informed consent signature date in the database.
- Being inoculated with PfSPZ-DVI Challenge is defined as having an exposure date of PfSPZ-DVI Challenge or any information confirming this exposure present in the database.
- Major protocol deviations with impact on PD data will be identified with DVSCAT. DVSCAT = 'MISSING DATA EXPECTED PER PROTOCOL' indicates no impact on PD.

Unless specified otherwise, the safety analysis set will be used for the analysis of demographics and other general characteristics and for the safety/tolerability analysis. The PD analysis set will be used for pharmacodynamic statistical analysis. The modified PD analysis set will be used as a sensitivity analysis for the pharmacodynamic statistical analysis.

Protocol deviations will be reviewed and exclusion of subjects from the analysis sets will be decided during final data review prior to database lock.

## 5.1.2 As planned versus as actual analysis

Not applicable.

### 5.2 Phases and time points

#### **5.2.1 Phases**

All events and assessments will be allocated to phases. Seconds in the time part will be ignored.



| Phase | Start | End |
|---|---|---|
| Screening | Date of signing the ICF, with 00:00 added as time part | First inoculation date(time) – 1 minute |
| Challenge | First inoculation date(time) | First antimalarial treatment administration date(time) – 1 minute |
| Rescue | First antimalarial treatment administration date(time) | Date of last contact, with 23:59 added as time part |

Per definition, and for each subject, the first phase starts on the date of the earliest available ICF signature, and the last available phase ends on the date of last contact, with 23:59 added as time part.

AEs and concomitant therapies will be allocated to phases as described in sections 3.1.2 and 4.5.2 respectively. All other assessments will be allocated to phases based on the assessment date(time).

In case of (partially) missing date(time) fields, the visit label will be used to allocate to the correct phase. If this is not possible (unscheduled visits or visits on a turning point between phases), assessments will be handled as follows:

- Screening phase vs. challenge phase: assessments will be allocated to the challenge phase unless the available parts of the assessments start or stop date(time) provide evidence for allocating to the screening phase.
- Challenge phase vs. rescue phase: assessments will be allocated to the rescue phase unless the available parts of the assessments start or stop date(time) provide evidence for allocating to the challenge phase.

## 5.2.2 Baseline and change from baseline

The baseline value is the last available and non-missing value before the inoculation of PfSPZ-DVI Challenge. If all values are missing, the baseline will be reported as missing.

Change from baseline is defined as:

Change from baseline at time point t = value at time point t - baseline value.

## 5.2.3 Relative day

Relative days (DY) will be calculated according to the following rule:

- Concerned date < reference date: DY = concerned date reference date
- Concerned date  $\geq$  reference date: DY = concerned date reference date + 1

The reference date is the date of inoculation of PfSPZ-DVI Challenge.

## 5.2.4 Analysis visits

For assessments after the reference date, the analysis will use the visits and time points indicated on the subject's case report form (CRF). Unscheduled assessments after the reference date will only be listed.



The screening value is the last available and non-missing value before day -1. This value corresponds to the screening visit, except in case of retesting. Reason for this approach is the use of retest results for subject eligibility assessment.

The day -1 value is the last available and non-missing value performed on the date of day -1.

Baseline is defined in section 5.2.2.

## 5.2.5 Worst-case

A worst-case analysis visit will be created for parameters for which abnormalities are defined to summarise values considered as the worst-case. For abnormalities it is derived per parameter and in case both the lowest and the highest values are considered abnormal, a subject can have two worst-case analysis visits for a same parameter, which will be shown in tables as a combined high+low category. For malaria signs and symptoms, the worst-case corresponds to the highest score and is also derived per sign/symptom.

All non-missing post-baseline values, including unscheduled assessments and followup will be considered when deriving the worst-case analysis visit.

Worst-case will be derived both by phase (challenge/rescue) as relevant and overall.

#### 5.3 IMPUTATION AND ROUNDING RULES

## 5.3.1 Missing values

For the calculation of the malaria clinical score, missing individual signs and symptom scores will be imputed with the mean of all non-missing scores.

No other imputation will be done of missing values.

# 5.3.2 Handling partially or completely missing dates in calculations

For the time to event parasitaemia parameters, assessment datetimes used in the figures and AE onset hours, partially missing time parts will be imputed with zero (e.g. if minutes and seconds are missing time will be set to hh:00:00).

Note: If imputation of the start datetime results in a start datetime posterior to the stop datetime, the start datetime will be imputed with the stop datetime. If imputation of the stop datetime results in a stop datetime anterior to the start datetime, the stop datetime will be imputed with the start datetime.

No other date(time) imputation will be performed.

### 5.3.3 Values below or above a threshold

Safety values expressed as below (or above) the limit of quantification will be imputed by the value of the quantification limit itself.

Parasitaemia values below the limit of quantification (50 parasites/mL) will be imputed by 1 parasite per mL blood, which is equivalent to zero in the logarithmic scale.

Listings will always show the non-imputed values.



## 5.3.4 Rounding of derived variables

Derived variables will be rounded to the appropriate number of significant digits (see Definition of terms) at display level:

- Malaria clinical score will be rounded to 1 decimal.
- Mean of triplicates, mean scores and BMI will be rounded to 1 decimal.
- AE onset hour will be rounded to 1 decimal.
- Time to event parameters and log10(parasitaemia) will be rounded to 1 decimal.
- Other derived PD parameters will be rounded to 2 decimals.

Rounding will be done using the round half to up rule (see Definition of terms).

## 5.3.5 Outliers

There will be no outlier detection. All measured values will be included in the analyses.

## 5.4 Presentation of results

## 5.4.1 Calculation of descriptive statistics and percentages

For continuous parameters, full descriptive statistics will only be presented if there are at least 2 non-missing observations. Alternatively, only the number of non-missing data points and mean are shown.

Descriptive statistics of the general and safety parameters will include the number of non-missing data points, the arithmetic mean, the standard deviation (SD), the median, minimum and maximum.

Descriptive statistics of the pharmacodynamic endpoints will include the number of non-missing data points, the arithmetic or geometric mean and SD, the corresponding 95% confidence interval (CI), minimum and maximum. Geometric mean, geometric SD and CI are calculated as the exponentials of the arithmetic mean, SD and corresponding CI (based on t-distribution, without continuity correction) of the log-transformed data.

Mean, geometric mean, median, SD, geometric SD and CI will be presented with one more decimal place than the individual values. Minimum and maximum will be presented with the same number of decimal places than the individual values.

P-values will be presented with four decimal places, ratios with three decimal places and test statistics with two decimal places.

For event-type data, the denominator will be all subjects in the analysis set and phase. All cohorts will be shown, even if no events are present.

For frequency tabulations and cross-tabulations, missing values will not be included in the denominator count when computing percentages. For cross-tabulations of post-baseline results versus baseline results, a 'missing' category will be shown for baseline results if applicable.

Percentages will be shown with one decimal place.



## 5.4.2 Presentation of treatments

The following labels will be used in the tables, listings and figures:

- Cohort 1
- Cohort 2

In the analysis, a grand total will be added to summarise all subjects over cohorts except for parameters defined only for cohort 2. Grand totals will be shown last.

## 5.4.3 Ordering in tables, figures and listings

All tables and figures will be presented per cohort, unless specified otherwise.

All listings will be ordered by cohort, subject, analysis visit and time point, unless specified otherwise.

Tables will be sorted first by cohort, then by time point.

In tables and figures showing several parameters, each parameter will begin on a new page and parameters will be sorted alphabetically, within the parameter category if applicable.


### 6. CHANGES TO THE PLANNED ANALYSIS

### 6.1 CHANGES NOT COVERED BY PROTOCOL AMENDMENTS BEFORE DATABASE LOCK

- The inoculation set is renamed as safety analysis set and will be used for the general and safety analyses instead of the safety analysis set defined in the protocol as "all inoculated participants who received any treatment" (see protocol section 9.1).
- Time to first PCR positivity (defined as qPCR outcome ≥ 250 asexual parasites per mL blood): in the absence of positive PCR, the endpoint will not be derived instead of imputing the duration by 28 days.
- Time to parasitaemia of >= 5000 parasites per mL blood: summarised using Kaplan Meier estimates instead of geometric mean (95% CI), SD and range.
- Endpoints related to the 10000 parasites per mL blood are removed from the analysis since the threshold for Cohort 2 was modified to 5000 parasites per mL blood.
- log10PRR48, PC50 and PC99 are estimated using the weighted average slope and standard error of the subjects with the optimal regression model having a p-value <0.001.

### 6.2 CHANGES NOT COVERED BY PROTOCOL AMENDMENTS AFTER DATABASE LOCK

Not applicable.

6.3 CHANGES TO THE FINAL STATISTICAL ANALYSIS PLAN

Not applicable.



### 7. REFERENCES

ICH Topic E6(R2) Guideline for Good Clinical Practice – Step 4, 9 November 2016.

ICH guideline E14: the clinical evaluation of QT/QTc interval prolongation and proarrhythmic potential for non-antiarrhythmic drugs (R3) – questions and answers, January 2016.

ICH Topic E9 Statistical Principles for Clinical Trials – Step 5 – Note for Guidance on Statistical Principles for Clinical Trials (CPMP/ICH/363/96), September 1998.

Hartung J, Knapp G, Sinha B. 2008. Statistical meta-analysis with applications, p 35–41. John Wiley & Sons, Inc, Hoboken, NJ.

Leesa F Wockner, Isabell Hoffmann, Lachlan Webb, Benjamin Mordmüller, Sean C Murphy, James G Kublin, Peter O'Rourke, James S McCarthy, Louise Marquart, Growth Rate of Plasmodium falciparum: Analysis of Parasite Growth Data From Malaria Volunteer Infection Studies, The Journal of Infectious Diseases, Volume 221, Issue 6, 15 March 2020, Pages 963–972, <a href="https://doi.org/10.1093/infdis/jiz557">https://doi.org/10.1093/infdis/jiz557</a>.

Marquart, L.C., Baker, M., O'Rourke, P., & McCarthy, J.S. (2015). Evaluating the pharmacodynamic effect of antimalarial drugs in clinical trials by quantitative PCR. Antimicrobial agents and chemotherapy, 59 7, 4249-59.

### 8. LIST OF TABLES, LISTINGS AND FIGURES

### 8.1 TABLES

### GENERAL CHARACTERISTICS 14.1.1.1 Analysis Sets **SCR** 14.1.1.2 First and Last Contact in the Study **SCR** 14.1.1.3 SAF Study Discontinuation 14.1.1.4 Major Protocol Deviations SAF 14.1.2.1 Demographic Data SAF 14.1.2.2 Orthostatic Change in Vital Signs at Screening SAF 14.1.2.3 SAF Beck Depression Inventory at Screening 14.1.2.4 Medical History SAF 14.1.2.5 Concomitant Diseases SAF 14.1.2.6 Prior and Concomitant Therapies by ATC Class (Level 4) and Generic SAF 14.1.2.7 Antimalarial Treatment SAF 14.1.2.8 Antimalarial Treatment Discontinuation SAF **PHARMACODYNAMICS** 14.2.3.1.1 PD Time to First PCR Positivity (days): Descriptive Statistics 14.2.3.1.2 m-PD Time to First PCR Positivity (days): Descriptive Statistics 14.2.3.2.1 PD Parasitaemia at First PCR Positivity (parasites/mL): Descriptive Statistics 14.2.3.2.2 Parasitaemia at First PCR Positivity (parasites/mL): Descriptive Statistics m-PD 14.2.3.3.1 Time to Parasitaemia of ≥5000 Parasites per mL Blood (days): Kaplan PD Meier Estimates 14.2.3.3.2 m-PD Time to Parasitaemia of ≥5000 Parasites per mL Blood (days): Kaplan Meier Estimates 14.2.3.4.1 Parasitaemia at the Time of ≥5000 Parasites per mL Blood (parasites/mL): PD Descriptive Statistics 14.2.3.4.2 Parasitaemia at the Time of ≥5000 Parasites per mL Blood (parasites/mL): m-PD Descriptive Statistics 14.2.3.5.1 PD Time to First Dose of Treatment with Riamet (days): Descriptive Statistics 14.2.3.5.2 Time to First Dose of Treatment with Riamet (days): Descriptive Statistics m-PD 14.2.3.6.1 Parasitaemia at First Dose of Treatment with Riamet (Parasites/mL): PD **Descriptive Statistics** 14.2.3.6.2 Parasitaemia at First Dose of Treatment with Riamet (Parasites/mL): m-PD Descriptive Statistics 14.2.3.7.1 PD Incidence of Parasitaemia 14.2.3.7.2 Incidence of Parasitaemia m-PD 14.2.3.8.1 Blood-Stage Parasite Profile: Log-Linear Mixed Model Estimates PD 14.2.3.8.2 Blood-Stage Parasite Profile: Log-Linear Mixed Model Estimates m-PD



| 14.2.3.9.1 | Blood-Stage Parasite Profile: Extended Log-Linear Mixed Model Estimates | PD |
|---|---|---|
| 14.2.3.9.2 | Blood-Stage Parasite Profile: Extended Log-Linear Mixed Model Estimates | m-PD |
| 14.2.3.10.1 | Blood-Stage Parasite Profile: Model Derived Population Parameters | PD |
| 14.2.3.10.2 | Blood-Stage Parasite Profile: Model Derived Population Parameters | m-PD |
| 14.2.3.11.1 | Blood-Stage Parasite Profile: Model Derived Parameters Based on<br>Individual Parameter Estimates | PD |
| 14.2.3.11.2 | Blood-Stage Parasite Profile: Model Derived Parameters Based on<br>Individual Parameter Estimates | m-PD |
| 14.2.3.12.1 | Blood-Stage Parasite Profile: Model Derived Parameters Based on<br>Simulated Individual Parameter Values | PD |
| 14.2.3.12.2 | Blood-Stage Parasite Profile: Model Derived Parameters Based on<br>Simulated Individual Parameter Values | m-PD |
| 14.2.3.13.1 | Blood-Stage Parasite Clearance Profile: Individual Log-Linear Model Estimates | PD |
| 14.2.3.13.2 | Blood-Stage Parasite Clearance Profile: Individual Log-Linear Model Estimates | m-PD |
| 14.2.3.14.1 | Blood-Stage Parasite Clearance Profile: Descriptive Statistics | PD |
| 14.2.3.14.2 | Blood-Stage Parasite Clearance Profile: Descriptive Statistics | m-PD |
| 14.2.3.15.1 | Descriptive Statistics of log10(Parasitaemia) Actual Values | PD |
| 14.2.3.15.2 | Descriptive Statistics of log10(Parasitaemia) Actual Values | m-PD |
| SAFETY | | |
| ADVERSE I | EVENTS | |
| 14.3.1.1 | Adverse Events Overview | SAF |
| 14.3.1.2 | Adverse Events by MedDRA System Organ Class and Preferred Term | SAF |
| 14.3.1.3 | Adverse Events by MedDRA Preferred Term by Descending Order of Frequency | SAF |
| 14.3.1.4 | Serious Adverse Events by MedDRA System Organ Class and Preferred Term | SAF |
| 14.3.1.5 | Grade 3 or More Adverse Events by MedDRA System Organ Class and Preferred Term | SAF |
| 14.3.1.6 | PfSPZ Inoculum Related Adverse Events by MedDRA System Organ<br>Class and Preferred Term | SAF |
| 14.3.1.7 | Antimalarial Treatment Related Adverse Events by MedDRA System<br>Organ Class and Preferred Term | SAF |
| 14.3.1.8 | Serious PfSPZ Inoculum Related Adverse Events by MedDRA System<br>Organ Class and Preferred Term | SAF |
| 14.3.1.9 | Adverse Events for which the Antimalarial Treatment Was Discontinued by MedDRA System Organ Class and Preferred Term | SAF |
| 14.3.1.10 | Adverse Events of Special Interest Related to PfSPZ Inoculum by<br>MedDRA System Organ Class and Preferred Term | SAF |
| 14.3.1.11 | Adverse Events of Special Interest Related to Antimalarial Treatment by MedDRA System Organ Class and Preferred Term | SAF |



| I ADODA' | TORY DATA | |
|---|---|---|
| | | CAE |
| 14.3.2.1<br>14.3.2.2 | Descriptive Statistics of Laboratory Test Results | SAF<br>SAF |
| _ | Cross-Tabulation of Laboratory Abnormalities Versus Baseline | |
| 14.3.2.3 | Liver Enzyme Elevation Categories | SAF |
| VITAL SI | | CAE |
| 14.3.3.1 | Descriptive Statistics of Vital Signs | SAF |
| 14.3.3.2 | Cross-Tabulation of Vital Signs Abnormalities Versus Baseline | SAF |
| ECG | D. J. J. G. J. J. ADGG | G A F |
| 14.3.4.1 | Descriptive Statistics of ECG | SAF |
| 14.3.4.2 | Cross-Tabulation of ECG Abnormalities Versus Baseline | SAF |
| 14.3.4.3 | Tabulation of QTc Change Abnormalities | SAF |
| | A CLINICAL SCORE | |
| 14.3.5.1 | Descriptive Statistics of Malaria Clinical Score | SAF |
| 14.3.5.2 | Frequency Table of the Worst-Case Individual Malaria Signs and Symptoms | SAF |
| 8.2 L | ISTINGS | |
| GENERA | L CHARACTERISTICS | |
| 16.2.1.1 | Allocation | SCR |
| 16.2.1.2 | Analysis Phases | SAF |
| 16.2.1.3 | Study and Antimalarial Treatment Discontinuation | SAF |
| 16.2.2.1 | Major Protocol Deviations | SAF |
| 16.2.2.2 | Violations on Eligibility Criteria | SAF |
| 16.2.2.3 | No-Inoculated Subjects | SCR<br>minus<br>SAF |
| 16.2.4.1 | Demographic Data | SAF |
| 16.2.4.2 | Smoking History | SAF |
| 16.2.4.3 | Orthostatic Change in Vital Signs at Screening | SAF |
| 16.2.4.4 | Beck Depression Inventory at Screening | SAF |
| 16.2.4.5 | Screening Laboratory Tests | SAF |
| 16.2.4.6 | Pregnancy Tests | SAF |
| 16.2.4.7 | rRT-PCR Tests for SARS-CoV-2 Infection | SAF |
| 16.2.4.8 | Medical History | SAF |
| 16.2.4.9 | Concomitant Diseases | SAF |
| 16.2.4.10 | Prior and Concomitant Therapies | SAF |
| 16.2.4.11 | Antimalarial Treatment | SAF |
| 16.2.4.12 | Comments | SAF |
| 16.2.5.1 | Exposure to Challenge Agent | SAF |



| PHARMA | ACODYNAMICS | |
|---|---|---|
| 16.2.6.1 | Parasitaemia | PD |
| 16.2.6.2 | Parasitaemia Endpoints | PD |
| 16.2.6.3 | Blood-Stage Parasite Clearance Profile: Iteration Process to Determine the Optimal Log-Linear Model | PD |
| SAFETY | | |
| ADVERS | E EVENTS | |
| 16.2.7.1 | Adverse Events | SAF |
| 16.2.7.2 | Serious Adverse Events | SAF |
| 16.2.7.3 | Fatal Adverse Events | SAF |
| 16.2.7.4 | Adverse Events for Which the Study Was Discontinued | SAF |
| 16.2.7.5 | Adverse Events for Which the Antimalarial Treatment Was Discontinued | SAF |
| 16.2.7.6 | Adverse Events after Administration of Antimalarial Treatment | SAF |
| 16.2.7.7 | Adverse Events for Which Another Action Is Taken | SAF |
| 16.2.7.8 | Adverse Events: Coding Information | SAF |
| 16.2.7.9 | Physical Examinations Abnormalities | SAF |
| LABORA | TORY DATA | |
| 16.2.8.1 | Laboratory Test Results for Subjects with Abnormal Values | SAF |
| VITAL SI | GNS | |
| 16.2.9.1 | Vital Signs Results for Subjects with Abnormal Values | SAF |
| ECG | | |
| 16.2.10.1 | ECG Results for Subjects with Abnormal Values | SAF |
| 16.2.10.2 | ECG Interpretation and Morphology for Subjects with any Abnormal Interpretation | SAF |
| MALARI | A CLINICAL SCORE | |
| 16.2.11.1 | Malaria Signs and Symptoms | SAF |
| 16.2.11.2 | Malaria Clinical Scores > 6 and Parasitaemia | SAF |
| 8.3 I | FIGURES | |
| PHARMA | ACODYNAMICS | |
| 14.2.3.1.1 | Blood-Stage Parasite Profile: Median Parasitaemia Actual Values over Time | PD |
| 14.2.3.1.2 | Blood-Stage Parasite Profile: Median Parasitaemia Actual Values over Time | m-PD |
| 14.2.3.2.1 | Blood-Stage Parasite Profile: Individual Parasitaemia Actual Values over Time | PD |
| 14.2.3.2.2 | Blood-Stage Parasite Profile: Individual Parasitaemia Actual Values over Time | m-PD |
| 14.2.3.3.1 | Time to first PCR positivity: Kaplan Meier Plot | PD |
| 14.2.3.3.2 | Time to first PCR positivity: Kaplan Meier Plot | m-PD |



| 14.2.3.4.1 | Time to parasitaemia of $\geq$ 5000 parasites per mL blood: Kaplan Meier Plot | PD |
|---|---|---|
| 14.2.3.4.2 | Time to parasitaemia of $\geq$ 5000 parasites per mL blood: Kaplan Meier Plot | m-PD |
| 14.2.3.5.1 | Time to First Dose of Treatment with Riamet: Kaplan Meier Plot | PD |
| 14.2.3.5.2 | Time to First Dose of Treatment with Riamet: Kaplan Meier Plot | m-PD |
| 14.2.3.6.1 | Time to Parasite Clearance: Kaplan Meier Plot | PD |
| 14.2.3.6.2 | Time to Parasite Clearance: Kaplan Meier Plot | m-PD |
| LABORAT | FORY DATA | |
| 14.3.2.1 | Individual Laboratory Test Actual Values over Time | SAF |
| VITAL SIC | GNS | |
| 14.3.3.1 | Individual Vital Signs Actual Values over Time | SAF |
| ECG | | |
| 14.3.4.1 | Individual ECG Actual Values over Time | SAF |
| MALARIA | CLINICAL SCORE | |
| 14.3.5.1 | Individual Malaria Clinical Score Actual Values over Time | SAF |
| 14.3.5.2 | Individual Malaria Clinical Score and Parasitaemia Actual Values over Time | SAF |
| 14.3.5.3 | Individual Malaria Clinical Score and CRP Actual Values over Time | SAF |



### 9. APPENDICES

### 9.1 SAS CODE

Blood-stage parasite clearance profile:

```
data ds;
    set ...;
    laval = log10(aval);
run;

proc glm data = ds alpha = 0.05;
    by usubjid;
    model laval = areltm / clparm;
run;
```

| Statistical Analysis Plan | MMV PfSPZ-DVI Blood<br>Stage_19_01 |
|---------------------------|------------------------------------|
| Ses | MMV_PfSPZ-DVI Blood<br>Stage_19_01 |

## 9.2 SCHEDULE OF ASSESSMENTS

| | EOS Visit y 28 <sup>Error! Reference sour</sup> | ce not found | × | | | 8 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | ı | | L | | | | | | | | | |
| | Day of Discharge From<br>Confinement: Day of<br>Parasite Clearance<br>(0 Parasites/mL) AND ≥72<br>h After Initiating<br>Antimalarial Therapy | Estimated On or Before<br>Day 19 | | | (X) | × | | | | | | |
| ۵. | Day of First PCR<br>≥5000 Parasites/mL Until≥72 h<br>After Initiating Antimalarial<br>Therapy | | | | X | | | | | | | |
| Challenge, treatment and follow-up | Day of First PCR<br>≥250 Parasites/mL Until<br>Day of First PCR<br>≥5000 Parasites/mL | | | | X | | | | | | | |
| Challe | Day 10: Start of<br>Confinement in<br>Clinical Unit | | | | X | | | | | | | |
| | Day 7-9 | | X | X | | | | | | | | |
| | Day 2-6 | | | | | | Х | | | | | |
| | 1 | 7 | | | | × | | | | | | |
| | Day 1 | 0 Errαt! Reference source not found. | | | × | | | | | | | |
| | Day -1 <sup>Er</sup> ror! Reference source not found. | | | | × | | | X | | | | |
| | Screening Vis Day -28 to Day | | × | × | | | | × | × | × | × | × |
| Assessments | Study Day/Event | Time point (h) in relation to PfSPZ-DVI Challenge | Ambulatory visit | Ambulatory visit (SARS-CoV-2 test) | Confinement in clinical unit <sup>Error!</sup> | Discharge from clinical unit | Telephonic<br>Monitoring for AEs | Eligibility criteria | Informed consent <sup>Error!</sup><br>Reference source not found. | Demographics | Medical and social history | Beck Depression<br>Inventory |

| SES | <br>MMV_PfSPZ-DVI Blood | Stage 19_01 |
|-----|-------------------------|-------------|
| | <br> | |

### Statistical Analysis Plan

Final 1.0 of 11FEB2021

| | EOS Visit | | Π | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Da | y 28 <sup>Error!</sup> Reference source | ce not found. | | × | × | × | | | × | | | × | X |
| | Day of Discharge From<br>Confinement: Day of<br>Parasite Clearance<br>(0 Parasites/mL) AND ≥72<br>h After Initiating<br>Antimalarial Therapy | Estimated On or Before<br>Day 19 | | | X | X | | | | | | X | X |
| a | Day of First PCR<br>≥5000 Parasites/mL Until ≥72 h<br>After Initiating Antimalarial<br>Therapy | | | | X | X | X | | | | X | × | X |
| Challenge, treatment and follow-up | Day of First PCR<br>≥250 Parasites/mL Until<br>Day of First PCR<br>≥5000 Parasites/mL | | | | × | X | | | | | | × | × |
| Challe | Day 10: Start of<br>Confinement in<br>Clinical Unit | | | | X | X | | | | | | X | X |
| | Day 7-9 | | | | | | | | | | | × | X |
| | Day 2-6 | | | | | | | | | | | | |
| | - | 2 | | | | × | | | | | | | |
| | Day 1 | OError!<br>Reference<br>source not<br>found. | | | | × | | | | × | | × | |
| | Day -1 Er ror! Reference source not found. | | × | × | × | × | | | × | | | | X |
| | Screening Vis<br>Day -28 to Day | | × | × | × | × | × | × | × | | | | X |
| Assessments | Study Day/Event | Time point (h) in relation to PfSPZ-DVI Challenge | Alcohol & drug<br>ScreenError! Reference<br>source not found. | Height & weightError!<br>Reference source not found. | Physical examination | Vital signs <sup>Error!</sup><br>Reference source not found. | 12-lead ECG <sup>Error!</sup><br>Reference source not found. | Viral serology Error!<br>Reference source not found. | Pregnancy test <sup>Error!</sup> Reference source not found. | DVI of P/SPZ<br>Challenge | Riamet® | Malaria Clinical<br>Score Error! Reference source<br>not found. | Haematology & liver biochemistry |

| SES | V_PfSPZ-DVI Blood | Stage_19_01 |
|----------|-------------------|-------------|
| <b>O</b> | MMV | Stage |

Statistical Analysis Plan

Final 1.0 of 11FEB2021

| Assessments | | | | | | | Challe | Challenge, treatment and follow-up | di di | | Da |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day/Event | Screening Vis<br>Day -28 to Day | Day -1 <sup>Er</sup> ror! Reference source not found. | Day 1 | y 1 | Day 2-6 | Day 7-9 | Day 10: Start of<br>Confinement in<br>Clinical Unit | Day of First PCR 2250 Parasites/mL Until Day of First PCR 25000 Parasites/mL | Day of First PCR<br>>5000 Parasites/mL Until >72 h<br>After Initiating Antimalarial<br>Therapy | Day of Discharge From Confinement: Day of Parasite Clearance (0 Parasites/mL) AND > 72 h After Initiating Antimalarial Therapy | EOS Visit |
| Time point (h) in relation to PASPZ-DVI Challenge | -2 | | 0 Error!<br>Reference<br>source not<br>found. | 2 | | | | | | Estimated On or Before<br>Day 19 | ce not found. |
| Biochemistry other<br>than liverError! Reference<br>source not found. | × | × | | | | | × | | × | | X |
| CRP analysis Error!<br>Reference source not found. | | × | | | | X | × | X | X | X | × |
| Coagulation<br>parameters Error!<br>Reference source not found. | × | × | | | | X | × | X | × | X | X |
| rRT-PCR for SARS-<br>CoV-2 | X | | | | | Xs | | | | | |
| qPCR for<br>parasitesError! Reference<br>source not found. | | | × | | | X | X | X | × | X | × |
| Parasite Transcriptomics | | | | | | X | × | X | × | X | × |
| Previous medications | × | | | | | | | | | | |
| Concomitant<br>medications | | X | | | | | | | | Χ | |
| AEs | | XX | | | | | | | | Χ | |
| SAE reporting | | XX | | | XX | | | | | X | |

β-HCG: β-human chorionic gonadotropin, AE: adverse event, aPTT: activated partial thromboplastin time, CMV: cytomegalovirus, CRP: C-reactive protein, DVI: direct venous inoculation, EBV: Epstein Barr Virus, ECG: electrocardiogram, EOS: end of study, FSH: follicle stimulating hormone, HbsAg: hepatitis B surface antigen, HCV: hepatitis C virus, HIV: human immunodeficiency virus, IgM: immunoglobulin M, INR: international normalized ratio, *P/SPZ: Plasmodium falciparum* sporozoites, PT: prothrombin time, qPCR: quantitative polymerase chain reaction, rRT-PCR: real-time reverse transcription polymerase chain reaction, SAEs: serious adverse event, SARS-CoV-2: severe acute respiratory syndrome coronavirus 2



- a. Assessments begin as of participant confinement in the clinical unit and must be completed and safety assessment outcomes must be available before PfSPZ-DVI Challenge on Day 1.
- b. On Day 1, assessments begin as of 3 h before challenge (except for urinalysis assessments, morning void allowed). The assessments indicated must be completed and safety assessment outcomes must be available before PfSPZ-DVI Challenge inoculation.
- c. Confinement to the clinical unit will occur as follows:
- Participants will be admitted to the clinical unit in the morning of Day -1 and discharged from confinement 2 h post P/SPZ-DVI Challenge on Day 1.
- antimalarial therapy), estimated to occur on or before Day 19. Of note, participants who commence antimalarial therapy on Day 24 (see ) will only be Participants will be admitted to the clinical unit in the morning of Day 10 and discharged on Day of discharge from confinement (Day of parasite clearance AND \( \geq 72\) hafter initiating discharged from confinement at the end of the EOS visit on Day 28.
- d. No study-related procedure is to be performed before voluntarily signing of the informed consent form.
- e. Alcohol breath test and urine dipstick screening for drug abuse.
- f. Height to be measured at screening only; body weight to be measured at screening, at admission on Day -1 and at the EOS visit.
- g. Physical examination will be conducted:
- once at screening and once on Day -1;
- once on Day 10 (upon admission to clinical unit for confinement);
- once within 24 h after first PCR > 250 parasites/mL;
- once within 24 h after first PCR >5000 parasites/mL;
- once at pre-discharge from clinical unit on Day of discharge from confinement (Day of parasite clearance AND  $\geq$ 72 h after initiating antimalarial therapy); and
- once at the EOS.

Full physical examination will be conducted at screening, on Day -1, within ±24 h after first PCR ≥250 parasites/mL and at the EOS visit on Day 28. Targeted (symptom-driven) physical examination will be performed on the other time points in case malaria clinical score >6.

- h. Vital signs (blood pressure and pulse) will be measured after remaining in a supine position for at least 10 min. All measurements will be performed as follows:
- once at screening and once on Day -1;
- on Day 1 (pre and post *Pf*SPZ-DVI Challenge);
- twice daily from Day 10 (admission to clinical unit for confinement) onwards until Day of discharge from confinement (Day of parasite clearance AND >72 h after initiating antimalarial
- once at the EOS.

At screening, orthostatic changes to blood pressure and pulse rate will also be assessed: participants will be requested to stand after completion of the supine measurements and blood pressure Body temperature (sublingual) will also be assessed, and this whenever the malaria clinical score will be evaluated (see ).

and pulse rate will be recorded after at least 2 min in the standing position.



- i. 12-lead ECGs recordings will be performed in triplicate after participants have remained in a supine position for at least 10 min. All recordings will be performed as follows:
- once at screening; and
- once on Days 2 and 3 of antimalarial therapy.
- Serological testing for HIV, hepatitis A IgM antibody, HbsAg, anti-HCV antibody, hepatitis D antibody (only in subjects positive for HbsAg), hepatitis E IgM antibody, CMV IgM antibody and EBV IgM antibody, to determine eligibility for the study.
- k. Pregnancy testing consists of serum  $\beta$ -HCG assessments at screening and at the EOS visit and a urine  $\beta$ -HCG assessment on Day-1.
- P/SPZ-DVI Challenge will commence antimalarial therapy no later than Day 24, regardless if they reach the pre-defined cohort-specific PCR parasitaemia/malaria clinical score thresholds (i.e., possible when a PCR threshold of 5000 parasites/mL is achieved or earlier if a participant has a malaria clinical score >6 or at Investigator's discretion. Of note, all participants inoculated with 1. Every participant will be prescribed a 3-day oral course of Riamet® (20 mg artemether and 120 mg lumefantrine tablets) (see Protocol Section 5.1). The first dose should be taken as soon as 5000 parasites/mL blood and/or a malaria clinical score ≥6) (see Protocol Section 4.3).

If an intolerance or contraindication to Riamet® develops since inclusion, Malarone® will be administered (see Protocol Section 5.1).

m.Malaria clinical score for malaria signs and symptoms and the vital sign parameter body temperature (sublingual) (see ) are assessed:

- on Day 1 (pre-PfSPZ-DVI Challenge);
- once daily during ambulatory visits on Day 7, 8 and 9;
- twice daily from Day 10 (admission to clinical unit for confinement) onwards until Day of discharge from confinement (Day of parasite clearance AND \( \geq 72\) h after initiating antimalarial
- once at the EOS.

n. Haematology and liver biochemistry laboratory tests will be performed after overnight fast for at least 8 h (see Protocol Section 4.3):

- once at screening and once on Day -1;
- once during ambulatory visit on Day 7
- once on Day 10 (upon admission to clinical unit for confinement);
- once within 24 h after first PCR > 250 parasites/mL;
- once at pre-discharge from clinical unit on Day of discharge from confinement (Day of parasite clearance AND \( \geq 72\) h after initiating antimalarial therapy); and once on Day of first PCR ≥5000 parasites/mL AND prior to initiating antimalarial therapy (non-fasted state allowed);
- FSH will be measured at screening in all women.

Troponin T will be measured at screening (fasted state), at baseline prior to inoculation on Day -1 (fasted state), and on Days 1, 2 and 3 of antimalarial therapy (non-fasted state).

o. Biochemistry laboratory tests other than liver (including urinalysis, morning void allowed) will be performed after overnight fast for at least 8 h (see Protocol Section 4.3):

- once at screening and once on Day -1;
- once on Day 10 (upon admission to clinical unit for confinement);
- once on Day of first PCR ≥5000 parasites/mL AND prior to initiating antimalarial therapy (non-fasted state allowed); and
- once at the EOS

| SGS Statistical Analysis Plan | MMV_PRPZ-DVI Blood<br>Stage_19_01 |
|-------------------------------|------------------------------------|
| Ses | MMV_PfSPZ-DVI Blood<br>Stage_19_01 |

p. CRP laboratory tests will be performed at the following time points:

- once during ambulatory visit on Day 7;
- once on Day 10 (upon admission to clinical unit for confinement);
- once within 24 h after first PCR > 250 parasites/mL;
- once on Day of first PCR >5000 parasites/mL AND prior to initiating antimalarial therapy;

- once at pre-discharge from clinical unit on Day of discharge from confinement (Day of parasite clearance AND \( \geq 72\) h after initiating antimalarial therapy); and

- q. INR, PT and aPTT laboratory tests will be performed once at screening and once on Day -1. On the other time points thereafter, only the INR test will be performed.
- r. A nasopharyngeal swab will be taken at an ambulatory visit during screening up to Day -2 (preferably as close as possible to the day of admission, based on test capacity and according to national laws) from participants who are still eligible to be enrolled in the study after completing all other screening tests. An rRT-PCR test will be performed on these swabs to screen for infection with
- s. A nasopharyngeal swab will be taken prior to confinement to the study site on Day 10, based on test capacity and according to national laws.
- t. Blood samples for the assessment of parasitaemia by qPCR will be drawn at the following time points:
- on Day 1 (pre-PfSPZ-DVI Challenge);
- once daily during ambulatory visits on Day 7, 8 and 9;
- twice daily from Day 10 (admission to clinical unit for confinement) onwards until Day of first PCR \$5000 parasites/mL AND prior to initiating antimalarial therapy;
- at multiple time points (2, 6, 8, 12, 16, 24, 36, 48 and 72 h) following initiation of Riamet®;
- once on Day of discharge from confinement (Day of parasite clearance AND  $\geq$ 72 h after initiating antimalarial therapy); and

once at the EOS.

- All qPCR blood samples will be drawn for immediate analysis, except for the ones drawn at the multiple time points during Riamet® therapy.
  - u. Blood samples for parasite transcriptomics will be drawn at the following time points:
- once daily during ambulatory visits on Day 7, 8 and 9;
- once daily from Day 10 (admission to clinical unit for confinement) onwards until Day of discharge from confinement (Day of parasite clearance AND ≥72 h after initiating antimalarial therapy); and
  - once at the EOS.
- v. All participants will be asked non-leading questions to determine the occurrence of any AEs at the EOS visit.

Of note, for participants who commence antimalarial therapy on Day 24 (), the Day of discharge from confinement will coincide with the EOS. In this case, applicable assessments will not be performed in duplicate

# MOCK TABLES, LISTINGS AND FIGURES

A single centre, open label, pilot phase Ib study to investigate blood stage malaria infection after Direct Venous Inoculation of cryopreserved Plasmodium falciparum (NF54 strain) Sporozoites (PfSPZ-DVI) in malaria naïve

healthy adult volunteers

Protocol: MMV\_PfSPZ-DVI Blood Stage\_19\_01

**SGS LS number:** BE-80-1914715

Development phase: Ib

Sponsor: Medicines for Malaria Venture (MMV)

Mock TLF version number: Final 1.0

SAP version date: 11FEB2021


### SIGNATURE PAGE

| Name and function | Date (ddMMMyyyy) | Signature |
|---|---|---|
| SGS-LS author(s): | | |
| Daniel Izquierdo<br>Juncàs, Biostatistician | 11FEB2021 | Daniel Izquierdo Juncas Daniel Izquierdo Juncas Signer Name: Daniel Izquierdo Juncas Signer Reason: I am the author of this document Signing Reason: I am the author of this document Signing Time: 11-Feb-2021 16:10 CET |
| Bastiaan Jansen,<br>Biostatistical<br>Coordinator | 11FEB2021 | DocuSigned by: bastiaan Jansen Signer Name: 11-Feb-2021 16.23 CET Signing Time: 11-Feb-2021 16.23 CET 15ADFC6D3E734686B167F978EA41202B |
| Sponsor's approval:<br>The approver agrees the ta | ables, listings and fi | Sponsor's approval:<br>The approver agrees the tables, listings and figures of the statistical analysis will be created according to this document. |
| Farouk Chughlay,<br>Project and Medical<br>Director | | DocuSigned by: Description Description |
| Myriam El Gaaloul<br>Director, Clinical<br>Sciences | | DocuSigned by: Myriam El Gaaloul Signing Reason: lapprove this document Signing Reason: lapprove this document Signing Time: 13-Feb-2021 01:24 PST C2CA71F33AA843DAB327CC3B36DFB37C |


### TABLE OF CONTENTS General Characteristics General Characteristics Table of contents of the Listings Table of contents of the Tables Malaria clinical score Pharmacodynamics Pharmacodynamics Laboratory data Laboratory data Adverse events Adverse events Vital signs Vital signs 1. Table of contents ECG Signature page 1.1.1 1.1.2 1.1.4 1.1.7 1.2.1 1.1.3 1.1.5 1.1.6 1.2.2 1.2.4 1.2.5 1.2.3 1.2

 $\infty$ 6 6 10

12 12 12 13 13 13 14 14

Table of contents of the Figures

1.3

Pharmacodynamics

1.3.1

Malaria clinical score

ECG

1.2.6 1.2.7

| MM | I-ZdSłd_/ | MMV_PfSPZ-DVI Blood Stage_19_01 Mock Tables, Listings and Figures | Final 1.0 of 11FEB2021 |
|---|---|---|---|
| | 1.3.2 | Laboratory data | 14 |
| | 1.3.3 | Vital signs | 14 |
| | 1.3.4 | ECG | 14 |
| | 1.3.5 | Malaria clinical score | 14 |
| 2. | General la | General layout of a TLF | 15 |
| 2.1 | Softwa | Software used | 15 |
| 2.2 | Layout | Layout specifications in SAS | 15 |
| 2.3 | Layout | Layout specifications in MS Word | 17 |
| 2.4 | Genera | General table layout | 18 |
| | 2.4.1 | Standard layout for descriptive statistics on continuous parameters | 18 |
| | 2.4.2 | Standard layout for frequency tabulations | 19 |
| | 2.4.3 | Standard layout for table containing descriptive statistics and frequency tabulations | 20 |
| | 2.4.4 | Standard layout of an analysis table of contents | 21 |
| 2.5 | Genera | General figure layout | 22 |
| 3. | Mock tables | les | 23 |
| 3.1 | Genera | General characteristics | 23 |
| | 3.1.1 | Subject disposition | 23 |
| | 3.1.2 | Protocol deviations and eligibility | 26 |
| | 3.1.3 | Demographic and other baseline characteristics | 27 |
| | 3.1.4 | Medical history and concomitant diseases | 31 |
| | 3.1.5 | Prior and concomitant therapies | 32 |

| MM | V_PfSPZ-Ľ | MMV_PfSPZ-DVI Blood Stage_19_01 Mock Tables, Listings and Figures | Final 1.0 of 11FEB2021 | 21 |
|---|---|---|---|---|
| 3.2 | Pharma | Pharmacodynamics | 3 | 35 |
| 3.3 | Safety | | 5 | 51 |
| | 3.3.1 | Adverse events | 5 | 51 |
| | 3.3.2 | Clinical laboratory evaluation | 5 | 28 |
| | 3.3.3 | Vital signs | 9 | 61 |
| | 3.3.4 | Electrocardiograms (ECG) | 9 | 62 |
| | 3.3.5 | Malaria clinical score | 9 | 65 |
| 4. | Mock listings | Säu | 9 | 89 |
| 4.1 | Genera | General characteristics | 9 | 89 |
| | 4.1.1 | Subject disposition | 9 | 89 |
| | 4.1.2 | Protocol deviations and eligibility | 7 | 71 |
| | 4.1.3 | Demographic and other baseline characteristics | 7 | 74 |
| | 4.1.4 | Medical history and concomitant diseases | 80 | 81 |
| | 4.1.5 | Prior and concomitant therapies | 8 | 83 |
| | 4.1.6 | Comments | 8 | 85 |
| | 4.1.7 | Exposure to challenge agent | 8 | 98 |
| 4.2 | Pharm | Pharmacodynamics | 8 | 87 |
| 4.3 | Safety | | 6 | 06 |
| | 4.3.1 | Adverse events | 6 | 06 |
| | 4.3.2 | Physical examinations | 6 | 95 |
| | 4.3.3 | Clinical laboratory evaluation | 6 | 96 |

| MM | V_PfSPZ-L | MMV_PfSPZ-DVI Blood Stage_19_01 | Mock Tables, Listings and Figures | Final 1.0 of 11FEB2021 | 021 |
|---|---|---|---|---|---|
| | 4.3.4 | 4.3.4 Vital signs | | | 26 |
| | 4.3.5 | ECG | | | 86 |
| | 4.3.6 | 4.3.6 Malaria clinical score | | 1 | 101 |
| S | Template figures | figures | | 1 | 103 |
| 5.1 | Pharma | Pharmacodynamics | | 1 | 103 |
| 5.2 | Safety | | | 1 | 111 |
| | 5.2.1 | Clinical laboratory evaluation | | 1 | 111 |
| | 5.2.2 | Vital signs | | 1 | 113 |
| | 5.2.3 | ECG | | 1 | 114 |
| | 5.2.4 | 5.2.4 Malaria clinical score | | 1 | 115 |

### TABLE 14.1.2.6: PRIOR AND CONCOMITANT THERAPIES BY ATC CLASS (LEVEL 4) AND GENERIC TERM.......................32 TABLE 14.1.2.1: DEMOGRAPHIC DATA 27 TABLE 14.1.2.4: MEDICAL HISTORY 31 IABLE 14.1.1.2: FIRST AND LAST CONTACT IN THE STUDY. TABLE 14.1.1: ANALYSIS SETS..... TABLE OF CONTENTS OF THE TABLES General Characteristics

## 1.1.2 Pharmacodynamics

TABLE 14.1.2.8; ANTIMALARIAL TREATMENT DISCONTINUATION 34

| 38 | STATISTICS |
|---|---|
| | TABLE 14.2.3.4.1: PARASITAEMIA AT THE TIME OF ≥5000 PARASITES PER mL BLOOD (PARASITES/mL): DESCRIPTIVE |
| 37 | TABLE 14.2.3.3.1: TIME TO PARASITAEMIA OF≥5000 PARASITES PER mL BLOOD (DAYS): KAPLAN MEIER ESTIMATES37 |
| 36 | TABLE 14.2.3.2.1: PARASITAEMIA AT FIRST PCR POSITIVITY (PARASITES/mL): DESCRIPTIVE STATISTICS36 |
| 36 | TABLE 14.2.3.1.1: TIME TO FIRST PCR POSITIVITY (DAYS): DESCRIPTIVE STATISTICS |

| RED TERM. 55 | TABLE 14.3.1.6: PfSPZ INOCULUM RELATED ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM. 55 |
|---|---|
| RM 55 | TABLE 14.3.1.5: GRADE 3 OR MORE ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM55 |
| 54 | TABLE 14.3.1.4: SERIOUS ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM |
| 53 | TABLE 14.3.1.3: ADVERSE EVENTS BY MEDDRA PREFERRED TERM BY DESCENDING ORDER OF FREQUENCY |
| 52 | TABLE 14.3.1.2: ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM |
| 51 | TABLE 14.3.1.1: ADVERSE EVENTS OVERVIEW |
| | Adverse events |
| 50 | TABLE 14.2.3.15.1: DESCRIPTIVE STATISTICS OF LOG10(PARASITAEMIA) ACTUAL VALUES |
| § <del>**</del> ********************************** | TABLE 14.2.3.14.1: BLOOD-STAGE PARASITE CLEARANCE PROFILE: DESCRIPTIVE STATISTICS |
| .S47 | TABLE 14.2.3.13.1: BLOOD-STAGE PARASITE CLEARANCE PROFILE: INDIVIDUAL LOG-LINEAR MODEL ESTIMATES |
| DIVIDUAL46 | TABLE 14.2.3.12.1: BLOOD-STAGE PARASITE PROFILE: MODEL DERIVED PARAMETERS BASED ON SIMULATED INDIVIDUAL PARAMETER VALUES |
| ARAMETER 45 | TABLE 14.2.3.11.1: BLOOD-STAGE PARASITE PROFILE: MODEL DERIVED PARAMETERS BASED ON INDIVIDUAL PARAMETER ESTIMATES |
| 44 | TABLE 14.2.3.10.1: BLOOD-STAGE PARASITE PROFILE: MODEL DERIVED POPULATION PARAMETERS |
| 42 | TABLE 14.2.3.9.1: BLOOD-STAGE PARASITE PROFILE: EXTENDED LOG-LINEAR MIXED MODEL ESTIMATES |
| 40 | TABLE 14.2.3.8.1: BLOOD-STAGE PARASITE PROFILE: LOG-LINEAR MIXED MODEL ESTIMATES |
| 39 | TABLE 14.2.3.7.1: INCIDENCE OF PARASITAEMIA |
| STATISTICS. 38 | TABLE 14.2.3.6.1: PARASITAEMIA AT FIRST DOSE OF TREATMENT WITH RIAMET (PARASITES/mL): DESCRIPTIVE STATISTICS.38 |
| 38 | TABLE 14.2.3.5.1: TIME TO FIRST DOSE OF TREATMENT WITH RIAMET (DAYS): DESCRIPTIVE STATISTICS |

| 'ABLE 14.3.4.1: DESCRIPTIVE STATISTICS OF ECG |
|---|
| 1.1.6 ECG |
| ABLE 14.3.3.2: CROSS-TABULATION OF VITAL SIGNS ABNORMALITIES VERSUS BASELINE |
| ABLE 14.3.3.1: DESCRIPTIVE STATISTICS OF VITAL SIGNS |
| 1.1.5 Vital signs |
| ABLE 14.3.2.3: LIVER ENZYME ELEVATION CATEGORIES |
| ABLE 14.3.2.2: CROSS-TABULATION OF LABORATORY ABNORMALITIES VERSUS BASELINE |
| ABLE 14.3.2.1: DESCRIPTIVE STATISTICS OF LABORATORY TEST RESULTS |
| YABLE 14.3.1.11: ADVERSE EVENTS OF SPECIAL INTEREST RELATED TO ANTIMALARIAL TREATMENT BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM |
| ABLE 14.3.1.10: ADVERSE EVENTS OF SPECIAL INTEREST RELATED TO PFSPZ INOCULUM BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM |
| ABLE 14.3.1.9: ADVERSE EVENTS FOR WHICH THE ANTIMALARIAL TREATMENT WAS DISCONTINUED BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM |
| 'ABLE 14.3.1.8: SERIOUS PFSPZ INOCULUM RELATED ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM |
| ABLE 14.3.1.7: ANTIMALARIAL TREATMENT RELATED ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM |

| 1 |
|----------------------|
| 0 |
| 19 |
| Stage_ |
| <b>7</b> 2 |
| looc |
| $\mathbf{B}$ |
| $\overline{\Lambda}$ |
| Ģ. |
| PZ. |
| PfSPZ-DVI Blo |
| > |
| $\geq$ |
| = |
| $\overline{}$ |

## Mock Tables, Listings and Figures

| TABLE 1 | TABLE 14.3.4.2: CROSS-TABULATION OF ECG ABNORMALITIES VERSUS BASELINE | 33 |
|---|---|---|
| TABLE 1 | TABLE 14.3.4.3: TABULATION OF QTC CHANGE ABNORMALITIES | 4 |
| 1.1.7 | Malaria clinical score | |
| TABLE 1 | TABLE 14.3.5.1: DESCRIPTIVE STATISTICS OF MALARIA CLINICAL SCORE | 55 |
| TABLE 1 | TABLE 14.3.5.2: FREQUENCY TABLE OF THE WORST-CASE INDIVIDUAL MALARIA SIGNS AND SYMPTOMS66 | 99 |

## 2 TABLE OF CONTENTS OF THE LISTINGS

## 1.2.1 General Characteristics

| LISTING 16.2.1.1: ALLOCATION | . 68 |
|--------------------------------------------------------------------|------|
| LISTING 16.2.1.2: ANALYSIS PHASES | 69 |
| LISTING 16.2.1.3: STUDY AND ANTIMALARIAL TREATMENT DISCONTINUATION | 70 |
| LISTING 16.2.2.1: MAJOR PROTOCOL DEVIATIONS | . 71 |
| LISTING 16.2.2.2: VIOLATIONS ON ELIGIBILITY CRITERIA | . 72 |
| LISTING 16.2.2.3: NO-INOCULATED SUBJECTS | . 73 |
| LISTING 16.2.4.1: DEMOGRAPHIC DATA | 74 |
| LISTING 16.2.4.2: SMOKING HISTORY | . 75 |
| LISTING 16.2.4.3: ORTHOSTATIC CHANGE IN VITAL SIGNS AT SCREENING | . 76 |
| LISTING 16.2.4.4: BECK DEPRESSION INVENTORY AT SCREENING | . 77 |
| LISTING 16.2.4.5: SCREENING LABORATORY TESTS | 78 |
| LISTING 16.2.4.6: PREGNANCY TESTS | . 79 |
| LISTING 16.2.4.7: rRT-PCR TESTS FOR SARS-CoV-2 INFECTION | . 80 |
| LISTING 16.2.4.8: MEDICAL HISTORY | . 81 |
| LISTING 16.2.4.9: CONCOMITANT DISEASES | . 82 |
| LISTING 16.2.4.10: PRIOR AND CONCOMITANT THERAPIES | . 83 |
| LISTING 16.2.4.11: ANTIMALARIAL TREATMENT | . 84 |
| LISTING 16.2.4.12: COMMENTS | . 85 |

| LISTINC | LISTING 16.2.5.1: EXPOSURE TO CHALLENGE AGENT | 0 |
|---|---|---|
| 1.2.2 | Pharmacodynamics | |
| LISTING | LISTING 16.2.6.1: PARASITAEMIA | _ |
| LISTING | LISTING 16.2.6.2: PARASITAEMIA ENDPOINTS | $\sim$ |
| LISTING | LISTING 16.2.6.3: BLOOD-STAGE PARASITE CLEARANCE PROFILE: ITERATION PROCESS TO DETERMINE THE OPTIMAL LOG-<br>LINEAR MODEL | $\overline{}$ |
| 1.2.3 | Adverse events | |
| LISTING | LISTING 16.2.7.1: ADVERSE EVENTS | |
| LISTING | LISTING 16.2.7.2: SERIOUS ADVERSE EVENTS | |
| LISTING | LISTING 16.2.7.3: FATAL ADVERSE EVENTS | $\sim$ 1 |
| LISTING | LISTING 16.2.7.4: ADVERSE EVENTS FOR WHICH THE STUDY WAS DISCONTINUED92 | $\sim$ 1 |
| LISTING | LISTING 16.2.7.5: ADVERSE EVENTS FOR WHICH THE ANTIMALARIAL TREATMENT WAS DISCONTINUED92 | <b>~</b> 1 |
| LISTING | LISTING 16.2.7.6: ADVERSE EVENTS AFTER ADMINISTRATION OF ANTIMALARIAL TREATMENT92 | <b>~</b> 1 |
| LISTING | LISTING 16.2.7.7: ADVERSE EVENTS FOR WHICH ANOTHER ACTION IS TAKEN93 | ~ |
| LISTING | LISTING 16.2.7.8: ADVERSE EVENTS: CODING INFORMATION | <del></del> |
| LISTING | LISTING 16.2.7.9: PHYSICAL EXAMINATIONS ABNORMALITIES | 10 |
| 1.2.4 | Laboratory data | |
| LISTINC | LISTING 16.2.8.1: LABORATORY TEST RESULTS FOR SUBJECTS WITH ABNORMAL VALUES | |

| 1.2.5 | Vital signs |
|---|---|
| LISTING | LISTING 16.2.9.1: VITAL SIGNS RESULTS FOR SUBJECTS WITH ABNORMAL VALUES |
| 1.2.6 ECG | ECG |
| <b>LISTING</b> | LISTING 16.2.10.1: ECG RESULTS FOR SUBJECTS WITH ABNORMAL VALUES |
| LISTING | LISTING 16.2.10.2: ECG INTERPRETATION AND MORPHOLOGY FOR SUBJECTS WITH ANY ABNORMAL INTERPRETATION 100 |
| 1.2.7 | Malaria clinical score |
| LISTING | LISTING 16.2.11.1: MALARIA SIGNS AND SYMPTOMS |
| <b>LISTING</b> | LISTING 16.2.11.2: MALARIA CLINICAL SCORES > 6 AND PARASITAEMIA |

## 1.3 TABLE OF CONTENTS OF THE FIGURES

## 1.3.1 Pharmacodynamics

| FIGURE 14.2.3.1.1: BLOOD-STAGE PARASITE PROFILE: MEDIAN PARASITAEMIA ACTUAL VALUES OVER TIME |
|---|
| FIGURE 14.2.3.2.1: BLOOD-STAGE PARASITE PROFILE: INDIVIDUAL PARASITAEMIA ACTUAL VALUES OVER TIME 106 |
| FIGURE 14.2.3.3.1: TIME TO FIRST PCR POSITIVITY: KAPLAN MEIER PLOT |
| FIGURE 14.2.3.4.1: TIME TO PARASITAEMIA OF ≥5000 PARASITES PER mL BLOOD: KAPLAN MEIER PLOT |
| FIGURE 14.2.3.5.1: TIME TO FIRST DOSE OF TREATMENT WITH RIAMET: KAPLAN MEIER PLOT |
| FIGURE 14.2.3.6.1: TIME TO PARASITE CLEARANCE: KAPLAN MEIER PLOT |

### 1.3.2 Laboratory data

| _ | |
|---------------------------------------------------|---|
| : | |
| (ד) | |
| 1F | |
| $\leq$ | |
| YY TEST ACTUAL VALUES OVER TIME. | |
| $\simeq$ | |
| H) | |
| $\geq$ | |
| $\circ$ | |
| S | |
| H | |
| 7 | |
| A | |
| $\geq$ | |
| | ı |
| $\triangleleft$ | ĺ |
| È | |
| 9 | |
| SE | |
| > | ١ |
| O | |
| $\leq$ | |
| K | |
| BC | ۱ |
| ٨ | |
| 1 | ĺ |
| | l |
| $\forall$ | ĺ |
| | ١ |
| 5 | |
| $\leq$ | |
| <u></u> | |
| 2 | |
| 3 | |
| <del>\ \ </del> | |
| 7 | |
| [I] | |
| $\simeq$ | |
| Ę | |
| 9 | |
| r- | |
| | ١ |

### 1.3.3 Vital signs

| 13 |
|-------------------------------------|
| — |
| i |
| : |
| i |
| : |
| : |
| : |
| S ACTUAL VALUES OVER TIME |
| : |
| : |
| : |
| : |
| i |
| : |
| : |
| ACTUAL VALUES OVER TIME |
| eq |
| 出 |
| $\geq$ |
| $\circ$ |
| S |
| 5 |
| $\Box$ |
| $\leq$ |
| A |
| $\Box$ |
| Ę |
| 7 |
| S |
| Ż |
| 9 |
| S |
| ٦ |
| $\frac{1}{1}$ |
| $\leq$ |
| $\Gamma$ |
| IAL |
| $\geq$ |
| $\prod$ |
| Ž |
| P |
| $\leq$ |
| $\vdots$ |
| ώ. |
| $\tilde{\omega}$ |
| 14 |
| IGURE 14.3.3.1: INDIVIDUAL VITAL SI |
| $\mathbb{R}$ |
| 3 |
| ĭ |
| _ |

### 1.3.4 ECG

| _ | 1 |
|---|---|
| _ | 117 |
| _ | _ |
| | : |
| | • |
| | : |
| Ľ | : |
| Ĺ | 15: |
| 117 | ME: |
| TAAT | |
| TIME | I IIME |
| מועד מ | K HIME |
| חיוד מיו | EK LIME |
| חאוד מחי | VEK LIME |
| מאמד ממער | JVEK LIME |
| TAUT GENT | OVER LIME |
| TAME GENERAL | SOVER LIME |
| THE CHANGE | ESOVEK LIME |
| THE OTHER PARTY | OES OVER LIME |
| THE OWNER THE | LUES OVER IIME |
| ATTES OTTES | ALUES OVER LIME |
| TATT GAMES OF TAKE | VALUES OVER I IIVIE |
| TATTER OXIED THAT | VALUES OVER LIME |
| TATTER OVER THAT | L VALUES OVER IIME |
| TAT THE CAME TAY | AL VALUES OVER LIME |
| TAT VALITES OVER TAIL | OAL VALUES OVER LIME |
| TATT TATTER OTTER | I UAL VALUES UVER I IIME |
| THAT THE OTHER PARTY | OIOAL VALUES OVER HIME |
| THE THE TAILED OFFER THE | ACTUAL VALUES OVER TIME |
| TATTO | ACTOAL VALUES OVER TIME |
| TATTO | G ACTOAL VALUES OVER TIME |
| TATTO | OR ACTORE VALUES OVER TIME |
| TATTO | JOG ACTOAL VALUES OVER TIME |
| TATTO | ECG ACTOAL VALUES OVER TIME |
| TATTO | LECGACIOAL VALUES OVER HIME |
| TATTO | AL ECG ACTUAL VALUES UVER TIME |
| TATTO | OAL ECG ACTOAL VALUES OVER TIME |
| TATTO | JOAL ECG ACTOAL VALUES OVER TIME |
| TATTO | IDOAL ECG ACTOAL VALUES OVER TIME |
| TATTO | VIDUAL ECG ACTUAL VALUES UVER TIME |
| TATTO | IVIDUAL ECG ACTOAL VALUES OVER TIME |
| TATTO | IVIDUAL ECG ACTUAL VALUES UVEK I |
| TATTO | NDIVIDUAL ECG ACTUAL VALUES OVER TIME |
| TATTO | IVIDUAL ECG ACTUAL VALUES UVEK I |
| TAIL TO STITLE TO A CTITAL VIALITIES OF TAIL THE | IVIDUAL ECG ACTUAL VALUES UVEK I |
| TATTO | IVIDUAL ECG ACTUAL VALUES UVEK I |
| TATTO | IVIDUAL ECG ACTUAL VALUES UVEK I |
| A 1. TAIL TAIL ECO A CITTAI | IVIDUAL ECG ACTUAL VALUES UVEK I |
| A 1. TAIL TAIL ECO A CITTAI | IVIDOAL ECG ACTOAL VALUES OVER I |
| A 1. TAIL TAIL ECO A CITTAI | IVIDOAL ECG ACTOAL VALUES OVER I |
| TATTO | IVIDOAL ECG ACTOAL VALUES OVER I |
| A 1. TAIL TAIL ECO A CITTAI | IVIDUAL ECG ACTUAL VALUES UVEK I |
| A 1. TAIL TAIL ECO A CITTAI | IVIDUAL ECG ACTUAL VALUES UVEK I |

## 1.3.5 Malaria clinical score

| FIGURE 14.3.5.1: INDIVIDUAL MALARIA CLINICAL SCORE ACTUAL VALUES OVER TIME | FIGURE 14.3.5.2: INDIVIDUAL MALARIA CLINICAL SCORE AND PARASITAEMIA ACTUAL VALUES OVER TIME | FIGURE 14.3.53: INDIVIDITAL MALARIA CLINICAL SCORE AND CRP ACTITAL VALUES OVER TIME |
|---|---|---|
| FIGURE 14.3.5.1: INDIVIDUAL MALARIA CLINIC | FIGURE 14.3.5.2: INDIVIDUAL MALARIA CLINIC | FIGURE 14353: INDIVIDITAL MALARIA CLINIC |

## **GENERAL LAYOUT OF A TLF**

### SOFTWARE USED

SAS version 9.4 or later will be used for programming. TLFs will be transferred to MS WORD.

## LAYOUT SPECIFICATIONS IN SAS

SAS TITLE1, left will identify the project by Sponsor protocol number. In case of a blinded testrun, the analysis version will be added, or a note that fake treatments were used.

SAS TITLE1, right will show the SAS datetime stamp of the table creation (batch submit datetime).

SAS TITLE2 will present the page numbering, right aligned, in the format "PAGE X OF Y"

SAS TITLE3 will contain the TLF's identification in the form TABLE 14.x.x.x, LISTING 16.2.x.x and FIGURE 14.x.x.x followed by the title. The title itself and the TLF number are copied from the SAP.

SAS TITLE4 will draw a horizontal dotted line ("-----") over the entire width of the page.

SAS TITLE5 will show the analysis population.

SAS TITLE6 through 10 may be used to provide further information, when deemed useful.

Example:

```
SAS DATE AND TIME PAGE X OF Y
1 STUDY IDENTIFIER - ANALYSIS VERSION
                                      3 TABLE 14.x.x.x: <TABLE TITLE>
                                                                        5 POPULATION: ALL SUBJECTS 6 7
```

Footnotes will be added in SAS, as deemed appropriate by the programmer. Footnotes will be used to improve the readability of the output. Output will be left-aligned and all text will be in CAPITALS, except for specific test units.

The following SAS page setup will be used:

- LSIZE = 139
- PSIZE = 43

Dates are formatted using the SAS date9. format: ddMMMyyyy . E.g., 16SEP1970.

The format of times follows a 24h clock as hh:mm, from 00:00 till 23:59. 24:00 equals 00:00 on the next day.

Datetime fields are formatted using the SAS datetime 13. or datetime 15. format: ddMMMyyyy:hh:mm

## LAYOUT SPECIFICATIONS IN MS WORD

All tables and listings will be generated in ASCII text files by SAS, and then converted into MS Word documents, using font COURIER NEW 8pt. (like in these Mock TLFs).

Page layout:

landscape

• paper size: A4

| <ul> <li>margins in N</li> </ul> | margins in MS Word, in cm: |
|----------------------------------|----------------------------|
| Top | 3.2 |
| Bottom | 3.2 |
| Left | 2.2 |
| Right | 2.2 |
| Gutter | 0 |
| Header, from edge | 76.0 |
| Trates from ale | 700 |

| • margins in MS word, in cm: | is word, in cm: |
|------------------------------|-----------------|
| Тор | 3.2 |
| Bottom | 3.2 |
| Left | 2.2 |
| Right | 2.2 |
| Gutter | 0 |
| Header, from edge | 76.0 |
| Footer, from edge | 0.94 |


## CENERAL TABLE LAYOUT

# Standard layout for descriptive statistics on continuous parameters

Use of decimal places in descriptive statistics:

- Mean, geometric mean, median, SD, geometric SD and CI will be presented with one more decimal place than the individual values.
- Minimum, maximum and range will be presented with the same number of decimal places than the individual values.
- P-values will be presented with four decimal places, ratios with three decimal places and estimates and test statistics with two decimal

places.

| | g | Mean | S.<br>田.<br>日. | S.D. | 95% C.I. * | | Min | Median<br> | Max<br> |
|---|---|---|---|---|---|---|---|---|---|
| COHORT 1 (N=XX) | | | | | | | | | |
| SCREENING | X | xx.xx | XXX.XX | XX.XXX | (XX.XXX) | XX.XXX) | XX.XX | xxx.xx | xx.xx |
| BASELINE | × | XXX.XXX | XX.XX | XXX.XX | (XXX.XXX) | XX.XXX) | XX.XX | XXX.XXX | XX.XX |
| TIME POINT 3 | × | XXX.XXX | XX.XX | XXX.XX | (XXX.XXX) | XX.XXX) | XX.XX | XXX.XXX | XX.XX |
| TIME POINT 4 | × | XX.XXX | XX.XX | XX.XXX | (XX.XXX) | XX.XXX) | XX.XX | XXX.XXX | XX.XX |
| FOLLOW-UP | × | XXX.XX | XXX.XXX | XX.XXX | (XXX.XX) | XX.XXX) | XX.XX | XXX.XX | XX.XX |
| COHORT 2 (N=XX) | | | | | | | | | |
| SCREENING | × | XXX.XXX | XX.XX | XX.XXX | (XXX.XXX) | XX.XXX) | XX.XX | XXX.XX | XX.XX |
| BASELINE | × | XX.XXX | XXX.XX | XX.XXX | (XX.XXX) | XX.XXX) | XX.XX | XX.XXX | XX.XX |
| TIME POINT 3 | × | XX.XXX | XX.XX | XX.XXX | ٠. | XX.XXX) | XX.XX | XXX.XXX | XX.XX |
| TIME POINT 4 | × | XX.XXX | XX.XX | XX.XXX | (XX.XXX) | XX.XXX) | XX.XX | XXX.XXX | XX.XX |
| FOLLOW-UP | × | XX.XXX | XX.XX | XX.XXX | (XX.XX) | XX.XXX) | XX.XX | XX.XXX | XX.XX |
| Etc. | | | | | | | | | |

<sup>\*</sup> CONFIDENCE INTERVAL FOR MEAN


## .4.2 Standard layout for frequency tabulations

It is possible that the width of tables is too much to fit on one page (due to the number of treatments / columns). In that case, the page break will attempt to keep information of one treatment together. I.e., the break will not be made between "n" and "%".

Zero frequencies are shown, but classes that were not observed in any treatment or missing values, are not presented.

Percentages will be shown with 1 decimal place (xx.x%). It is allowed that "100.0%" is presented as "100%" to save space.

An example for a categorical variable:

| | COHORT (N-XY) | COHORT 1 | COHO | COHORT 2 | ALL SU | ALL SUBJECTS |
|---|---|---|---|---|---|---|
| PARAMETER AND CLASS | n n | Q % | Z C | N-02) | % U | 00 ov |
| | <br> | <br> | <br> <br> <br> <br> <br> | <br> <br> <br> <br> | <br> | <br> |
| CLASS 1 | ×× | XX.X | × | $\times \times \times$ | XX | XX.X |
| CLASS 2 | XX | XX.X | × | XX.X | XX | XX.X |
| TOTAL | XX | 100 | ×× | 100 | XX | 100 |
| PARAMETER 2 | | | | | | |
| CLASS 1 | XX | XX.X | × | XX.X | XX | xx.x |
| CLASS 2 | XX | XX.X | × | XX.X | XX | XX.X |
| CLASS 3 | XX | XX.X | × | XX.X | XX | XX.X |
| TOTAL | XX | 100 | × | 100 | ×× | 100 |
| PARAMETER 3 | | | | | | |
| CLASS 1 | XX | XX.X | × | XX.X | XX | XX.X |
| TOTAL | XX | 100 | × | 100 | XX | 100 |


## Standard layout for table containing descriptive statistics and frequency tabulations 2.4.3

In case a table contains descriptive statistics as well as tabulations (for example for demographic parameters), the following presentation will be

| (N=xx) (X | | | COHORT 1 | | COHORT 2 | AL | ALL SUBJECTS |
|---|---|---|---|---|---|---|---|
| XX XX.X (XX.X) XX.X XX.X XX.X XX.X XX.X XX.X XX. | | | (N=XX) | | (N=XX) | | (N=XX) |
| XX | ER 1 (unit) | <br> | <br> | | <br> | | <br> |
| XXX (XX.X) XXX (XX.X; XX.X) XXX (XX.X; XX.X) XXX XX | | XX | | X | | XX | |
| X.X (XX.X; XX.X) (XX.X; XX.X) (XX.X; (XX,X) (XX,X; (XX,X) (XX,X) (XX,X; (XX,X) (XX,X; (XX,X) (XX,X; (XX,X) (XX,X; (XX,X) (XX,X) (XX,X; (XX,X) (XX,X; (XX,X) (XX,X) (XX,X; (XX,X) (XX,X) (XX,X; (XX,X) (XX,X) (XX,X; (XX,X) (XX,X) (XX,X) (XX,X) (XX,X; (XX,X) | (S.D) | XX. | (XX.XX) X | XX | (XXXX) X | XX | XX.X (XX.X) |
| (XX.X, XX.X) (XX.X, XX.X) (XX.X, XX.X) (XX.X, XX.X) (XX.X, XX.X) (XX.X, XX.X, XX.X) (XX.X, XX.X, XX.X, XX.X) (XX.X, XX.X, XX.X | | × | × | × | × | × | × |
| XX | . H. | (XX) | X; XX.X) | (XX | X; XX.X) | (XX) | (XX.X; XX.X) |
| (XX; XX) (XX; XX) XX XX.X (XX.X) XX.X (XX.X) XX.X (XX.X; XX.X) (XX.X; XX.X) XX.X (XX; XX) (XX; XX) XX XX.X (XX; XX) XX XX.X XX XX.X XX XX.X XX.X XX XX.X XX.X XX.X XX.X XX.X XX XX.X XX.X XX.X XX.X XX.X XX.X XX XX.X XX.X XX.X XX.X XX.X XX.X XX XX.X XX XX.X | an | XX. | × | XX. | × | XX | × |
| XX XX.X (XX.X) XX.X XX.X (XX.X; XX.X) XX.X (XX.X; XX.X) (XX.X; XX.X) (XX; XX) (XX; XX) (XX; XX) XX XX.X XX XX XX.X XX XX XX.X XX XX XX.X XX | Max | (XX) | XX) | (XX); | XX) | (XX) | XX) |
| XX | ER 2 (unit) | | | | | | |
| b) x.x (xx.x) x.x (xx.x)<br>x.x | | XX | | X | | XX | |
| * (XX.X; XX.X) (XX.X; XX.X) (XX.X; XX.X) (XX.X; XX.X) (XX; XX) (XX; XX) (XX; XX) (XX; XX.X; XX.X | (S.D) | XX | (XX.XX) X | XX | (XXXX) X | XX | XX.X (XX.X) |
| * (XX.X; XX.X) (XX.X; XX.X) XX.X (XX; XX) (XX; XX) XX XX.X XX XX XX.X XX XX XX XX.X XX X | | × | × | × | × | × | × |
| XX.X (XX, XX) (XX, XX) (XX, XX) (XX, XX) (XX, XX, | | (XX | X; XX.X) | (XX) | X; XX.X) | (XX) | (XX.X; XX.X) |
| (xx; xx) (xx; xx) (xx; xx) xx xx.x xx xx.x xx.x xx.x xx.x xx. | an | XX | × | ×× | × | XX | × |
| XX XX.X XX.X XX.X XX.X XX.X XX.X XX.X | Max | (XX) | (XX) | (XX) | (XX) | (XX) | (XX) |
| XX XX.X XX.X XX.X XX.X XX.X XX.X XX.X | ER 3 | | | | | | |
| XX XX.X XX XX.X XX | S 1 | × | XX.X | × | XX.X | × | XX.X |
| XX 100 XX 100 XX X | S 2 | × | XX.X | × | XX.X | × | XX.X |
| XX XX.X XX.X XX.X XX.X XX.X XX.X XX.X | H. | × | 100 | XX | 100 | XX | 100 |
| 1 | ER 4 | | | | | | |
| XX XX.X XX XX.X XX | S 1 | X | XX.X | × | XX.X | X | XX.X |
| XX 100 XX 100 XX | s 2 | X | XX.X | × | XX.X | X | XX.X |
| | Г | × | 100 | X | 100 | X | 100 |


<sup>\*</sup> CONFIDENCE INTERVAL FOR MEAN THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET, EXCLUDING MISSING VALUES.

## Standard layout of an analysis table of contents

Per section of the analysis a table of contents is created automatically. Below an example:

STUDY IDENTIFIER - ANALYSIS VERSION

SAS DATE AND TIME

TABLE 14.1.1.1: SUBJECT DISPOSITION: TABULATION OF THE STUDY TERMINATION
TABLE 14.1.1.2: SUBJECT DISPOSITION: TABULATION OF THE NUMBER OF SUBJECTS IN EACH ANALYSIS POPULATION
LISTING 16.2.1.2: SUBJECT DISPOSITION: STUDY TERMINATION LISTING 16.2.1.4: SUBJECT DISPOSITION: OVERALL LISTING OF VISITS AND ASSESSMENTS LISTING 16.2.1.5: SUBJECT DISPOSITION: ELIGIBILITY CRITERIA - VIOLATIONS LISTING 16.2.1.6: SUBJECT DISPOSITION: ELIGIBILITY CRITERIA - EXEMPTIONS LISTING 16.2.1.7: SUBJECT DISPOSITION: PROTOCOL DEVIATIONS LISTING 16.2.1.8: SUBJECT DISPOSITION: NO-TREATMENT SUBJECTS LISTING 16.2.1.9: SUBJECT DISPOSITION: COMMENTS LISTING 16.2.2.3: DEMOGRAPHIC DATA: MEDICAL HISTORY ABNORMALITIES LISTING 16.2.2.4: DEMOGRAPHIC DATA: CONCOMITANT DISEASES LISTING 16.2.2.5: PHYSICAL EXAMINATIONS LISTING 16.2.1.3: SUBJECT DISPOSITION: STUDY ANALYSIS PERIODS LISTING 16.2.2.1: DEMOGRAPHIC DATA: DEMOGRAPHIC PARAMETERS TABLE 14.1.2.1: DEMOGRAPHIC DATA: DESCRIPTIVE STATISTICS LISTING 16.2.1.10: USE OF STUDY MEDICATION: ACTUAL DATA LISTING 16.2.2.2: DEMOGRAPHIC DATA: SCREENING TESTS LISTING 16.2.1.1: SUBJECT DISPOSITION: ALLOCATION DISPLAY / LISTING TABLE OF CONTENTS


## S GENERAL FIGURE LAYOUT

Please be aware that all graphs shown in this document are mock-graphs. Points, lines, axes and legends are not always study specific and are therefore described explicitly below each graph.

### General programmer notes:

- Figures should be made at a high resolution and with an easily readable font size for legend and axis labels and values.
- Markers and lines should be of sufficient size and width.
- Labels of X- and Y-axis will be centred.
- Colours, line types and symbols should be used in a consistent way throughout the analysis.
- Colours, line types and symbols should be used keeping in mind figures are often printed in grey scale.

 document
#### 3. MOCK TABLES

#### GENERAL CHARACTERISTICS

#### Subject disposition

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

SAS DATE AND TIME PAGE X OF Y

TABLE 14.1.1.1: ANALYSIS SETS

ANALYSIS SET: ALL SCREENED SUBJECTS

ALL SUBJECTS XX XX 100 XX XX.X XX.X % U COHORT 2 n % ALL SCREENED SUBJECTS SET
SAFETY ANALYSIS SET
PHARMACODYNAMICS ANALYSIS SET
XX XX.X
MODIFIED PHARMACODYNAMICS ANALYSIS SET
XX XX.X COHORT 1 n % ANALYSIS SET

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET.


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.1.1.2: FIRST AND LAST CONTACT IN THE STUDY

ANALYSIS SET: ALL SCREENED SUBJECTS

ddMMMYYYY ddMMMyyyy ddMMMyyyy DATE OF FIRST ICF (1):
DATE OF LAST VISIT (2):
DATE OF LAST CONTACT (3):

NOTES: (1): SIGNATURE DATE ON THE INFORMED CONSENT FORM OF THE FIRST SUBJECT. (2): DATE OF THE LAST VISIT IN THE STUDY (INCLUDING UNSCHEDULED VISITS). (3): LAST DATE OF CONTACT WITH ANY SUBJECT IN THE STUDY.


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

MMV\_PfSPZ-DVI Blood Stage\_19\_01

TABLE 14.1.1.3: STUDY DISCONTINUATION

ANALYSIS SET: SAFETY

| | COH | COHORT 1 | COH | ORT 2 | AT.T. S | ALI, SUBJECTS |
|---|---|---|---|---|---|---|
| | = N) | XX) | = Z) | (N=XX) | =N) | (N=XX) |
| SUBJECT STATUS | Д | . %<br>. % | , u | 0/0 | % ۵ | 0/0 |
| | | | 1 1 1 1 1 1 | | 1 1 1 1 1 1 1 | |
| COMPLETED | XX | x.x. | XX | XX XX.X | XX | XX.X |
| DISCONTINUED | X | xx.x | XX | x.x. | XX | XX.X |
| ADVERSE EVENT | × | XX.X | XX | xx.x | XX | XX.X |
| SUBJECT LOST TO FOLLOW-UP | X | XX.X | ×× | xx.x | XX | XX.X |

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET.

## Protocol deviations and eligibility

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.1.1.4: MAJOR PROTOCOL DEVIATIONS

ANALYSIS SET: SAFETY

| ALL SUBJECTS (N=XX) | | xx xx xx | xxx xx | x.xx xx | xx xx.x |
|---|---|---|---|---|---|
| COHORT 2 (N=XX) | ₩<br>₩ | XX XX.X | XX XX.X | XX XX.X | XX XX.X |
| COHORT 1 (N=XX) | %<br>Cl | XX XX.X | XX XX.X | XX XX.X | XX XX.X |
| | ESENCE AND CLASS | NO MAJOR DEVIATIONS | ANY MAJOR DEVIATION | FORBIDDEN THERAPY | PROCEDURE DEVIATION |

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET.


# Demographic and other baseline characteristics

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.1.2.1: DEMOGRAPHIC DATA

ANALYSIS SET: SAFETY

| ALL SUBJECTS (N=XX) | XX<br>XX.X (X.X)<br>XX.X<br>(XX, XX) | XX<br>XX.X (X.X)<br>XX.X (XX) | XX<br>XX.X (X.X)<br>XX.X (XXX) | xx<br>xx.x (x.x)<br>xx.x (xx,x) | xx xx.x<br>xx xx.x<br>xx 100 | XX |
|---|---|---|---|---|---|---|
| COHORT 2<br>(N=XX) | XX<br>XX.X (X.X)<br>XX.X<br>(XX, XX) | xx<br>xx.x (x.x)<br>xx.x (xx,x) | xx<br>xx.x (x.x)<br>xx.x (xx.x) | xx<br>xx.x (x.x)<br>xx.x<br>(xx; xx) | XX XX.X<br>XX XX.X<br>XX 100 | XX XX.X<br>XX.X XX.X |
| COHORT 1 (N=XX) | XX<br>XX.X (X.X)<br>XX.X<br>(XX, XX) | xx<br>xx.x (x.x)<br>xx.x<br>(xx, xx) | (kg)<br>xx<br>xx.x (x.x)<br>xx.x<br>(xx, xx) | (kg/m²) | XX XX.X<br>XX XX.X<br>XX 100 | XX |
| | AGE (years) n Mean (S.D.) Median Min; Max | HEIGHT (cm) n Mean (S.D.) Median Min; Max | WEIGHT AT SCREENING<br>n<br>Mean (S.D.)<br>Median<br>Min; Max | BMI AT SCREENING (kg<br>n<br>Mean (S.D.)<br>Median<br>Min; Max | SEX (n %)<br>FEMALE<br>MALE<br>TOTAL | RACE (n %)<br>BLACK<br>CAUCASIAN/WHITE<br>TOTAL |


| | XX.X | XX.X | 100 | | XX.X | XX.X | XX.X | 100 |
|---|---|---|---|---|---|---|---|---|
| | ×× | ×× | XX | | XX | ×× | ×× | ×× |
| | XX.X | x.xx | 100 | | XX.X | XX.X | XX.X | 100 |
| | XX | ×× | XX | | XX | XX | XX | ×× |
| | XX.X | x.x. | 100 | | xx.x | xx.x | XX.X | 100 |
| _ | TINO XX | C/LATINO XX | ×× | (n %) | | XX | | |
| ETHNICITY (n % | HISPANIC/LA | NOT HISPANI | TOTAL | SMOKING STATUS (n | EX-SMOKER | NON-SMOKER | SMOKER | TOTAL |

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET, EXCLUDING MISSING VALUES.

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.1.2.2: ORTHOSTATIC CHANGE IN VITAL SIGNS AT SCREENING

ANALYSIS SET: SAFETY

SYSTOLIC BLOOD PRESSURE (mmHg)

| ALL SUBJECTS (N=XX) | XX<br>XX.X (X.X)<br>XX.X<br>(XX, XX) | XX<br>XX.X (X.X)<br>XX.X<br>(XX, XX) | XX<br>XX.X (X.X)<br>XX.X<br>(XX, XX) |
|---|---|---|---|
| COHORT 2<br>(N=XX) | XX<br>XX.X (X.X)<br>XX.X<br>(XX, XX) | XX<br>XX.X (X.X)<br>XX.X<br>(XX, XX) | XX<br>XX.X (X.X)<br>XX.X<br>(XX, XX) |
| COHORT 1 (N=XX) | XX<br>XX.X<br>XX.X<br>(XX, XX) | XX XXX | XX<br>XX.X (X.X)<br>XX.X<br>(XX, XX) |
| | SUPINE RESULT<br>n<br>Mean (S.D.)<br>Median<br>Min; Max | STANDING RESULT n Mean (S.D.) Median Min; Max | ORTHOSTATIC CHANGE n Mean (S.D.) Median Min; Max |

ORTHOSTATIC CHANGE = VALUE IN SUPINE POSITION - VALUE IN STANDING POSITION.

Programmer notes: repeat the table by parameter: systolic blood pressure, diastolic blood pressure and heart rate.

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.1.2.3: BECK DEPRESSION INVENTORY AT SCREENING

ANALYSIS SET: SAFETY

| | HOO<br>N) | COHORT 1 (N=XX) | COH<br>(N) | COHORT 2 (N=XX) | ALL SUBJ<br>(N=XX) | ALL SUBJECTS (N=XX) |
|---|---|---|---|---|---|---|
| BECK DEPRESSION INVENTORY TOTAL SCORE | | | | | | |
| | XX | | XX | | × | |
| Mean (S.D.) | XX. | (X.X) X | XX. | (X.X) X | XX | (X.X) |
| Median | XX. | XX.X | XX. | × | XX | × |
| Min; Max | (XX) | (XX; XX) | (XX) | (XX; XX) | (XX) | (XX; XX) |
| BECK DEPRESSION INVENTORY INTERPRETATION | | | | | | |
| NORMAL | ×× | XX.X | XX | XX.X | × | XX.X |
| MILD MOOD DISTURBANCE | XX | XX.X | XX | XX.XX | × | XX.X |
| BORDERLINE CLINICAL DEPRESSION | XX | XX.X | × | XX.X | × | XX.X |
| | × | 100 | × | 100 | × | 100 |

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET, EXCLUDING MISSING VALUES.

SAS DATE AND TIME PAGE X OF Y


# Medical history and concomitant diseases

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.1.2.4: MEDICAL HISTORY

ANALYSIS SET: SAFETY

| SYSTEM ORGAN CLASS AND PREFERRED TERM | COH<br>(N= | COHORT 1<br>(N=XX)<br>n % | COH<br>(N= | COHORT 2<br>(N=XX)<br>n % | ALL SUBJ<br>(N=XX)<br>n % | ALL SUBJECTS (N=XX) |
|---|---|---|---|---|---|---|
| NO MEDICAL HISTORY FINDINGS | l XX | XXXXXXX | × | x.x | ×× | XX XX XX |
| WITH ANY MEDICAL HISTORY FINDING | XX | XX.X | XX | xx.x | XX | XX.X |
| EYE DISORDERS | XX | XX.X | XX | xx.x | XX | XX.X |
| CATARACT | XX | XX.X | XX | XX.X | XX | XX.X |
| GASTROINTESTINAL DISORDERS | ×× | XX.X | XX | ××.× | XX | XX.X |
| DUODENAL ULCER | XX | XX.X | ×× | ××.× | ×× | XX.X |
| UMBILICAL HERNIA | XX | XX.X | XX | ×.×× | ×× | XX.X |
| INFECTIONS AND INFESTATIONS | XX | XX.X | XX | XX.X | XX | XX.X |
| APPENDICITIS | ×× | XX.X | XX | ××.× | XX | XX.X |
| TUBERCULOSIS | XX | XX.X | ×× | x.xx | ×× | XX.X |

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET.

# Programmer notes: repeat similar table for concomitant diseases:

TABLE 14.1.2.5: CONCOMITANT DISEASES

## 3.1.5 Prior and concomitant therapies

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.1.2.6: PRIOR AND CONCOMITANT THERAPIES BY ATC CLASS (LEVEL 4) AND GENERIC TERM

SAS DATE AND TIME PAGE X OF Y

ANALYSIS SET: SAFETY

ANALYSIS PHASE = OVERALL

ALL SUBJECTS (N=XX)\* \* COHORT 2 (N=XX)ᅄ \* COHORT 1 (N=XX)q \* WITH THERAPIES TAKEN ATC CLASS (LEVEL 4) AND GENERIC TERM NO THERAPIES TAKEN ZOLMITRIPTAN CARDIAC THERAPY PARACETAMOL CAFFEINE IBUFROFEN ULTRACET

ANALYSIS PHASE = SCREENING

Etc.

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT AND PER ANALYSIS PHASE IN THE SAFETY SET.


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.1.2.7: ANTIMALARIAL TREATMENT

ANALYSIS SET: SAFETY

| ALL SUBJECTS (N=XX) n % | XX XX.X<br>XX XX.X<br>XX 100 | XX XX.X<br>XX XX.X<br>XX 100 |
|---|---|---|
| COHORT 2<br>(N=XX)<br>n % | xx xx.x<br>xx xx.x<br>xx 100 | xx xx.x<br>xx xx.x<br>100 |
| COHORT 1 (N=XX) n % | XX XX.X<br>XX XX.X<br>XX 100 | XX XX.X<br>XX XX.X<br>100 |
| | START OF ANTIMALARIAL TREATMENT PRIOR TO DAY 24 ON DAY 24 TOTAL | ANTIMALARIAL TREATMENT ADMINISTERED<br>MALARONE 250/100 mg<br>RIAMET 20/120 mg<br>TOTAL |

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET.

MMV\_PfSPZ-DVI Blood Stage\_19\_01

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.1.2.8: ANTIMALARIAL TREATMENT DISCONTINUATION

ANALYSIS SET: SAFETY

| ALL SUBJECTS (N=XX) | 0/0 | | XX.X | XX XX.X | XX.X | XX.X |
|---|---|---|---|---|---|---|
| ALL S<br>(N= | Ц | 1 1 1 1 1 | XX | XX | XX | XX |
| ХТ 2<br>Х) | 90 | | XX.X | x.xx | XX.X | xx.x |
| COHORT<br>(N=XX) | ū | 111111 | ×× | | XX | |
| ORT 1<br>(X) | 0/0 | | XX.XX | XX.X | XX.X | xx.x |
| COHORT<br>(N=XX) | Ц | | × | XX | | × |
| | SUBJECT STATUS | | STED | JISCONTINUED | ADVERSE EVENT | SUBJECT LOST TO FOLLOW-UP |
| | SUBJEC | 1 | COMPLETED | DISCON | ADV | SUE |

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET.


#### 3.2 PHARMACODYNAMICS

Programmer note: all PD tables shown in this section will be repeated for the m-PD analysis set with adjusted numbering (e.g. 14.2.3.1.2).

MMV\_PfSPZ-DVI Blood Stage\_19\_01

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.2.3.1.1: TIME TO FIRST PCR POSITIVITY (DAYS): DESCRIPTIVE STATISTICS

ANALYSIS SET: PD

Geom S.D. Min; Max XX.XXX; XX.XXX XX.XXX; XX.XXX XX.XXX; XX.XXX Geom. Mean 95% C.I. <a>  $\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}$ g ¦ ALL SUBJECTS (N=XX) COHORT 1 (N=XX) COHORT 2 (N=XX)

<a> TWO-SIDED 95% CONFIDENCE INTERVAL ON THE GEOMETRIC MEAN.
POSITIVE PARASITAEMIA IS DEFINED AS QPCR OUTCOME 2 250 PARASITES PER ML BLOOD.
ONLY SUBJECTS THAT REACHED POSITIVE PARASITAEMIA ARE INCLUDED.

# Programmer note: repeat Table 14.2.3.1.1 excluding the last footnote for:

TABLE 14.2.3.2.1: PARASITAEMIA AT FIRST PCR POSITIVITY (PARASITES/ml): DESCRIPTIVE STATISTICS


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

SAS DATE AND TIME PAGE X OF Y

TABLE 14.2.3.3.1: TIME TO PARASITAEMIA OF 25000 PARASITES PER ML BLOOD (DAYS): KAPLAN MEIER ESTIMATES

ANALYSIS SET: PD

| ALL SUBJECTS (N=XX) | XX.X (XX.X; XX.X)<br>XX.X (XX.X; XX.X)<br>XX.X (XX.X; XX.X) | × × × |
|---|---|---|
| | XX.X (XX.X; XX.X)<br>XXX (XX.X; XX.X)<br>XXX (XX.X; XX.X) | * * * |
| | XX.X (XX.X; XX.X)<br>XX.X (XX.X; XX.X)<br>XX.X (XX.X; XX.X) | × × × |
| | 25th QUANTILE (95% CI)<br>MEDIAN (95% CI)<br>75th QUANTILE (95% CI) | NUMBER ASSESSED<br>NUMBER CENSORED<br>NUMBER OF EVENTS <a></a> |

<sup>&</sup>lt;a> SUBJECTS WITH PARASITAEMIA OF 25000 PARASITES PER mL BLOOD.


## Programmer note: repeat Table 14.2.3.1.1 for:

TABLE 14.2.3.4.1: PARASITAEMIA AT THE TIME OF 25000 PARASITES PER ML BLOOD (PARASITES/ML): DESCRIPTIVE STATISTICS TABLE 14.2.3.6.1: PARASITAEMIA AT FIRST DOSE OF TREATMENT WITH RIAMET (PARASITES/ML): DESCRIPTIVE STATISTICS TABLE 14.2.3.5.1: TIME TO FIRST DOSE OF TREATMENT WITH RIAMET (DAYS): DESCRIPTIVE STATISTICS

In the previous tables the footnotes will be adapted accordingly.


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.2.3.7.1: INCIDENCE OF PARASITAEMIA

ANALYSIS SET: PD

PARASITES PER ML BLOOD <b 90% C.I. <c> PARASITAEMIA OF 25000 % U POSITIVE PARASITAEMIA <a> XX.X XX.X; XX.X XX.X XX.X; XX.X XX.X XX.X; XX.X 90% C.I. <c> % U  $\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}$ COHORT 1 (N=XX)
COHORT 2 (N=XX)
ALL SUBJECTS (N=XX) <a> INCIDENCE OF POSITIVE PARASITAEMIA BETWEEN INOCULATION WITH PESPZ AND DAY 28.
<b><b> INCIDENCE OF PARASITAEMIA OF >5000 PARASITES PER mL BLOOD BETWEEN INOCULATION WITH PESPZ AND DAY 28.
<>> TWO-SIDED 90% EXACT CLOPPER-PEARSON CONFIDENCE INTERVAL.


SAS DATE AND TIME PAGE X OF Y

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.2.3.8.1: BLOOD-STAGE PARASITE PROFILE: LOG-LINEAR MIXED MODEL ESTIMATES

| i |
|---|
| i |
| İ |
| I |
| ŀ |
| i |
| i |
| İ |
| ļ |
| i |
| i |
| i |
| I |
| i |
| i |
| i |
| İ |
| ļ |
| i |
| i |
| İ |
| i |
| ŀ |
| i |
| İ |
| i |
| ŀ |
| i |
| İ |
| ļ |
| ŀ |
| i |
| İ |
| ļ |
| ŀ |
| i |
| į |
| ŀ |
| ŀ |

ANALYSIS SET: PD

| PARAMETER | VALUE | RSE | SHRINKAGE | COMMENT |
|---|---|---|---|---|
| **Typical parameters**<br>GR<br>Finoc<br>Pinoc | | | 1 1 1 | Parasite growth rate (1/hour) Inoculum viability (-) Inoculum size (-) |
| **Inter-individual variability** omega(GR) omega(Finoc) omega(Pinoc) | | | | LogNormal<br>LogNormal<br>LogNormal |
| **Correlation of random effects** corr(GR, Finoc) corr(GR, Pinoc) corr(Finoc, Pinoc) | | | 1.1.1.1 | Correlation coefficient Correlation coefficient Correlation coefficient |
| **Parameter-Covariate relationships** beta_GR(AGE) beta_GR(WT0) beta_GR(SEX_0) | | | 1 1 1 1 | AGE in Years on GR<br>Weight in kg on GR<br>Gender female on GR |
| **Residual variability**<br>error_PROP1<br>error_ADD1 | | | | Proportional Error (fraction) - Parasitemia<br>Absolute Error - Parasitemia |
| Objective function<br>AIC<br>BIC | | 1 1 1 | | |

Model: ../PATH/TO/MODEL/DIRECTORY, Significant digits: 3 (Objective function rounded to closest integer value), omega values reported in standard deviation.


Programmer note 1: In the previous table, rows for correlation of random effects and rows for Parameter-Covariate relationships can be added or removed, depending on the final selected model.

Programmer note 2: In the previous table, the path to the model directory in the footnote should be adapted accordingly.


SAS DATE AND TIME PAGE X OF Y


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.2.3.9.1: BLOOD-STAGE PARASITE PROFILE: EXTENDED LOG-LINEAR MIXED MODEL ESTIMATES ANALYSIS SET: PD

| <pre>vpical parameters** oc nter-individual variability** ad(GR) ga(Finoc) ga(Finoc) ga(Phi) ga(Phi) cr(GR, Finoc) r(GR, Finoc) r(GR</pre> | PARAMETER | VALUE | RSE | SHRINKAGE | COMMENT |
|---|---|---|---|---|---|
| <pre>dual variability** of random effects** co rariate relationships** ability** ion ion</pre> | **Typical parameters** GR Finoc Pinoc Fmax Phi Phi | <br> | <br> | 11111 | Parasite growth rate (1/hour) Inoculum viability (-) Inoculum size (-) Maximum fraction of hidden parasites (-) Oscillation phase (-) Period length of the oscillation (h) |
| <pre>f random effects** co) ariate relationships** lability** cion</pre> | **Inter-individual variability** omega(GR) omega(Finoc) omega(Pinoc) omega(Fmax) omega(Phi) omega(Plen) | | | | LogNormal<br>LogNormal<br>LogNormal<br>LogNormal<br>LogNormal |
| rariate relationships** ability** | **Correlation of random effects** corr(GR,Finoc) corr(GR,Pinoc) corr(Finoc,Pinoc) | | | 1 1 1 1 | |
| /ariability** unction | /ariate | | | 1 1 1 1 | AGE in Years on GR<br>Weight in kg on GR<br>Gender female on GR |
| ) ) | **Residual variability** error_RDD1 error_ADD1 Objective function AIC | | 1 1 1 | | Proportional Error (fraction) - Parasitemia<br>Absolute Error - Parasitemia<br>-<br>- |

Model: ../PATH/TO/MODEL/DIRECTORY, Significant digits: 3 (Objective function rounded to closest integer value), omega values reported in standard deviation. Programmer note 1: The table should be included only if such an extended log-linear model had been estimated (refer to SAP section 2.1.3.1).

Programmer note 2: In the previous table, rows for correlation of random effects and rows for Parameter-Covariate relationships can be added or removed, depending on the final selected model.

Programmer note 3: In the previous table, the path to the model directory in the footnote should be adapted accordingly.


```
SAS DATE AND TIME PAGE X OF Y
                                 TABLE 14.2.3.10.1: BLOOD-STAGE PARASITE PROFILE: MODEL DERIVED POPULATION PARAMETERS
                                                                                                                                                                                                                                                                                                     XXX.X<d>
                                                                                                                                                                                                                                                    XXX.X; XXX.X<d>
                                                                                                                                                                                                   X.XX; X.XX<c>
                                                                                                                                                                     X.XX; X.XX<c>
                                                                                                                                                                                                                                                                                                     XXX.X;
                                                                                                 95%-CI
                                                                                                                                                                                                                                                    xxx.xx
xxx.x
                                                                                                                                                                                                                                                                                                     x.xxx
x.xxx
                                                                                                 MEAN
                                                                                                                                                                                                     XX.X
                                                                                                                                                                     XXXX
                                                                                                                                                                                                                                      **Predicted time to reach parasitaemia thresholds (h)**
MMV_PFSPZ-DVI BLOOD STAGE_19_01 - ANALYSIS VERSION
                                                                                                                                                    **Parasitaemia multiplication rate (log10)**
                                                                                                                                                                                                                                                    TIME_PCRPOS <a>
TIME_PCR5000 <a>
                                                                                                                                                                                                                                                                                                     TIME_PCRPOS <b>TIME_PCR5000 <b>
                                                                  ANALYSIS SET: PD
                                                                                                                                                                                                     PMR_Plen <b>>
                                                                                                                                                                    PMR_48h <a>
                                                                                                 PARAMETER
```

<a> derivation based on the log-linear mixed model;
<b> derivation based on the extended log-linear mixed model.
<b> calculated as -1.96\*S.E.+MEAN; 1.96\*S.E.+MEAN, where S.E. denotes the standard error of MEAN, i.e. S.E.=S.D./SQRT(1'000) with S.D. denoting the POPULATION PARAMETER ESTIMATES OBTAINED UPON SAMPLING OF 1'000 SETS OF MODEL POPULATION PARAMETERS FROM THE UNCERTAINTY DISTRIBUTION: MEAN: SAMPLE ARITHMETIC MEAN FOR PARASITAEMIA MULTIPLICATION RATE; SAMPLE GEOMETRIC MEAN FOR PREDICTED TIME TO REACH PARASITAEMIA THRESHOLDS, I.E. 95%-CI: 95% CONFIDENCE INTERVAL FOR THE MEAN (SEE FOOTNOTES <c> and <d>). EXP (MEAN (LOG-TRANSFORMED TIMES)); sample standard deviation.

Programmer note 1: Rows corresponding to the extended log-linear model  $\langle b \rangle$  to be omitted if such model had not been inferred (refer to SAPsection 2.1.3.1).

 document

```
<d> relative standard error of GEOMETRIC MEAN in percentile calculated as S.D.(LOG-TRANSFORMED TIMES)/SQRT(N - 1)*100;
<d> 95% prediction interval calculated as -t(N-1,0.025,0.975)*S.D.+ ARITHMETIC MEAN; t(N-1,0.025,0.975)*S.D.+ ARITHMETIC MEAN, where t(N-1,0.025,0.975) denotes the Student t-value for N-1 degrees of freedom. Note that these procedure assumes normal distribution of the variable.
SAS DATE AND TIME PAGE X OF Y
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                              MEAN: ARITHMETIC MEAN FOR PARASITAEMIA MULTIPLICATION RATE; GEOMETRIC MEAN FOR PREDICTED TIME TO REACH PARASITAEMIA THRESHOLDS;
                                                                                                                                                                                                                                                                                                                                                                                                               XXX.X; XXX.X XXX.X XXX.X; XXX.X;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                               XXX.X; XXX.X XXX.X XXX.X
                                                                                                                                                                                                                                                                                                                                 X.XX; X.XX
                                                                                                                                                                                                                                                                              X.XX; X.XX
                                                        DERIVED PARAMETERS BASED ON INDIVIDUAL PARAMETER ESTIMATES
                                                                                                                                                                  RANGE
                                                                                                                                                                                                                                                                                                                                                                                                               XXX.X; XXX.X XXX.X XXX.X; XXX.X;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                               XXX.X; XXX.X
XXX.X; XXX.X
                                                                                                                                                                                                                                                                              X.XX; X.XX
                                                                                                                                                                                                                                                                                                                                 XXX; XXXX
                                                                                                                                                               95%-PI
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                          XXX.X
XXX.X
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                               XXX.X
XXX.X
                                                                                                                                                               S.D.
                                                                                                                                                                                                                                                                                                                                 \times
                                                                                                                                                                                                                                                                              \times \times \times
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                       RSE: RELATIVE STANDARD ERROR FOR MEAN (IN PERCENTILES; see footnotes <0> and <0>);
                                                                                                                                                                                                                                                                                                                                                                                                                 (%XXX X.XX
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                               XXX.X (XX%<d>)
                                                                                                                                                                                                                                                                                                                                                                                                                                           (%XXX) X.XXX
                                                                                                                                                                                                                                                                              X.XX (XX%<c>)
                                                                                                                                                                                                                                                                                                                                 X.XX (XX%<c>)
                                                                                                                                                               MEAN (RSE)
                                                                                                                                                                                                                                                                              ×
                                                                                                                                                                                                                                                                                                                                 \times
                                                                                                                                                                                                                                                                                                                                                                                                                    XX
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                   \stackrel{\times}{\times}\stackrel{\times}{\times}
                                                                                                                                                                  z
                                                                                                                                                                                                                                                                                                                                                                                       **Predicted time to reach parasitaemia thresholds (h) **
                                                      TABLE 14.2.3.11.1: BLOOD-STAGE PARASITE PROFILE: MODEL
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                             SUMMARY STATISTICS OF INDIVIDUAL PARAMETER ESTIMATES:
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                 95%-PI: 95% PREDICTION INTERVAL (see footnote <e>);
MMV_PFSPZ-DVI BLOOD STAGE_19_01 - ANALYSIS VERSION
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                   derivation based on log-linear mixed model;
                                                                                                                                                                                                                                                 **Parasitaemia multiplication rate (log10)**
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                           RANGE: OBSERVED MINIMUM AND MAXIMUM.
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                             S.D.: STANDARD DEVIATION;
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                       N: NUMBER OF INDIVIDUALS;
                                                                                                                                                                                                                                                                                                                                                                                                               TIME_PCRPOS <a>
TIME_PCR5000 <a>
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                               TIME_PCRFOS <b>TIME_PCR5000 <b>
                                                                                                              ANALYSIS SET: PD
                                                                                                                                                                                                                                                                                                                                 PMR Plen <b>
                                                                                                                                                                                                                                                                              PMR_48h <a>
                                                                                                                                                               PARAMETER
```

Programmer note 1: Derived parameters for the extended log-linear model <b> should be omitted if such model had not been inferred (refer to SAP section 2.1.3.1).

 document


SAS DATE AND TIME PAGE X OF Y MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.2.3.12.1: BLOOD-STAGE PARASITE PROFILE: MODEL DERIVED PARAMETERS BASED ON SIMULATED INDIVIDUAL PARAMETER VALUES

ANALYSIS SET: PD

| PARAMETER | MEAN | 95%-PI |
|---|---|---|
| **Parasitaemia multiplication rate (log10)**<br>PMR_48h <a></a> | ×.×. | x.xx; x.xx |
| PMR_Plen <b>&gt;</b> | XX.XX | X.XX; X.XX |
| **Predicted time to reach parasitaemia thresholds (h)** TIME_PCRS000 <a> TIME_PCRS000 <a></a></a> | × | XXX.X; XXX.X<br>XXX.X; XXX.X |
| TIME_PCRPOS <b>TIME_PCR5000 <b></b></b> | XXXX<br>XXXX | XXX.X; XXX.X<br>XXX.X; XXX.X |

PARAMETER VALUES (SAMPLING FROM IIV DISTRIBUTION) FOR EACH POPULATION (IN TOTAL 1'000'000 SETS OF INDIVIDUAL PARAMETER VALUES): MEAN: SAMPLE ARITHMETIC MEAN FOR PARASITAEMIA MULTIPLICATION RATE; SAMPLE GEOMETRIC MEAN FOR PREDICTED TIME TO REACH PARASITAEMIA THRESHOLDS; 95%-PI: 95% PREDICTION INTERVAL CALCULATED FROM THE 0.025TH AND 0.975TH SAMPLE QUANTILES. SUMMARY STATISTICS UPON SIMULATING 1'000 SETS OF POPULATION PARAMETERS (SAMPLING FROM UNCERTAINTY DISTRIBUTION) AND 1'000 SETS OF INDIVIDUAL

<a> derivation based on log-linear mixed model;
<b> derivation based on extended log-linear mixed model.

Programmer note 1: The table should be included only if the model parameter IIV distribution could be estimated for all model parameters (refer to SAP section 2.1.3.1). Programmer note 2: Derived parameters for the extended log-linear model <b> should be omitted if such model had not been inferred (refer to SAP section 2.1.4).

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

SAS DATE AND TIME PAGE X OF Y

TABLE 14.2.3.13.1: BLOOD-STAGE PARASITE CLEARANCE PROFILE: INDIVIDUAL LOG-LINEAR MODEL ESTIMATES

ANALYSIS SET: PD

COHORT = COHORT 1 SUBJECT = XXX

| | ESTIMATE S.E. | S. I. E. I. | 95% C.I. | . | 95% C.I. P-VALUE |
|---|---|---|---|---|---|
| MODEL ESTIMATES:<br>INTERCEPT<br>TIME | × | × × × × | X.XX ;X.XX XX.XX XX.XX | × × | XX.X; XX.X<br>XX.X; XX.X X.XX <a></a> |
| DERIVED PARAMETERS:<br>LOG10PRR48 | ×.×. | | x , x, x | × | |
| PC50 | XX.X | | XX.X; XX.X | × | |
| PC99 | xx.x | | XX.X; | xx.x | |
| TYPE 3 TESTS OF FIXED EFFECTS: | | | | | <q> xx.x</q> |

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.2.3.14.1: BLOOD-STAGE PARASITE CLEARANCE PROFILE: DESCRIPTIVE STATISTICS

ANALYSIS SET: PD

TIME TO PARASITE CLEARANCE (DAYS)

n Geom. Mean 95% C.I. <a> Geom. S.D. Min; Max

<a> TWO-SIDED 95% CONFIDENCE INTERVAL ON THE GEOMETRIC MEAN.


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.2.3.14.1: BLOOD-STAGE PARASITE CLEARANCE PROFILE: DESCRIPTIVE STATISTICS

ANALYSIS SET: PD

LOG10 PARASITE REDUCTION RATIO PER 48h (LOG10PRR48)

| Mın; Max | | xx;xx | XX;XX | |
|----------|---|-----------------|-----------------|---------------------|
| | | XXX.XXX | XX.XXX | XXX.XX |
| 95% C.I. | | XX.XX; | XX.XXX; XX.XXX | XX.XX; |
| n Mean | | XX.XXX | | XX.XXX |
| п | - | XX | × | XX |
| | | COHORT 1 (N=XX) | COHORT 2 (N=XX) | ALL SUBJECTS (N=XX) |

SUMMARY STATISTICS ESTIMATED BY USING THE INVERSE-VARIANCE METHOD TO CALCULATE THE WEIGHTED AVERAGE LINEAR RECRESSION SLOPE AND CORRESPONDING STANDARD ERROR.

ONLY SUBJECTS WHOSE OPTIMAL LOG-LINEAR REGRESSION MODEL OVERALL P-VALUE < 0.001 ARE INCLUDED.

#### Programmer notes:

Show the table for all parameters starting in a new page in the following order: time to parasite clearance,  $log_{10}PRR_{46}$ , PC50, PC99.


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.2.3.15.1: DESCRIPTIVE STATISTICS OF LOG10(PARASITAEMIA) ACTUAL VALUES

ANALYSIS SET: PD

| ANALYSIS PHASE<br>ANALYSIS VISIT | COHORT 1 (N=XX) | COHORT 2<br>(N=XX) | ALL SUBJECTS (N=XX) |
|---|---|---|---|
| SCREENING<br>DAY 1, PREDOSE | | | |
| | × | ×× | × |
| Mean (S.D) | XX.X (X.X) | XX.X (X.X) | XX.X (X.X) |
| Median | ×.×× | ××.× | ××.×× |
| Min; Max | (XX; XX) | (XX; XX) | (XX; XX) |
| 95% C.I. <a></a> | (XX; XX) | (XX; XX) | (XX :XX) |
| CHALLENGE | | | |
| | XX | XX | ×× |
| Mean (S.D) | (X.X) XX | (X.X) XX | XX.X (X.X) |
| Median | XX.X | XX.X | XX.XX |
| Min; Max | (XX; XX) | (XX; XX) | (XX; XX) |
| 95% C.I. <a></a> | (XX; XX) | (XX; XX) | (XX; XX) |
| | ×× | ×× | ×× |
| Mean (S.D) | (X.X) XX | XX.X (X.X) | XX.X (X.X) |
| Median | ××.×× | x.xx | xx.x |
| Min; Max | (XX; XX) | (XX; XX) | (XX; XX) |
| 95% C.I. <a></a> | (XX; XX) | (XX; XX) | (XX; XX) |
| RIAMET DAY 1, 2H | | | |
| | XX | XX | XX |
| Mean (S.D) | (X.X) XXX | XX.X (X.X) | XX.X (X.X) |
| Median | XX.X | XX.X | XX.X |
| Min; Max | (XX; XX) | (XX; XX) | (XX; XX) |
| 95% C.I. <a></a> | (XX; XX) | (XX; XX) | (XX; XX) |

<sup>&</sup>lt;a> TWO-SIDED 95% CONFIDENCE INTERVAL ON THE ARITHMETIC MEAN.


#### SAFETY

#### Adverse events

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

SAS DATE AND TIME PAGE X OF Y

TABLE 14.3.1.1: ADVERSE EVENTS OVERVIEW

ANALYSIS SET: SAFETY

| | ) | (N=XX) | <b>-</b> | Ś | (N=XX) | | Ç | (N=XX) | )<br>H |
|---|---|---|---|---|---|---|---|---|---|
| z | С | 0/0 | ш | С | 0/0 | E | С | 0/0 | Ħ |
| AT LEAST ONE AE | !<br>! X | XX | XX | i<br>! X | | i<br>! X | ! X | . x . x x | × |
| AT LEAST ONE SERIOUS AE | × | XX.X | XX | X | XX.X | × | X | XX.X | X |
| AT LEAST ONE GRADE 2 3 AE | × | XX.X | ×× | × | XX.X | × | × | XX.X | × |
| AT LEAST ONE FATAL AE | × | XX.X | ×× | × | XX.X | × | × | XX.X | × |
| AT LEAST ONE AE RELATED TO PÉSPZ INOCULUM | × | XX.X | ×× | × | XX.X | × | × | XX.X | × |
| AT LEAST ONE AE RELATED TO ANTIMALARIAL TREATMENT | × | XX.X | XX | × | XX.X | XX | × | XX.X | × |
| AT LEAST ONE AE RELATED TO RIAMET | XX | x.xx | × | × | XX.X | × | × | XX.X | $\times$ |
| AT LEAST ONE AE RELATED TO MALARONE | × | XX.X | ×× | × | XX.X | XX | × | XX.X | $\times$ |
| AT LEAST ONE SERIOUS AE RELATED TO PÉSPZ INOCULUM | XX | XX.X | XX | X | XX.X | XX | XX | XX.X | X |
| AT LEAST ONE AE FOR WHICH THE STUDY WAS DISCONTINUED | × | XX.X | XX | × | XX.X | × | × | XX.X | × |
| AT LEAST ONE AE FOR WHICH THE ANTIMALARIAL TREATMENT WAS DISCONTINUED | × | XX.X | ×× | × | XX.X | XX | × | XX.X | $\times$ |
| AT LEAST ONE AE FOR WHICH RIAMET WAS DISCONTINUED | × | XX.X | ×× | × | XX.X | × | × | XX.X | $\times$ |
| AT LEAST ONE AE FOR WHICH MALARONE WAS DISCONTINUED | × | XX.X | XX | × | XX.X | × | × | XX.X | X |
| AT LEAST ONE AE OF SPECIAL INTEREST | × | XX.X | ×× | × | XX.X | × | × | XX.X | XX |
| AT LEAST ONE AE OF SPECIAL INTEREST RELATED TO PESPZ INOCULUM | × | XX.X | ×× | × | XX.X | × | × | XX.X | $\times$ |
| AT LEAST ONE AE OF SPECIAL INTEREST RELATED TO ANTIMALARIAL TREATMENT | ×× | ××× | ×× | ×× | > >> | ** | > | > >> | > |

n= NUMBER OF SUBJECTS WITH EVENT, m = NUMBER OF EVENTS, AE = ADVERSE EVENT.

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET.

ONLY ADVERSE EVENTS THAT STARTED AFTER PESPZ INOCULATION ARE SHOWN.

RELATED IS DEFINED AS RELATED/SUSPECTED TO CHALLENGE AGENT/ANTIMALARIAL TREATMENT ACCORDING TO THE INVESTIGATOR, OR A MISSING RELATEDNESS.

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.3.1.2: ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM

ANALYSIS SET: SAFETY

| | | COHORT 1 | | O | COHORT 2 | <b>⊘</b> I | AL | ALL SUBJECTS | ECIS |
|---|---|---|---|---|---|---|---|---|---|
| AND PREFERRED TERM | п | % % % | Е | | (N-N) | Е | | (VV-VI) | ш |
| ANY AE | i × | XX XX.XX XX | | | XXXXXXX | <br> | | XX XX.X XX | × |
| GASTROINTESTINAL DISORDERS | × | XX.X | × | × | XX.X | × | X | XX.X | × |
| DIARRHOEA | × | XX.X | × | × | XX.X | × | × | XX.X | × |
| GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS | × | XX.X | × | X | XX.X | × | × | XX.X | × |
| FATIGUE | × | XX.X | × | × | XX.X | × | × | XX.X | X |
| FEELING HOT | × | XX.X | × | × | XX.X | × | × | XX.X | × |
| INJECTION SITE ERYTHEMA | × | XX.X | XX | XX | XX.X | XX | × | XX.X | × |
| INFECTIONS AND INFESTATIONS | × | XX.X | × | × | XX.X | × | × | XX.X | × |
| RHINITIS | × | XX.X | × | × | XX.X | × | × | XX.X | × |
| ATMOMITAN | × | ××× | × | × | × | × | >> | > >> | × |

Etc.

n= NUMBER OF SUBJECTS WITH EVENT, m = NUMBER OF EVENTS, AE = ADVERSE EVENT. THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET. ONLY ADVERSE EVENTS THAT STARTED AFTER PISPZ INOCULATION ARE SHOWN.

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.3.1.3: ADVERSE EVENTS BY MEDDRA PREFERRED TERM BY DESCENDING ORDER OF FREQUENCY

ANALYSIS SET: SAFETY

| PREFERRED TERM DIARRHOEA FALIGUE FEDITING HOT | COHO<br>N N N N N N N N N N N N N N N N N N N | COHORT 1 (N=XX) n % XX XX.X XX XX.X XX XX.X XX XX.X XX XX.X | OHOOO I XXXX | COHORT 2 (N=XX) N % XX XX.X XX XX.X XX XX.X XX XX.X XX XX.X | ALL AKK | ALL SUBJECTS (N=XX) n % XX XX.X XX XX.X XX XX.X XX XX.X XX XX.X |
|---|---|---|---|---|---|---|
| INDECTION SITE ENTINEMS PREUMONIS | < × × | < × × | < × × | < × × | < | < × × × |

Etc.

n= NUMBER OF SUBJECTS WITH EVENT, AE = ADVERSE EVENT. THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET. ONLY ADVERSE EVENTS THAT STARTED AFTER PÉSPZ INOCULATION ARE SHOWN.

Programmer note: the adverse events will be sorted by descending order of frequency in the all subjects group.


MMV\_PfSPZ-DVI Blood Stage\_19\_01

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.3.1.4: SERIOUS ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM

ANALYSIS SET: SAFETY

| SYSTEM ORGAN CLASS AND PREFERRED TERM | 0 Z q | COHORT 1 (N=XX) | 8 g | COHORT 2<br>(N=XX) | | ALL SUBJECTS<br>(N=XX)<br>n % |
|---|---|---|---|---|---|---|
| ANY AE | | | | XX XX XX | | |
| GASTROINTESTINAL DISORDERS | × | XX.X | XX | XX.X | X | xx.x |
| DIARRHOEA | × | XX.X | × | XX.X | × | XX.X |
| GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS | × | XX.X | × | xx.x | × | xx.x |
| FATIGUE | × | XX.X | × | ××.× | × | xx.x |
| FEELING HOT | × | XX.X | × | XX.X | × | XX.X |
| INJECTION SITE ERYTHEMA | × | XX.X | × | XX.X | × | XX.X |
| INFECTIONS AND INFESTATIONS | × | XX.X | X | XX.X | X | XX.X |
| RHINITIS | × | XX.X | × | ××.× | × | xx.x |
| PNEUMONIA | × | XX.X | × | ××.× | × | xx.x |
| Etc. | | | | | | |

n= NUMBER OF SUBJECTS WITH EVENT, AE = ADVERSE EVENT. THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET. ONLY ADVERSE EVENTS THAT STARTED AFTER PÉSPZ INOCULATION ARE SHOWN.

### Programmer note: repeat Table 14.2.1.4 for:

TABLE 14.3.1.6: PfSPZ INOCULUM RELATED ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM TABLE 14.3.1.5: GRADE 3 OR MORE ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

SAS DATE AND TIME PAGE X OF Y

TABLE 14.3.1.7: ANTIMALARIAL TREATMENT RELATED ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM

ANALYSIS SET: SAFETY

ANTIMALARIAL TREATMENT = RIAMET OR MALARONE

| | 8 | OHORT 1 | 8 | COHORT 2 | | ALL SUBJECTS |
|---|---|---|---|---|---|---|
| | 2 | (N=XX) | Z) | (N=XX) | Ξ | (N=XX) |
| SYSTEM ORGAN CLASS AND PREFERRED TERM | Д | 0/0 | Д | 0/0 | Ц | 0/0 |
| | i | | | | | |
| ANY AE | × | XX.X | × | XX.X | × | XX.X |
| GASTROINTESTINAL DISORDERS | × | XX.X | × | XX.X | × | XX.X |
| DIARRHOEA | X | XX.X | × | XX.X | X | XX.X |
| GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS | XX | XX.X | XX | XX.X | XX | XX.X |
| FATIGUE | XX | XX.X | × | XX.X | XX | XX.X |
| FEELING HOT | X | x.xx | X | ××.× | XX | XX.X |
| INJECTION SITE ERYTHEMA | X | XX.X | X | XX.X | X | XX.X |
| INFECTIONS AND INFESTATIONS | XX | XX.X | XX | XX.X | XX | XX.X |
| RHINITIS | XX | XX.X | × | XX.X | XX | XX.X |
| PNEUMONIA | × | XX.X | × | XX.X | × | XX.X |

ANTIMALARIAL TREATMENT = RIAMET

n= NUMBER OF SUBJECTS WITH EVENT, AE = ADVERSE EVENT. THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET. ONLY ADVERSE EVENTS THAT STARTED AFTER PÍSPZ INOCULATION ARE SHOWN.

#### Programmer note: repeat Table 14.2.1.4 for:

TABLE 14.3.1.8: SERIOUS PÍSPZ INOCULUM RELATED ADVERSE EVENTS BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM

### Programmer note: repeat Table 14.2.1.8 for:

TABLE 14.3.1.9: ADVERSE EVENTS FOR WHICH THE ANTIMALARIAL TREATMENT WAS DISCONTINUED BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM

#### Programmer note: repeat Table 14.2.1.4 for:

TABLE 14.3.1.10: ADVERSE EVENTS OF SPECIAL INTEREST RELATED TO PESPZ INOCULUM BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM

### Programmer note: repeat Table 14.2.1.8 for:

TABLE 14.3.1.11: ADVERSE EVENTS OF SPECIAL INTEREST RELATED TO ANTIMALARIAL TREATMENT BY MEDDRA SYSTEM ORGAN CLASS AND PREFERRED TERM


## 3.3.2 Clinical laboratory evaluation

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.3.2.1: DESCRIPTIVE STATISTICS OF LABORATORY TEST RESULTS

SAS DATE AND TIME PAGE X OF Y

ANALYSIS SET: SAFETY

LABORATORY CATEGORY: LABORATORY PARAMETER 1 (unit)

| | | ACTUAL VALUES | | CH | CHANGES FROM BASELINE | E |
|---|---|---|---|---|---|---|
| | COHORT 1 (N=XX) | COHORT 2<br>(N=XX) | ALL SUBJECTS (N=XX) | COHORT 1 (N=XX) | COHORT 2 (N=XX) | ALL SUBJECTS (N=XX) |
| BASELINE<br>n | × | XX | × | | | |
| Mean (S.D) | XX.X (X.X) | XX.X (X.X) | XX.X (X.X) | | | |
| Median | XX.X | XX.XX | XX.XX | | | |
| Min; Max | (XX; XX) | (XX; XX) | (XX; XX) | | | |
| AY X | | | | | | |
| и | XX | XX | XX | XX | XX | XX |
| Mean (S.D) | (X.X) XX | XX.X (X.X) | (X.X) XXX | XX.X (X.X) | (X.X) XXX | XX.X (X.X) |
| Median | xx.x | XX.X | x.xx | XX.X | XX.X | XX.X |
| Min; Max | (XX; XX) | (XX; XX) | (XX; XX) | (XX; XX) | (XX; XX) | (XX; XX) |
| AY X | | | | | | |
| п | ×× | XX | XX | XX | XX | XX |
| Mean (S.D) | (X.X) XX | XX.X (X.X) | (X.X) XXX | XX.X (X.X) | (X.X) XXX | XX.X (X.X) |
| Median | XX.X | xx.xx | XX.XX | XX.X | XX.X | XX.X |
| Min; Max | (XX ; XX) | (XX; XX) | (XX; XX) | (XX; XX) | (XX; XX) | (XX; XX) |
| AY X | | | | | | |
| п | XX | XX | XX | XX | XX | XX |
| Mean (S.D) | (X.X) | XX.X (X.X) | XX.X (X.X) | XX.X $(X.X)$ | XX.X (X.X) | XX.X (X.X) |
| Median | xx.x | XX.X | x.xx | XX.X | XX.X | XX.X |
| Min; Max | (XX; XX) | (XX; XX) | (XX; XX) | (XX; XX) | (XX; XX) | (XX; XX) |

Etc.


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.3.2.2: CROSS-TABULATION OF LABORATORY ABNORMALITIES VERSUS BASELINE

SAS DATE AND TIME PAGE X OF Y

ANALYSIS SET: SAFETY

LABORATORY CATEGORY: LABORATORY PARAMETER 1 (unit)

ABNORMALITY AT BASELINE

| COHORT/<br>ANALYSIS VISIT | ABNORMALITY | z | 0/0 | Z | 0/0 | LOW | ⊗ °/° | N C | NORMAL<br>n % | H | HIGH<br>n % | MIS | MISSING<br>n % |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| COHORT 1 (N=XX) | | <br> | <br> | <br> | <br> | <br> <br> <br> | <br> <br> <br> <br> | <br> | <br> <br> <br> <br> | <br> | <br> <br> <br> <br> | <br> | <br> |
| DAY 7 | LOW | × | ××. | × | ×.× | × | ××. | × | ××. | × | ×.× | × | ×.× |
| | NORMAL | × | XX.X | | | XX | XX.X | XX | XX.X | X | XX.X | XX | XX.X |
| | HIGH | × | XX.X | X | XX.X | X | XX.X | X | XX.X | X | XX.X | X | XX.X |
| | TOTAL | × | XX.X | X | XX.X | X | XX.X | X | XX.X | X | XX.X | X | XX.X |
| WORST-CASE POST-BASELINE | TOW | × | ××.× | X | XX.X | $\times$ | XX.X | $\times$ | XX.X | × | XX.X | $\times$ | XX.X |
| | NORMAL | × | XX.X | | | X | XX.X | X | XX.X | X | XX.X | X | $\times \times \times$ |
| | HIGH | × | XX.X | X | XX.X | X | XX.X | X | XX.X | X | XX.X | X | $\times \times \times$ |
| | TOM + HIGH | × | XX.X | X | XX.X | $\times$ | XX.X | $\times$ | XX.X | $\times$ | XX.X | $\times$ | XX.X |
| | TOTAL | × | XX.X | X | XX.X | $\times$ | XX.X | $\times$ | XX.X | $\times$ | XX.X | $\times$ | XX.X |
| WORST-CASE CHALLENGE | TOW | × | $\times \times \times$ | X | XX.X | X | XX.X | $\times$ | XX.X | $\times$ | XX.X | X | XX.X |
| | NORMAL | X | XX.X | | | X | XX.X | X | XX.X | X | XX.X | X | XX.X |
| | TOM + HIGH | × | XX.X | X | XX.X | $\times$ | XX.X | $\times$ | XX.X | $\times$ | XX.X | $\times$ | XX.X |
| | TOTAL | × | XX.X | X | XX.X | $\times$ | XX.X | $\times$ | XX.X | $\times$ | XX.X | $\times$ | XX.X |
| WORST-CASE RESCUE | TOM | × | XX.X | $\times$ | XX.X | $\times$ | XX.X | × | XX.X | X | XX.X | $\times$ | XX.X |
| | NORMAL | X | XX.X | | | X | XX.X | X | XX.X | X | XX.X | X | XX.X |
| | TOTAL | × | XX.X | ×× | XX.X | $\times$ | XX.X | × | хх.х | $\stackrel{\times}{\times}$ | ХХ.Х | × | хх.х |
| COHORT 2 (N=XX) | | | | | | | | | | | | | |
| | TANGON | >> | > | | | 2 | > | 2 | > | 2 | 2 | 2 | > |
| DAI / | NORMAL | V > | ۷٠,۷ | > | > | < > | ۷٠٧ | < > | ۷٠,۷ | \<br>\<br>\<br>\ | ۷٠٧ | < > | ۷٠,۷ |
| | H D I H | <b>4</b> | ۷٠,۷ | < ? | ۷٠,۷ | < ? | < :>< :> | 4 3 | ۷٠,۷ | 4 3 | < > | 4 3 | < : > |
| | TOTAL | ΥΥ | XX.X | ΥX | ٧٧٠٧ | ΥX | YY.Y | ΥX | ٧٧٠٧ | ΥX | ٧٧٠٧ | ΥX | YY.Y |

Etc.

N = TOTAL NUMBER OF SUBJECTS PER ABNORMALITY WITHIN EACH COHORT AND ANALYSIS VISIT
N' = TOTAL NUMBER OF SUBJECTS WITH A POST-BASELINE EMERGENT ABNORMALITY WITHIN EACH COHORT AND ANALYSIS VISIT
THE WORST-CASE ANALYSIS VISIT CONSIDERS ALL POST-BASELINE ASSESSMENTS, INCLUDING UNSCHEDULED ASSESSMENTS, AND IS SHOWN OVERALL

AND BY ANALYSIS PHASE. THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT AND PER ANALYSIS VISIT IN THE SAFETY SET, EXCLUDING SUBJECTS WITH MISSING VALUES PER COHORT AND PER ANALYSIS VISIT.

SAS DATE AND TIME PAGE X OF Y


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.3.2.3: LIVER ENZYME ELEVATION CATEGORIES

ANALYSIS SET: SAFETY

| | 8 | COHORT 1 | COH | COHORT 2 | ALL | ALL SUBJECTS |
|---|---|---|---|---|---|---|
| | _ | (X=XX) | Z) | (N=XX) | Ż) | (N=XX) |
| CRITERION | П | 0/0 | П | 0/0 | п | 0/0 |
| TIV | | | <br> | | <br> | |
| NIDX8 < | X | XX.X | X | XX.X | × | XX.X |
| > 5XULN | × | XX.X | X | XX.X | ×× | xx.x |
| > 3XULN | XX | ××.× | XX | XX.X | XX | XX.X |
| AST | | | | | | |
| > 8XULN | × | XX.X | X | XX.X | × | XX.X |
| > 5XULN | × | xx.x | × | XX.X | × | XX.X |
| > 3XULN | × | xx.x | × | XX.X | × | XX.X |
| ALT OR AST | | | | | | |
| > 8XULN | × | xx.x | × | XX.X | × | XX.X |
| > 5XULN | × | xx.x | × | XX.X | × | XX.X |
| > 3XULN | × | xx.x | × | XX.X | × | XX.X |
| TOTAL BILIRUBIN > 2XULN | × | x.x. | × | XX.X | × | XX.X |
| CONJUGATED BILIRUBIN FRACTION >35% | × | XX.X | × | XX.X | × | XX.X |
| POTENTIAL HY'S LAW CASE | X | XX.X | X | XX.X | × | XX.X |

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET, EXCLUDING SUBJECTS WITH MISSING VALUES. FOR EACH OF THE CRITERIA, THE HIGHEST POST-BASELINE VALUE IS CONSIDERED.

POTENTIAL HY'S LAW CASE: ALT OR AST > 3XULN AND TOTAL BILIRUBIN > 2XULN AT THE SAME SAMPLE, TOGETHER WITH A CONJUGATED BILIRUBIN FRACTION >358.

#### 3.3.3 Vital signs

The analysis tables for vital signs parameters are largely identical to the laboratory tables.

TABLE 14.3.3.1: DESCRIPTIVE STATISTICS OF VITAL SIGNS

TABLE 14.3.3.2: CROSS-TABULATION OF VITAL SIGNS ABNORMALITIES VERSUS BASELINE


The analysis tables for ECG parameters are largely identical to the laboratory tables.

TABLE 14.3.4.1: DESCRIPTIVE STATISTICS OF ECG


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.3.4.2: CROSS-TABULATION OF ECG ABNORMALITIES VERSUS BASELINE

ANALYSIS SET: SAFETY

ECG PARAMETER 1 (unit)

| | | | | | | | | BNOR | MALITY | . AT | ABNORMALITY AT BASELINE | NE | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| COHORT /<br>ANALYSIS VISIT | ABNORMALITY | Z | 0/0 | Ż | 0/0 | LOW | <br> -<br> % | | NORMAL<br>n % | HI | HIGH<br>n % | MIS | MISSING<br>n % |
| COHORT 1 (N=XX) | | <br> <br> <br> | | i<br>!<br>! | | <br> | <br> | <br> <br> | <br> | <br> | <br> | !<br>!<br>! | <br> |
| RIAMET DAY 2 | TOM | × | ×.× | × | XX.X | × | ×.× | × | XXX.X | × | XX.X | × | ×.× |
| | NORMAL | × | XX.X | | | X | XX.X | X | $\times \times \times$ | X | XX.X | X | XX.X |
| | HIGH | × | XX.X | XX | XX.X | X | XX.X | X | $\times \times \times$ | XX | XX.X | XX | XX.X |
| | TOTAL | × | XX.X | $\times$ | XX.X | X | XX.X | $\times$ | XX.X | X | XX.X | $\times$ | XX.X |
| RIAMET DAY 3 | LOW | × | XX.X | X | XX.X | X | XX.X | X | $\times \times \times$ | X | XX.X | X | XX.X |
| | NORMAL | × | XX.X | | | X | XX.X | X | $\times \times \times$ | X | XX.X | X | XX.X |
| | HIGH | × | XX.X | × | $\times \times \times$ | X | XX.X | $\times$ | $\times \times \times$ | × | XX.X | $\times$ | XX.X |
| | TOTAL | × | XX.X | × | XX.X | X | XX.X | $\times$ | $\times \times \times$ | $\times$ | XX.X | × | XX.X |
| WORST-CASE POST-BASELINE | LOW | × | XX.X | X | XX.X | X | XX.X | $\times$ | $\times \times \times$ | X | XX.X | X | XX.X |
| | NORMAL | × | XX.X | | | X | XX.X | X | $\times \times \times$ | XX | XX.X | XX | XX.X |
| | HIGH | × | XX.X | $\times$ | XX.X | X | XX.X | $\times$ | XX.X | X | XX.X | $\times$ | XX.X |
| | LOW + HIGH | × | XX.X | $\times$ | XX.X | X | XX.X | $\times$ | XX.X | X | XX.X | $\times$ | XX.X |
| | TOTAL | × | XX.X | X | XX.X | × | XX.X | × | XX.X | × | XX.X | × | ×.× |
| COHORT 2 (N=XX) | | | | | | | | | | | | | |
| RIAMET DAY 2 | LOW<br>NORMAL | ×× | × × × | $\stackrel{\times}{\times}$ | ×. × | ×× | × × × | $\stackrel{\times}{\times}\stackrel{\times}{\times}$ | × × × | ×× | × × | X X | × × × |
| | HIGH<br>TOTAL | $\stackrel{\times}{\times}\stackrel{\times}{\times}$ | ××.×<br>××.× | $\stackrel{\times}{\scriptscriptstyle \times}$ | × | $\overset{\times}{\times}\overset{\times}{\times}$ | ××.×<br>××.× | $\stackrel{\times}{\times}\stackrel{\times}{\times}$ | × | $\stackrel{\times}{\times}\stackrel{\times}{\times}$ | × | $\stackrel{\times}{\times}\stackrel{\times}{\times}$ | ××.×<br>××.× |

Etc.

N = TOTAL NUMBER OF SUBJECTS PER ABNORMALITY WITHIN EACH COHORT AND ANALYSIS VISIT

N' = TOTAL NUMBER OF SUBJECTS WITH A POST-BASELINE EMERGENT ABNORMALITY WITHIN EACH COHORT AND ANALYSIS VISIT

THE WORST-CASE ANALYSIS VISIT CONSIDERS ALL POST-BASELINE ASSESSMENTS, INCLUDING UNSCHEDULED ASSESSMENTS.

THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT AND PER ANALYSIS VISIT IN THE SAFETY SET, EXCLUDING SUBJECTS WITH MISSING VALUES PER COHORT AND PER ANALYSIS VISIT.

MMV\_PfSPZ-DVI Blood Stage\_19\_01

MMV PFSPZ-DVI BLOOD STAGE 19 01 - ANALYSIS VERSION

TABLE 14.3.4.3: TABULATION OF QTC CHANGE ABNORMALITIES

QTCB INTERVAL (ms)

ANALYSIS SET: SAFETY

0/0 ALL SUBJECTS CN, ××  $\stackrel{\times}{\times}\stackrel{\times}{\times}$  $\stackrel{\times}{\times}\stackrel{\times}{\times}$ (N=XX) XX.X XX.X 100 × × ×  $\overset{\times}{\times}\overset{\times}{\times}$ XX.X 100 0//0 q X X X X\* \* \* \* \* \* \* \* ××.× ××.×  $\overset{\times}{\overset{\times}{\cdot}}\overset{\times}{\overset{\times}{\cdot}}$ 0/0 CN,  $\stackrel{\times}{\times}\stackrel{\times}{\times}$  $\stackrel{\times}{\times}\stackrel{\times}{\times}$  $\stackrel{\times}{\times}\stackrel{\times}{\times}$ COHORT 2 (N=XX)  $\overset{\times}{\times}\overset{\times}{\times}$ XX.X 100  $\overset{\times}{\times}\overset{\times}{\cdot}$ 100 0/0 × × × × ¤ X X X X\* \* \* \* XX.X XX.X 0/0 CN, ×× ×× ×× COHORT 1 (N=XX) XX.XX XX.XX 1000 100 0/0 q X X X XX X X XX X X XWORST-CASE POST-BASELINE ]30,60] <= 30 (NORMAL) ]30,60] <= 30 (NORMAL) <= 30 (NORMAL) RIAMET DAY 2 RIAMET DAY 3 130,60] TOTAL TOTAL TOTAL 09 < 09 <

CN' = CUMULATIVE NUMBER OF SUBJECTS WITH A QTC CHANGE ABNORMALITY WITHIN EACH COHORT AND ANALYSIS VISIT
THE WORST-CASE ANALYSIS VISIT CONSIDERS ALL POST-BASELINE ASSESSMENTS, INCLUDING UNSCHEDULED ASSESSMENTS.
THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT AND PER ANALYSIS VISIT IN THE SAFETY SET, EXCLUDING SUBJECTS WITH MISSING VALUES PER COHORT AND PER ANALYSIS VISIT.

#### Malaria clinical score 3.3.5

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

TABLE 14.3.5.1: DESCRIPTIVE STATISTICS OF MALARIA CLINICAL SCORE

SAS DATE AND TIME PAGE X OF Y

ANALYSIS SET: SAFETY

ALL SUBJECTS XX XX.X (X.X) XX.X XX XX.X (X.X) XX.X (XX, XX) XX XX.X (X.X) XX.X (XX; XX) (XX; XX) CHANGES FROM BASELINE XX XX.X (X.X) XX.X (XX, XX) XX XX.X (X.X) XX.X XX XX.X XX.X XX.X COHORT 2 (N=XX)(XX; XX) (XX; XX) XX XX.X (X.X) XX.X (X.X) X.XX XX.X (X.X) COHORT 1 (XX; XX) (XX; XX) (XX; XX) XX.X XX.X ALL SUBJECTS XX.X (X.X) XX.X (XX, XX) XX XX.X (X.X) XX.X XX XX.X (X.X) XX.X (X.X) XX.X (XX; XX) (XX; XX) XX; XX) XX.X XX XX.X (X.X) XX.X (XX; XX) XX XX.X (X.X) XX.X (XX; XX) ACTUAL VALUES XX XX.X (X.X) XX.X XX XX.X (X.X) XX.X (XX; XX) COHORT 2 (N=XX) (XX; XX) XX XX.X (X.X) XX.X XX XX.X (X.X) XX.X XX XX.X (X.X) XX.X XX XX.X (X.X) XX.X COHORT 1 (N=XX)(XX; XX) (XX; XX) (XX; XX) (XX; XX) Min; Max WORST-CASE POST-BASELINE Mean (S.D) Median Min; Max Mean (S.D) Mean (S.D) Mean (S.D) Min; Max Min; Max Median Median BASELINE DAY 7 DAY 8


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

ANALYSIS SET: SAFETY

ANALYSIS PHASE = CHALLENGE + RESCUE

| ALL SUBJECTS (N=XX) | XX.X<br>XX.X<br>XX.X<br>100 | XXXXX<br>XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX<br>XXXXXX<br>100 | XX.X<br>XX.X<br>XX.X<br>100 |
|---|---|---|---|---|
| ALL SUBJ | * * * * * | X X X X X | * * * * * | $\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}$ |
| ORT 2<br>XX) | X X X X X X 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | X X X X X X X X X X X X X X X X X X X | X X X X X X X X X X X X X X X X X X X | XX |
| COHORT<br>(N=XX)<br>n % | | $\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}$ | * * * * * | X X X X X |
| RT 1<br>XX) | X X X X X 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | X X X X X X X X X X X X X X X X X X X | X X X X X X X X X X X X X X X X X X X | XX.X<br>XX.X<br>XX.X<br>100 |
| COHORT<br>(N=XX)<br>n % | * * * * * | X X X X X | $X \times X \times X$ | * * * * * |
| MALARIA SIGN/SYMPTOM | 1 А 1 | HEADACHE<br>0<br>1<br>2<br>3<br>TOTAL | MYALGIA<br>0<br>1<br>2<br>3<br>3<br>TOTAL | ARTHRALGIA<br>0<br>1<br>2<br>3<br>TOTAL<br>Etc. |

ANALYSIS PHASE = CHALLENGE

Etc.


TABLE 14.3.5.2: FREQUENCY TABLE OF THE WORST-CASE INDIVIDUAL MALARIA SIGNS AND SYMPTOMS

0-ABSENT; 1=MILD; 2=MODERATE; 3=SEVERE
THE DENOMINATOR FOR THE PERCENTAGE CALCULATIONS IS THE TOTAL NUMBER OF SUBJECTS PER COHORT IN THE SAFETY SET, EXCLUDING SUBJECTS WITH MISSING VALUES.
THE WORST-CASE IS THE HIGHEST POST-BASELINE SCORE WITHIN THE ANALYSIS PHASE AND IS DERIVED PER SIGN/SYMPTOM.
ANY SYMPTOM SHOWS THE WORST-CASE SEVERITY OF THE SIGN/SYMPTOM WITH THE HIGHEST SEVERITY.

#### Programmer notes:

• All malaria signs and symptoms will be shown (headache, myalgia, arthralgia, fatigue/lethargy, malaise, chills/shivering/rigors, sweating/hot spells, anorexia, nausea, vomiting, abdominal discomfort, fever, tachycardia and hypotension)


## **MOCK LISTINGS**

# GENERAL CHARACTERISTICS

## Subject disposition

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

SAS DATE AND TIME PAGE X OF Y

LISTING 16.2.1.1: ALLOCATION

ANALYSIS SET: ALL SCREENED SUBJECTS

m-PD NO
YES
YES
YES
YES
NO
YES
NO
YES
NO
NO
NO
NO SAF PD COHORT 2 COHORT 2 COHORT 1 COHORT 2 COHORT 1 COHORT 2 COHORT 1 COHORT 1 COHORT 1 SUBJECT DATETIME OF SIGNING NUMBER INFORMED CONSENT [1] COHORT ddMMMYyyy;hh:mm ddMMMyyyy;hh:mm ddMMyyyy;hh:mm ddMMyyyy;hh:mm ddMMyyyy:hh:mm ddMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm XXXX


<sup>[1]</sup> DATETIME OF THE EARLIEST AVAILABLE INFORMED CONSENT FORM SIGNATURE.

| SAS DATE AND TIME | PAGE X OF Y | |
|---|---|---|
| MMV_PFSPZ-DVI BLOOD STAGE_19_01 - ANALYSIS VERSION | | LISTING 16.2.1.2: ANALYSIS PHASES |

| DURATION<br>(DAYS) | ××× | × × × | × × × | * * * |
|---|---|---|---|---|
| DI START STOP | ddMwMyyyy;hh:mm ddMwMyyyy;hh:mm ddMMMyyyy;hh:mm ddMMMyyyy;hh:mm ddMMMyyyy;hh:mm | | | |
| ANALYSIS<br>PHASE | SCREENING<br>CHALLENGE<br>RESCUE | SCREENING<br>CHALLENGE<br>RESCUE | SCREENING<br>CHALLENGE<br>RESCUE | SCREENING<br>CHALLENGE<br>RESCUE |
| DISCONTINUATION ANALYSIS DATE | ddMMMyyyy | ddMMyyyy | ddMMyyyy | ddMMMyyyy |
| LAST USE OF ANTIMALARIAL TREATMENT | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyyy:hh:mm | ddMMyyyy:hh:mm |
| FIRST USE OF ANTIMALARIAL TREATMENT | ddMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm |
| ET: SAFETY SUBJECT DATETIME OF NUMBER INOCULATION | COHORT 1 XXXXXX ddMMMyyyy;hh:mm | xxxxxx ddMMMyyyy:hh:mm | XXXXXX ddMMMyyyy:hh:mm | COHORI 2 XXXXXX ddMMMyyyyy:hh:mm |
| SET: SAFETY SUBJECT DA NUMBER IN | XXXXX | XXXXXX | XXXXXX | XXXXX |
| ANALYSIS S COHORT | COHORT 1 | | | COHORT 2 |

ETC...

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.1.3: STUDY AND ANTIMALARIAL TREATMENT DISCONTINUATION

ANALYSIS SET: SAFETY

| ECTT CITY | 1 | DATE OF DISCONTINUATION | ر<br>د<br>د | STUDY D | STUDY DISCONTINUATION | ANTIMALARIAL | ANTIMALARIAL TREATMENT DISCONTINUATION |
|---|---|---|---|---|---|---|---|
| | STUDY | L TREATMENT | [1] | TYPE | REASON | TYPE | REASON |
| | OHORT 1 XXXXXX ddMMMyyyy | ddMMMyyyy | × | COMPLETED | | COMPLETED | |
| | ddMMMyyyy<br>ddmmmyyyyy | ddMMMYYYY<br>Admmaterree | × > | COMPLETED | · / >> CES/ HNEZIE ESCETION | COMPLETED | · /vv CGS/ Whatte godation |
| | A & & VINITALIA | | << | DISCONTINCED | PREFERRED TERM | | |
| | COHORT 2 XXXXXX ddMMMyyyy | ddMMMyyyy ddMMMyyyyy | XX | ONGOING | | ONGOING | |

<sup>[1]</sup> NUMBER OF DAYS IN STUDY AT DATE OF DISCONTINUATION, CALCULATED WITH REFERENCE TO THE DATE OF INOCULATION.


# Protocol deviations and eligibility

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.2.1: MAJOR PROTOCOL DEVIATIONS

| ANALYSIS | ANALYSIS SET: SAFETY | TI | | | |
|---|---|---|---|---|---|
| COHORT | SUBJECT<br>NUMBER | TYPE | DEVIATION CLASS | DEVIATION | DEVIATION (SPECIFICATION) |
| COHORT 1 XXXX | ×××× 1 | MAJOR | PROCEDURE DEVIATION | NO COMPLIANCE WITH ASSESSMENT WINDOW NO COMPLIANCE WITH VISIT | PK URINE COLLECTION X-XH POSTDOSE,<br>STARTED XH XXMIN. EARLIER<br>VISIT X DONE X DAY LATER |
| | XXXX | MAJOR | PROCEDURE DEVIATION | SCHEDOLES NO COMPLIANCE WITH ASSESSMENT WINDOW | ECG PXDX XX MIN.POSTDOSE, DONE XX MIN. EARLIER |
| | | | | TO COMPLIANCE WITH VICTURE | EAGLIER FARIER FAURINE COLLECTION X-XH POSTDOSE, STARTED XXMIN. EARLIER VICTH Y DONE Y DAY IARED |
| | XXXX | MAJOR | TREATMENT DEVIATION | NO COMPLIANCE WITH VISIT SCHEDULES NO COMPLIANCE WITH STUDY MED. | MEDICATION XX MIN. INFUSION, DOSE NOT |
| | | MAJOR | PROCEDURE DEVIATION | INITARE NO COMPLIANCE WITH ASSESSMENT WINDOW | PK BLOOD SAMPLING XH POSTDOSE, DONE X MIN. EARLING SAMPLING SAMPLI |
| | | | | NO COMPLIANCE WITH VISIT | ECG XXMIN. FOSIDOSE, DONE XX MIN. EARLIER ECG X.H. POSIDOSE, DONE XX MIN. EARLIER VISIT X. DONE X DAY LATER |
| | XXXX | MAJOR | SELECTION CRITERIA | SCHEDULES<br>SELECTION CRITERIA NOT MET | SELECTION CRITERIA ARE NOT MET (EX03, EX10) |

ETC...


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.2.2: VIOLATIONS ON ELIGIBILITY CRITERIA

ANALYSIS SET: SAFETY

ANSWER YES 0 N 8 9.BODY WEIGHT OF AT LEAST 50 KG AND A BODY MASS INDEX (BMI) OF 19.0 TO 30.0 KG/M2 9.BODY WEIGHT OF AT LEAST 50 KG AND A BODY MASS INDEX (BMI) OF 19.0 TO 30.0 KG/M2 17.PERSONAL HISTORY OF MALARIA CRITERION INCLUSION INCLUSION EXCLUSION TYPE SUBJECT NUMBER XXXX XXXX COHORT 2 COHORT 1 COHORT

NOTE: ONLY VIOLATIONS ARE SHOWN.


MMV\_PfSPZ-DVI Blood Stage\_19\_01

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

ANALYSIS SET: ALL SCREENED SUBJECTS MINUS SAFETY

LISTING 16.2.2.3: NO-INOCULATED SUBJECTS

SUBJECT NUMBER

STUDY TERMINATION REASON

OTHER: PERSONAL REASON
SUBJECT DID NOT FULFILL ALL INCLUSION/EXCLUSION CRITERIA
OTHER: PERSONAL REASON
SUBJECT DID NOT FULFILL ALL INCLUSION/EXCLUSION CRITERIA
SUBJECT DID NOT FULFILL ALL INCLUSION/EXCLUSION CRITERIA
OTHER: BLOOD SAFETY RESULTS
OTHER: BLOOD SAFETY RESULTS
SUBJECT MITHDREW CONSENT 

ETC...


# Demographic and other baseline characteristics

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.4.1: DEMOGRAPHIC DATA

ANALYSIS SET: SAFETY

| COUNTRY RACE ETHNICITY | BELGIUM WHITE HISPANIC OR LATINO BELGIUM WHITE NOT HISPANIC OR LATINO FRANCE WHITE HISPANIC OR LATINO BELGIUM WHITE HISPANIC OR LATINO BELGIUM WHITE HISPANIC OR LATINO FRANCE WHITE NOT HISPANIC OR LATINO FRANCE WHITE HISPANIC OR LATINO FRANCE WHITE HISPANIC OR LATINO FRANCE WHITE NOT HISPANIC OR LATINO |
|---|---|
| COUNTRY | BELGIUM<br>BELGIUM<br>FRANCE<br>BELGIUM<br>BELGIUM<br>FRANCE<br>FRANCE |
| SEX | MALE MALE MALE MALE MALE MALE FEMALE |
| BMI<br>(kg/m²) | ****** |
| WEIGHT<br>(kg) | ***** |
| HEIGHT<br>(cm) | |
| AGE<br>(years) | *** |
| DATE OF<br>SIGNING<br>INFORMED<br>CONSENT | ddmmmyyyy<br>ddmmyyyyy<br>ddmmhyyyy<br>ddmmhyyyy<br>ddmmyyyyy<br>ddmmyyyyy |
| PD | S S S S S K K K K K K K K K K K K K K K |
| SUBJECT<br>NUMBER<br> | 1 XXX X |
| COHORT | COHORT 1 COHORT 2 ETC |

SCREENING HEIGHT, WEIGHT AND BMI ARE LISTED.


SAS DATE AND TIME PAGE X OF Y


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.4.2: SMOKING HISTORY

ANALYSIS SET: SAFETY

SMOKING HABITS

| STOP DATE | ddMMMyyyy | ddMMMyyyy |
|---|---|---|
| START DATE | ddMMMyyyy | ddMMMyyyy<br>ddMMMyyyyy<br>ddMMMyyyyy |
| FREQUENCY | QD<br>QD | 00<br>00<br>00<br>00 |
| QUANTITY<br> | 4 CIGARETTE QD<br>1 CIGARETTE QD | 3 CIGARETTE<br>2 CIGARETTE<br>7 CIGARETTE |
| STATUS | SMOKER<br>EX-SMOKER<br>NON-SMOKER | SMOKER<br>SMOKER<br>EX-SMOKER |
| SUBJECT<br>NUMBER | × | × |
| COHORT | COHORT 1 | COHORT 2<br>ETC |

SAS DATE AND TIME PAGE X OF Y

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

| NG |
|-------------|
| SCREENI |
| ΑT |
| SIGNS |
| VITAL |
| Z |
| CHANGE |
| ORTHOSTATIC |
| ٠.<br>٣ |
| 4. |
| 5.2 |
| 1 |
| ISTING |

LIS

ANALYSIS SET: SAFETY

| | | | | HEART F | HEART RATE (beats/min) | | SYSTOLIC | BLOOD PR | SYSTOLIC BLOOD PRESSURE (mmHg) DIASTOLIC BLOOD PRESSURE | DIASTOL | IC BLOOD PI | RESSURE (mmHg) | (b) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| COHORT | NUMBER | SUBUECT ASSESSMENT<br>TUMBER DATE | USE<br>[1] | SUPINE | SUPINE STANDING CHANGE | ı | SUPINE | SUPINE STANDING CHANGE | <br>CHANGE | SUPINE | SUPINE STANDING CHANGE | CHANGE | ! |
| OHORT 1 | XXX | ddMMyyyy | | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| | XXX | ddMMYYYY | | XXX | XXX | XXX | XXX | XXX | ××× | XXX | XXX | XXX | |
| OHORT 2 | XXX | ddMMMyyyy | | XXX | XXX | XXX | XXX | XXX | ××× | XXX | XXX | XXX | |
| | XXX | ddMMMyyyy | | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| | XXX | ddMMMyyyy | | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| | XXX | ddMMMyyyy | | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| | | ddMMMyyyy | NO | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |

<sup>[1]</sup> NO = SAMPLE NOT USED IN ANALYSIS TABLES AND FIGURES. ORTHOSTATIC CHANGE = VALUE IN SUPINE POSITION - VALUE IN STANDING POSITION.


| MMV_PFSPZ-DVI | BLOOD ST. | MMV_PFSPZ-DVI BLOOD STAGE_19_01 - ANALYSI | KSIS VERSION | | SAS DATE | SAS DATE AND TIME |
|---|---|---|---|---|---|---|
| LISTING 16.2.4 | 1.4: BECK | LISTING 16.2.4.4: BECK DEPRESSION INVENTORY AT SCREENING | NTORY AT SCREENI | DNG | FA | FAGE A OF 1 |
| ANALYSIS SET: SAFETY | SAFETY | | <br> | <br> | | <br> |
| COHORT | SUBJECT<br>NUMBER | SUBJECT ASSESSMENT NUMBER DATETIME | SUICIDAL TOTAL THOUGHTS? (Q9) SCORE | TOTAL<br>SCORE | INTERPRETATION | |
| COHORT 1 | XXX | ddMMMyyyy:hh:mm XXX<br>ddMMMyyyy:hh:mm XXX | XXX | × | NORMAL<br>MILD MOOD DISTURBANCE | |
| COHORT 2 | × | ddMMMyyyy:hh:mm XXX<br>ddMMyyyy:hh:mm XXX<br>ddMMyyyy:hh:mm XXX<br>ddMMMyyyy:hh:mm XXX | XXX<br>XXX<br>XXX | X | NORMAL<br>BORDERLINE CLINICAL DEPRESSION<br>NORMAL<br>NORMAL | |

ETC...


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.4.5: SCREENING LABORATORY TESTS

ANALYSIS SET: SAFETY

A) URINE DRUG SCREEN AND ETHANOL

| OL | RESULT | NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE | NEGATIVE<br>NEGATIVE | |
|---|---|---|---|---|
| | ASSESSMENT DATETIME RESULT | ddwMyyyyy:hh:mm<br>ddwMyyyy;hh:mm<br>ddwMyyyy;hh:mm<br>ddwMyyyy;hh:mm<br>ddwMyyyy;hh:mm | ddMMMyyyy:hh:mm<br>ddMMyyyyy:hh:mm | |
| NING | RESULT | NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE | NEGATIVE<br>NEGATIVE | |
| DRUG SCREENING | ASSESSMENT DATETIME RESULT | ddMMMyyyy:hh:mm<br>ddMMMyyyy:hh:mm<br>ddMMMyyyy:hh:mm<br>ddMMMyyyy:hh:mm<br>ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm<br>ddMMyyyyy:hh:mm | |
| | SUBJECT ANALYSIS<br>NUMBER VISIT | SCREENING<br>DAY -1<br>SCREENING<br>DAY -1<br>SCREENING<br>SCREENING | SCREENING<br>DAY -1 | |
| | | × × ××<br>× × ×× | XXX | |
| | COHORT | СОНОКТ 1 | COHORT 2 | ETC |

되

B) VIRAL SEROLOGY AT SCREENING

| X 1 | | |
|---|---|---|
| HIV SEROLOGY | NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE | NEGATIVE<br>NEGATIVE |
| EPSTEIN BARR<br>VIRUS<br>ANTIBODY | NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE | NEGATIVE<br>NEGATIVE |
| CYTOMEGALOVIRUS<br>ANTIBODY | NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE | NEGATIVE<br>NEGATIVE |
| HEPATITIS E<br>VIRUS<br>ANTIBODY | NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE | NEGATIVE<br>NEGATIVE |
| HEPATITIS C<br>VIRUS<br>ANTIBODY | NEGATIVE NEGATIVE NEGATIVE NEGATIVE NEGATIVE NEGATIVE | NEGATIVE<br>NEGATIVE |
| HEPATITIS B<br>SURFACE<br>ANTIGEN | NEGATIVE NEGATIVE NEGATIVE NEGATIVE NEGATIVE | NEGATIVE<br>NEGATIVE |
| HEPATITIS A<br>VIRUS<br>ANTIBODY | POSITIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE<br>NEGATIVE | NEGATIVE<br>NEGATIVE |
| SUBJECT ASSESSMENT NUMBER DATETIME | ddMMMyyyy;hh;mm<br>ddMMMyyyy;hh;mm<br>ddMMMyyyy;hh;mm<br>ddMMMyyyy;hh;mm<br>ddMMMyyyy;hh;mm | ddMMMyyyy:hh:mm<br>ddMMMyyyy:hh:mm |
| SUBJECT<br>NUMBER | × | XXX |
| COHORT | сонокт 1 | COHORT 2 |

ETC...

| MMV_PFSPZ-DVI BLOOD STAGE_19_01 - ANALYSIS | STAGE_19 | _01 - ANALYSIS VERSION | | | SAS DATE AND TIME | CME |
|---|---|---|---|---|---|---|
| LISTING 16.2.4.6: PREGNANCY TESTS | REGNANCY | | | | | - |
| ANALYSIS SET: SAFETY | | | | | | !<br>! |
| COHORT | SUBJECT<br>NUMBER | ANALYSIS VISIT | ASSESSMENT<br>DATETIME | SPECIMEN TYPE | HCG RESULT | |
| COHORT 1 | × × × | SCREENING DAY -1 END OF STUDY SCREENING | ddMMMyyyy;hh:mm<br>ddMMMyyyy;hh:mm<br>ddMMMyyyy;hh:mm<br>ddMMMyyyy;hh:mm | SERUM<br>URINE<br>SERUM<br>SERUM | XX<br>NEGATIVE<br>XX<br>XX<br>NEGATIVE | |
| ETC | | | | | 7,115,011 | |

SAS DATE AND TIME PAGE X OF Y

ANALYSIS SET: SAFETY

| RESULT | NEGATIVE | NEGATIVE | NEGATIVE | NEGATIVE | |
|---|---|---|---|---|---|
| ASSESSMENT<br>DATETIME | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | |
| ANALYSIS VISIT | SCREENING | DAY 9 | SCREENING | DAY 9 | |
| SUBJECT | XXX | | XXX | | |
| COHORT | COHORT 1 | | | | ETC |


SAS DATE AND TIME PAGE X OF Y

COMMENTS

END DATE

START DATE

VERBATIM

PREFERRED TERM

## Medical history and concomitant diseases 4.1.4

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.4.8: MEDICAL HISTORY

SYSTEM ORGAN CLASS SUBJECT NUMBER XXXANALYSIS SET: SAFETY COHORT 1 COHORT

XXXXXXXXXXXXXXX ddMMMyyyy ddMMMyyyy ddMMMyyyy ddMMMyyyy ddMMMyyyy ddMMMYYYY ddMMMYYYY ddMMMYYYY ddMMMyyyy ddMMYYYYDIARRHOEA ABDOMINAL HERNIA ABSCESES DEPRESSION INSOMNIA GASTROONTESTINAL DISORDERS DIARRHOEA ABDOMINAL HERNIA INFECTIONS AND INFESTATIONS ABSCESS DEPRESSION INSOMNIA

PSYCHIATRIC DISORDERS PSYCHIATRIC DISORDERS

XXX XXX

ETC...


| MMV_PFSPZ-DVI BLOOD STAGE_19_01 - ANALYSIS | GE_19_01 · | - ANALYSIS VERSION | | | | SAS DATE AND TIME |
|---|---|---|---|---|---|---|
| LISTING 16.2.4.9: CONCOMITANT DISEASES | MITANT DI: | SEASES | | | | PAGE X OF Y |
| ANALYSIS SET: SAFETY | <br> | | | | 1<br>1 | |
| COHORT | SUBJECT<br>NUMBER<br> | SYSTEM ORGAN CLASS | PREFERRED TERM | VERBATIM | START DATE | COMMENTS |
| COHORT 1 | XXX | GASTROINTESTINAL DISORDERS | DIARRHOEA | DIARRHOEA | ddMMMyyyy | |
| | | ABDOMINA INFESTATIONS ABSCESS | ABDOMINAL HERNIA<br>ABSCESS | ABDOMINAL HERNIA<br>ABSCESES | ddMMMyyyy<br>ddMMMyyyy | |
| | XXX | PSYCHIATRIC DISORDERS | DEPRESSION | DEPRESSION | ddMMYYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXX | PSYCHIATRIC DISORDERS | INSOMNIA | INSOMNIA | ddMMMyyyy | |

ETC...


### Prior and concomitant therapies 4.1.5

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

SAS DATE AND TIME PAGE X OF Y

LISTING 16.2.4.10: PRIOR AND CONCOMITANT THERAPIES

ANALYSIS SET: SAFETY

COHORT 1

COMMENTS HIGH BLOOD PRESSURE (MEDICAL HISTORY) AE (SEQ X): PREFERRED TERM (SEQ X): PREFERRED TERM AE (SEQ X): PREFERRED TERM CONTRACEPTIVE CONTRACEPTIVE CONTRACEPTIVE START DATE END DATE DOSE, FREQ, ROUTE INDICATION ΑE PO PO PO T.I.D. ddMMMyyyy 375 mg T.I.D. ddMMMyyyy 250 mg T.I.D. ddMMMyyyy 150 mg 1X IM mg 1X IM mg 1X IM SCREENING DIHYDROPYRIDINE DERIVATIVES ddMMMyyyy ddMMMyyyy 10 mg QD PO ddMMMyyyy 1000 mg 150 ddMMMyyyy 150 ----THERAPY----ONGOING ddMMMyyyy ddMMMyyyy ddMMMyyyy ddMMMyyyy CHALLENGE PROGESTOGENS
MEDROXYPROGESTERONE ACETATE
RESCUE
PROGESTOGENS MEDROXYPROGESTERONE ACETATE SCREENING PROGESTOGENS MEDROXYPROGESTERONE ACETATE PENICILLINS WITH EXTENDED AMASE INHIBITORS AUGMENTIN /00756801/ ATC CLASS (LEVEL 4) GENERIC TERM PARACETAMOL AMOXICILLIN AMLODI PINE SPECTRUM ANILIDES SUBJECT ANALYSIS NUMBER PHASE CHALLENGE RESCUE XXXX XXXX ETC...

COHORT 2

ETC...

Mock Tables, Listings and Figures

SAS DATE AND TIME PAGE X OF Y

MMV\_PfSPZ-DVI Blood Stage\_19\_01

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.4.11: ANTIMALARIAL TREATMENT

ANALYSIS SET: SAFETY

| | 20/120 MG/TABLET | 20/120 MG/TABLET | 20/120 MG/TABLET | 20/120 MG/TABLET | 20/120 MG/TABLET | 20/120 MG/TABLET | 20/120 MG/TABLET | 250/100 MG/TABLET |
|---|---|---|---|---|---|---|---|---|
| NUMB | <br> | ×× | ×× | ×× | ×× | ×× | ×× | ×× |
| G DATETIME | ddMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMVvvvv:hh:mm |
| ENER | RIAMET | RIAMET | RIAMET | RIAMET | RIAMET | RIAMET | RIAMET | MAT, ARONE |
| DAY IN<br>STUDY[1] | 12 | 13 | 14 | 13 | 14 | 15 | 18 | 18 |
| SUBJECT DAY IN NUMBER STUDY[] | XXXX | | | XXXX | | | XXXX | |
| COHORT | COHORT 1 | | | | | | | |

ETC...


<sup>[1]</sup> NUMBER OF DAYS IN STUDY AT DATE OF ANTIMALARIAL TREATMENT, CALCULATED WITH REFERENCE TO THE DATE OF INOCULATION.

SAS DATE AND TIME PAGE X OF Y

#### Comments 4.1.6

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.4.12: COMMENTS

ANALYSIS SET: SAFETY

| COHORT | SUBJECT<br>NUMBER | REFERENCE | <br> -<br> -<br> -<br> -<br> -<br> - | COMMENT |
|---|---|---|---|---|
| COHORT 1 | XXXX | LBSEQ: XX | ×× | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| COHORT 2 | XXXX<br>XXXX | EGSEQ: XX<br>LBSEQ: XX<br>EGSEQ: XX | * * * * * | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

ETC...


MMV\_PfSPZ-DVI Blood Stage\_19\_01

# Exposure to challenge agent

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.5.1: EXPOSURE TO CHALLENGE AGENT

ANALYSIS SET: SAFETY

| COHORT | SUBJECT<br>NUMBER | SUBJECT PÍSPZ CHALLENGE<br>NUMBER DATETIME | 1<br>1<br>1<br>1<br>1<br>1<br>1<br>1 | ADMINISTRATION<br>ROUTE | FORMULATION |
|---|---|---|---|---|---|
| COHORT 1 | X X X X X X X X X X X X X X X X X X X | ddMMyyyy;hh:mm<br>ddMMyyyy;hh:mm<br>ddMMyyyy;hh:mm<br>ddMMyyyy;hh:mm<br>ddMMyyyy;hh:mm | × | XXXXXXX<br>XXXXXXX<br>XXXXXXXX | XXXXXXXX<br>XXXXXXXX<br>XXXXXXXXX |

ETC...


SAS DATE AND TIME PAGE X OF Y


## **PHARMACODYNAMICS**

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.6.1: PARASITAEMIA

COHORT 1

ANALYSIS SET: PD

RESULT (p/mL) [3] **GPCR** \* USE [2] ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm SAMPLE DATETIME DAY [1] DAY 8
DAY 9
DAY 10
DAY 11
DAY 12
DAY 12
DAY 13 ANALYSIS VISIT BASELINE DAY 7 FIRST ANTIMALARIAL TREATMENT DATETIME ddMMMyyyy:hh:mm m-PD YES SUBJECT XXXX

ddMMMyyyy:hh:mm UNSCHEDULED DAY 21

ETC...

0 N

ddMMyyyy:hh:mm

ddMMyyyy:hh:mm ddMMyyyy:hh:mm

UNSCHEDULED

<sup>[1]</sup> DAY VS. INOCULATION, DAYS ON WHICH ANTIMALARIAL TREATMENT IS TAKEN ARE FLAGGED (\*). [2] NO = NOT USED IN ANALYSIS TABLES AND FIGURES. [3] POSITIVE QPCR RESULTS (250 PARASITES PER ML BLOOD) ARE FLAGGED (\$).


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.6.2: PARASITAEMIA ENDPOINTS

ANALYSIS SET: PD

COHORT 1

| TIME TO PARASITE<br>CLEARENCE (DAYS) | *** |
|---|---|
| PARASITAEMIA<br>AT FIRST DOSE<br>OF RIAMET TI<br>(PARASITES/ML) CI | ××××<br>×××××<br>××××××××××××××××××××××××××× |
| O<br>DOSE<br>MET | *** |
| PARASITAEMIA TIME TA 25000 FIRST PARASITES OF RIA! (PARASITES/ML) (DAYS) | ××××<br>××××<br>- |
| TIME TO >5000 PARASITES ) (DAYS) [1] | ×××× |
| PARASITAEMIA TIME TO AT FIRST 25000 POSITIVE PCR PARASITES (PARASITES/ML) (DAYS)[1] | ××××<br>××××<br>××××× |
| TIME TO POSITIVE PARASITAEMIA (DAYS) | × × × × |
| m-PD | YES<br>YES<br>NO<br>YES |
| SUBJECT<br>NUMBER | XXXX<br>XXXX<br>XXXX |

<sup>[1]</sup> ABSENCE OF EVENT IS FLAGGED (°). POSITIVE PARASITAEMIA IS DEFINED AS QPCR OUTCOME 2250 PARASITES PER ML BLOOD. PARASITE CLEARANCE IS DEFINED AS QPCR OUTCOME BELOW THE LIMIT OF QUANTIFICATION (<50 PARASITES PER ML BLOOD).

ETC...


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

SAS DATE AND TIME PAGE X OF Y

LISTING 16.2.6.3: BLOOD-STAGE PARASITE CLEARANCE PROFILE: ITERATION PROCESS TO DETERMINE THE OPTIMAL LOG-LINEAR MODEL

ANALYSIS SET: PD

COHORT 1

| 1 | | |
|---|---|---|
| OPTIMAL<br>FLAG<br>[3] | YES | S<br>El |
| P-VALUE<br>[2]<br> | X | × |
| LOG10PRR48<br>(95% CI)<br> | (XX;XX)<br>(XX;XX)<br>(XX;XX)<br>(XX;XX) | (XX;XX)<br>(XX;XX)<br>(XX;XX)<br>(XX;XX) |
| LOG1<br>(95% | $\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}$ | $\overset{\times}{\times}\overset{\times}{\times}\overset{\times}{\times}\overset{\times}{\times}\overset{\times}{\times}$ |
| TIME<br>ESTIMATE<br>(95% CI) | (XX;XX)<br>(XX;XX)<br>(XX;XX) | (XX;XX)<br>(XX;XX)<br>(XX;XX)<br>(XX;XX)<br>(XX;XX) |
| TIIM<br>EST<br>(95 | $\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}$ | $\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}\stackrel{\times}{\times}$ |
| ITERATION | L 0 6 4 | 1 2 6 4 5 9 |
| USE<br>[1] | X E S | YES |
| m-PD | YES | S<br>H<br>X |
| SUBJECT<br>NUMBER | XXXX | ×××× |

<sup>[1]</sup> YES = SUBJECT INCLUDED IN THE DESCRIPTIVE STATISTICS OF DERIVED PARAMETERS OF THE LOG-LINEAR MODEL FOR PARASITE CLEARANCE. A SUBJECT IS INCLUDED WHEN THE OPTIMAL LOG-LINEAR REGRESSION MODEL P-VALUE <a href="https://document.org/linear/nobel">0.001</a>.

[2] OVERALL MODEL P-VALUE BASED ON F-TEST.

[3] OPTIMAL MODEL IS DEFINED BY THE MINIMUM OVERALL MODEL P-VALUE.

#### SAFETY

#### Adverse events 4.3.1

MMV PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

SAS DATE AND TIME PAGE X OF Y

DUR [14]

 $\overset{\times}{\underset{\times}{\times}}\overset{\times}{\underset{\times}{\times}}\overset{\times}{\underset{\times}{\times}}$ 

XXX

LISTING 16.2.7.1: ADVERSE EVENTS

ANALYSIS SET: SAFETY

COHORT

ONSET [13] ONSET [12] [11] RX ACT [10] REL ACT ACT [7] [8] [9] REL [6] REL [5] SI [4] TOX [3] OUT [2] STOP DATETIME -- ADVERSE EVENT START DATETIME PREFERRED TERM (VERBATIM) [1] ANALYSIS PHASE SUBJECT XXXX

\* \* \* \* \* NO YES NO NO 0 0 0 0 0 0 0 0 9 9 9 9 0 0 0 0 0 0 0 0 NO NO YES NO GR1 1 GR1 1 GR2 ' REC REC REC ddMMyyyy:hh:mm ddMMyyyy:hh:mm ddMMyyyy:hh:mm ONGOING ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMyyyy:hh:mm ddMMMyyyy:hh:mm VEIN WALL HYPERTROPHY (XXXXXXXX) PULMONARY EMBOLISM (XXXXXXXXX) \* TINEA PEDIS (XXXXXXXXX) PAIN NOS (XXXXXXXXX) SCREENING NONE CHALLENGE XXXX

ddMMMyyyy:hh:mm UNKNOMN PAIN IN FOOT (XXXXXXXX) ! DIARRHOEA NOS (XXXXXXXXX) VOMITING NOS (XXXXXXXX) DIZZINESS (XXXXXXXXX) NONE SCREENING NONE CHALLENGE

ETC...

 $\overset{\times}{\times}\overset{\times}{\times}$ XXX  $\overset{\times}{\times}\overset{\times}{\times}$ XXX NO NO YES NO NO NO PER NO NO NO PER NO NO NO PER YES ON ON YES 0 N YES YES 0 N YES NO NO NO MMMyyyyy
ddMMMyyyy;hh:mm REC GR1 N
ddMMMyyyy;hh:mm REC GR1 N
ddMMMyyyy;hh:mm REC GR1 N GR3 GR1 1 ddMMyyyy:hh:mm ddMMyyyy:hh:mm


<sup>[1]</sup> SAES ARE FLAGGED WITH \*. AES FOR WHICH ANOTHER ACTION IS TAKEN ARE FLAGGED WITH (!).

[2] OUTCOME: REC = RECOVERED/RESOLVED; RECI = RECOVERING/RESOLVING; NREC = NOT RECOVERED/NOT RESOLVED; RECS = RECOVERED WITH SEQUELAE;

[2] OUTCOME: REC = RECOVERED WITH SEQUELAE;

[3] AE TOXICITY: GRI = GRADE 1-MILD; GR2 = GRADE 2-MODERATE; GR3 = GRADE 3-SEVERE; GR4 = GRADE 4-LIFE-THREATENING; GR5 = GRADE 5-DEATH.

[4] SI: ADVERSE EVENT OF SPECIAL INTEREST.

[5, 6, 7] RELATIONSHIP TO PESPZ INOCULUM, RIAMET, MALARONE: NO=NOT RELATED/NOT SUSPECTED; NO=NO ACTION TAKEN; UNK=UNKNOWN; NAP=NOT APPLICABLE.

[8, 9, 10] ACTION TAKEN TOWARDS PISPZ INOCULUM, RIAMET, MALARONE: PER=PERMANENTLY DISCONTINUED; NO=NO ACTION TAKEN; UNK=UNKNOWN; NAP=NOT APPLICABLE.

[11] RX: CONCOMITANT THERAPY STARTED BECAUSE OF THE AE.

<sup>[12]</sup> ONSET: DAY OF ONSET VERSUS FIRST PESPZ INOCULATION, OR TIME OF ONSET IF ON DAY 1. [13] ONSET: DAY OF ONSET VERSUS START OF THE ANALYSIS PHASE, OR TIME OF ONSET IF ON DAY OF START OF THE ANALYSIS PHASE. [14] DURATION: DURATION (DAYS) OF THE INDIVIDUAL EVENT.

MMV PFSPZ-DVI BLOOD STAGE 19 01 - ANALYSIS VERSION

LISTING 16.2.7.2: SERIOUS ADVERSE EVENTS

ANALYSIS SET: SAFETY

COHORT

DUR [14] >XXX XXX XXX XXX [13] X X X XXXXXX ONSET [12] XXX X X X XXX EXX [11] YES 9 N 9 N [10] Q N 0 N 0N ACT [9] 0 N ON. 0N REL ACT [7] [8] 0 0 0 8 YES 0 0 0 0 0 0 YES REL [6] 0N 0 N REL [5] YES ON. 0 N NO NO YES [4] 0N OUT TOX [2] GR1 GR1 GR2 GR1 REC REC REC REC REASON [1] ddMMMyyyy;hh:mm ddMMMyyyy;hh:mm OMI adwwwyyyy:hh:mm ONGOING HOS ddMMMyyyy:hh:mm ddWMMyyyy:hh:mm OMI ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm OMI START DATETIME STOP DATETIME -- ADVERSE EVENT VEIN WALL HYPERTROPHY (XX) PULMONARY EMBOLISM (XXXXX) PREFERRED TERM (VERBATIM) VOMITING NOS (XXXXXXXX) PAIN NOS (XXXXXXXXX) CHALLENGE ANALYSIS RESCUE PHASE SUBJECT NUMBER XXXX XXXX

ETC...

[1] DTH = RESULTS IN DEATH; LIF = LIFE-THREATENING; HOS = REQUIRES OR PROLONGS HOSPITALISATION; DIS = RESULTS IN DISABILITY; CON = CONGENITAL

ANOMALY; OMI = OTHER MEDICAL IMPORTANT AE.

[2] OUTCOME: REC = RECOVERED/RESOLVED; RECI = RECOVERING/RESOLVING; NREC = NOT RECOVERED/NOT RESOLVED; RECS = RECOVERED WITH SEQUELAE; = FATAL; UNK = UNKNOWN. FAT

[3] AE TOXICITY: GR1 = GRADE 1-MILD; GR2 = GRADE 2-MODERATE; GR3 = GRADE 3-SEVERE; GR4 = GRADE 4-LIFE-THREATENING; GR5 = GRADE 5-DEATH.
[4] SI: ADVERSE EVENT OF SPECIAL INTEREST.
[5,6,7] RELATIONSHIP TO PESPZ INOCULUM, RIAMET, MALARONE: NO=NOT RELATED/NOT SUSPECTED; YES=RELATED/SUSPECTED; NAP=NOT APPLICABLE.
[8,9,10] ACTION TAKEN TOWARDS PESPZ INOCULUM, RIAMET, MALARONE: PER=PERMANENTLY DISCONTINUED; NO=NO ACTION TAKEN; UNK=UNKNOWN; NAP=NOT APPLICABLE.
[11] RX: CONCOMITANT THERAPY STARTED BEGAUSE OF THE AE.
[12] ONSET DAY OF ONSET VERSUS START OF THE ANALYSIS PHASE, OR TIME OF ONSET IF ON DAY 1.
[13] ONSET: DAY OF ONSET VERSUS START OF THE ANALYSIS PHASE, OR TIME OF ONSET IF ON DAY OF START OF THE ANALYSIS PHASE.


# Programmer note: repeat listing 16.2.7.1 for:

LISTING 16.2.7.3: FATAL ADVERSE EVENTS

LISTING 16.2.7.4: ADVERSE EVENTS FOR WHICH THE STUDY WAS DISCONTINUED

LISTING 16.2.7.5: ADVERSE EVENTS FOR WHICH THE ANTIMALARIAL TREATMENT WAS DISCONTINUED

LISTING 16.2.7.6: ADVERSE EVENTS AFTER ADMINISTRATION OF ANTIMALARIAL TREATMENT


MMV\_PfSPZ-DVI Blood Stage\_19\_01

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.7.7: ADVERSE EVENTS FOR WHICH ANOTHER ACTION IS TAKEN

ANALYSIS SET: SAFETY

COHORT 1

OTHER ACTION TAKEN PREFERRED TERM (VERBATIM) SUBJECT ANALYSIS NUMBER PHASE RESCUE XXXX XXXX ETC...


| MMV_PFSPZ-DVI BLOOD STAGE_19_01 | _01 - ANALYSIS VERSION | | | | SAS DATE AND | TIM |
|---|---|---|---|---|---|---|
| LISTING 16.2.7.8: ADVERSE EVE | EVENTS: CODING INFORMATION | | | | PA | PAGE X OF Y |
| ANALYSIS SET: SAFETY | | | <br> | | <br> | |
| COHORT 1 | | | | | | |
| SYSTEM ORGAN CLASS | HIGH LEVEL GROUP TERM | HIGH LEVEL TERM | PREFERRED TERM | LOWER LEVEL TERM VERBATIM | VERBATIM<br> | SUBJECT<br>NUMBER |
| GASTROINTESTINAL DISORDERS | DENTAL AND GINGIVAL CONDITIONS | DENTAL AND PERIODONTAL INFECTIONS AND INFLAMMATIONS | DENTAL CARIES | CARIES DENTAL | CARIES DENTAL | XXX |
| | | DENTAL DISORDERS NEC | TOOTH DISORDER | TOOTH DISORDER | TOOTH DISORDER | XXX |
| | GASTROINTESTINAL MOTILITY AND DEFAECATION | DIARRHOEA (EXCL<br>INFECTIVE) | DIARRHOEA | DIARRHOEA | DIARRHEA | XXX |
| | 0 NO | | | LOOSE STOOLS | LOOSE STOOLS | X |
| INFECTIONS AND INFESTATIONS | INFESTATIONS - PATHOGEN | UPPER RESPIRATORY TRACT | NASOPHARYNGITIS | COMMON COLD | COMMON COLD | XXX |
| | ONSFECIFIED | INFECTIONS | | | | XXX<br>XXX<br>XXX |
| | VIRAL INFECTIOUS<br>DISORDERS | VIRAL INFECTIONS NEC | GASTROENTERITIS<br>VIRAL | GASTROENTERITIS<br>VIRAL | GASTROENTERITIS<br>VIRAL | XXX |
| BTC | | | VIRAL UPPER<br>RESPIRATORY<br>TRACT INFECTION | UPPER<br>RESPIRATORY<br>TRACT INFECTION<br>VIRAL NOS | UPPER<br>RESPIRATORY<br>TRACT<br>INFECTION VIRAL | XXX |


## 4.3.2 Physical examinations

| MW_PFSPZ-DVI | BLOOD SI | MMV_PFSPZ-DVI BLOOD STAGE_19_01 - ANALYSIS | ALYSIS VERSION | | SAS D | SAS DATE AND TIME |
|---|---|---|---|---|---|---|
| ISTING 16.2.7 | 7.9: PHYS | LISTING 16.2.7.9: PHYSICAL EXAMINATIONS | ONS ABNORMALITIES | | | |
| ANALYSIS SET: SAFETY | SAFETY | <br> | <br> | | | <br> |
| COHORT | SUBJECT<br>NUMBER | SUBJECT ANALYSIS<br>NUMBER VISIT | ASSESSMENT<br>DATETIME | CRF BODY SYSTEM | DESCRIPTION (VERBATIM) | CLINICAL<br>SIGNIFICANT |
| сонокт 1 | XXXXXX<br>XXXXXX<br>XXXXXX | DAY -1<br>DAY -1<br>DAY 10<br>END OF STUDY<br>DAY 10 | ddMMyyyy;hh:mm<br>ddMMyyyyy;hh:mm<br>ddMMyyyyy;hh:mm<br>ddMMyyyy;hh:mm<br>ddMMyyyy;hh:mm | EARS, NOSE & THROAT MUSCULOSKELETAL SKIN MUSCULOSKELETAL MUSCULOSKELETAL MUSCULOSKELETAL MUSCULOSKELETAL | ANGINA (NOT TREATED) BACK PAIN SCARS (UPPER THORAX) CNS MOVEMENT-PAIN + CREPITATIO IN BOTH KNEES CNS HIGH MUSCULAR TENSION (NECK) MUSC. TENSION SHOULDER-NECK-MUSC. (NCS) | NO<br>NO<br>NO<br>NO<br>NO |
| ETC | | | | | | |

ONLY ABNORMALITIES ARE SHOWN.


SAS DATE AND TIME PAGE X OF Y

## Clinical laboratory evaluation 4.3.3

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.8.1: LABORATORY TEST RESULTS FOR SUBJECTS WITH ABNORMAL VALUES

ANALYSIS SET: SAFETY

COHORT 1 SUBJECT NUMBER (SEX) = XXXXXXXXX (MALE)

| LABORATORY TEST (UNIT) | ANALYSIS<br>PHASE<br> | ANALYSIS<br>VISIT<br> | SAMPLE<br>DATETIME | USE<br>[1] RESULT<br> | CHG<br>[2] | A<br>NORMAL RANGE [<br> | ABN FAS CSA<br>[3] TED [4] | COMMENT |
|---|---|---|---|---|---|---|---|---|
| TEST 1 (UNIT) | SCREENING | SCREENING<br>DAY -1 | ddMMMyyyy:hh:mm | ×× | | XX-XX<br>XX-XX | YES NO | ********** |
| | CHALLENGE | DAY X | ddMMyyyy:hh:mm | × | × > | H XX-XX | Y ES | |
| | | DAY X | ddMMyyyy:hh:mm | XXX | ×× | | XES | |
| | RESCUE | DAY X | ddMMMyyyy:hh:mm | XX | XX | XX-XX | YES NO | |
| | | DAY X | ddMMMyyyy:hh:mm | XX | X | XX-XX | YES NO | |
| | | DAY X | ddMMMyyyy:hh:mm | XX | X | XX-XX | YES NO | |
| | | DAY X | ddMMMyyyy:hh:mm | ×× | × | XX-XX | NO NO | |
| TEST 2 (UNIT) | SCREENING | SCREENING | ddMMyyyy:hh:mm | XX | | XX-XX | YES NO | |
| | | DAY -1 | ddMMMyyyy:hh:mm | XX | | XX-XX | YES NO | |
| | CHALLENGE | DAY X | ddMMMyyyy:hh:mm | XX | X | XX-XX | YES NO | |
| | | DAY X | ddMMMyyyyy:hh:mm | NO XX | XX | XX-XX | YES NO | |
| | | DAY X | ddMMyyyy:hh:mm | ×× | XX | XX-XX | YES NO | |
| ETC | | | | | | | | |

<sup>[1]</sup> NO = SAMPLE NOT USED IN ANALYSIS TABLES AND FIGURES.
[2] CHANGE FROM BASELINE VALUE.
[3] ABNORMALITY: H = ABNORMALLY HIGH VALUE / L = ABNORMALLY LOW VALUE COMPARED TO THE NORMAL RANGE.
[4] SAMPLE WITH CLINICALLY SIGNIFICANT ABNORMALITIES (CRF DATA).

SAS DATE AND TIME PAGE X OF Y

## Vital signs 4.3.4

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.9.1: VITAL SIGNS RESULTS FOR SUBJECTS WITH ABNORMAL VALUES

ANALYSIS SET: SAFETY

COHORT 1

| (kg) | CHG ABN<br>[3] [4] | | > | ~ | > | > | ~ | > | > | > | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| WEIGHT | ST C | ×× | XX XX | | XX | | | | | | |
| TEMPERATURE (°C) WEIGHT (kg) | ABN<br>[4] | ×× | | | H | H | H | | | | |
| TEMPERATI | | × × × × | | | x.x x.x | | | | | x.x x.x | |
| HEART RATE (bpm) | ABN<br>[4] | ~ ~ ~ | ī | | | | | | | | |
| HEART F | | ×× | XX XX | | XX XX | | | | | | |
| SUPINE<br>DBP (mmHg) | 4 J | | | | XX | | | | | | |
| | TEST<br>RESULT | ×× | ×× | XX | ×× | ×× | ×× | ×× | ×× | XX | |
| SUPINE<br>SBP (mmHg) | CHG<br>[3] | | XX | XX | XX | XX | XX | XX | XX | XX | |
| & & & | CSA TEST<br>[2] RESULT | ×× | NO XX | XX | XX | XX | XX | XX | XX | XX | |
| | USE<br>[1] | | | | ON | | | | | | |
| | VITAL SIGN<br>DATETIME | ddMMyyyy:hh:mm<br>ddMMyyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | |
| | ANALYSIS<br>VISIT | SCREENING<br>DAY -1 | BASELINE | TIME POINT 4 | TIME POINT 5 | SCREENING | DAY -1 | BASELINE | TIME POINT 4 | TIME POINT 5 | |
| | SUBJECT ANALYSIS<br>NUMBER PHASE | SCREENING | CHALLENGE | | | SCREENING | | CHALLENGE | | | |
| | SUBJECT<br>NUMBER | XXXX | | | | XXXX | | | | | ETC |


<sup>[1]</sup> NO = NOT USED IN ANALYSIS TABLES AND FIGURES.
[2] CLINICALLY SIGNIFICANT ABNORMALITY (CRF DATA).
[3] CHANGE FROM BASELINE VALUE.
[4] ABNORMALITY: H = ABNORMALLY HIGH VALUE / L = ABNORMALLY LOW VALUE COMPARED TO THE NORMAL RANGE.

SAS DATE AND TIME PAGE X OF Y

## 4.3.5

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.10.1: ECG RESULTS FOR SUBJECTS WITH ABNORMAL VALUES

ANALYSIS SET: SAFETY

COHORT 1 SUBJECT NUMBER (SEX) =XXXXXXXX (MALE)

| | COMMENT/MORPHOLOGY | | | | XXXXXXXX | | | | | | | XXXXXXXXXXXXX | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (S) | ABN [4] | | | | | | | | | | Ή | Η | н | н |
| QRS (ms) | CHG<br>[3] | - | | | | | | | | | X | XX | XX | × |
| <br> | ABN TEST<br>[4] RESULT | | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | ××× | XXX | XXX |
| (S) | | i<br>¦ | | | | | | | | | H | H | H | Ξ |
| PR (ms) | CHG | }<br>! | | | | | | | | | XX | XX | XX | × |
| | TEST<br>RESULT | | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| (mdq) | ABN<br>[4] | | ⊣ | П | П | П | | | | | П | Ц | П | П |
| RATE | CHG<br>[3] | | | | | | | | | | XXX | XXX | XXX | XXX |
| HEART RATE (bpm) | TEST<br>RESULT | | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | CSA<br>[2] | - | NO<br>NO | ON | NO<br>No | NO | | | | | ON | NO | NO | NO |
| | USE<br>[1] | - | ON<br>N | ON | NO<br>NO | | ON | ON | ON | | ON | ON | ON | |
| | : ECG DATETIME | | ddMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMMyyyy:hh:mm | ddMMyyyy:hh:mm |
| | ECG<br>TRIPLET | | ECG 1 | ECG 2 | ECG 3 | MEAN | ECG 1 | ECG 2 | ECG 3 | MEAN | 3 ECG 1 | ECG 2 | ECG 3 | MEAN |
| | ANALYSIS<br>VISIT | | SCREENING | | | | BASELINE | | | | TIME POINT | ECG | | |
| | ANALYSIS<br>PHASE | | SCREENING | | | | CHALLENGE | | | | | | | |

ETC...


<sup>[1]</sup> NO = NOT USED IN ANALYSIS TABLES AND FIGURES.
[2] CLINICALLY SIGNIFICANT ABNORMALITY (CRF DATA).
[3] CHANGE FROM BASELINE VALUE.
[4] ABNORMALITY: H = ABNORMALLY HIGH VALUE / L = ABNORMALLY LOW VALUE COMPARED TO THE NORMAL RANGE.

| SAS | |
|--------------------|---|
| VERSION | |
| ANALYSIS . | |
| I | |
| 19 01 | 1 |
| STAGE | |
| PFSPZ-DVI BLOOD ST | |
| PFSPZ-DVI | |
| PFSP2 | ı |

| MMV_PESPZ-DV. | I BLOOD STA | 4GE_19_01 | MMV_PFSPZ-DVI BLOOD STAGE_19_01 - ANALYSIS VERSION | NO | | | | | | | | | | SAS D | SAS DATE AND | D TIME |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| LISTING 16.2. | .10.1: ECG | RESULTS 1 | LISTING 16.2.10.1: ECG RESULTS FOR SUBJECTS WITH ABNORMAL VALUES | ABNO | RMAL \ | ALUES | | | | | | | | | 1000 | |
| ANALYSIS SET: SAFETY | SAFETY | <br> | | <br> | <br> | <br> | <br> | <br> | <br> | ;<br> <br> | <br> | i<br> <br> | <br> | <br> | <br> | <br> |
| COHORT 1<br>SUBJECT NUMBER (SEX) = XXXXXXXX (MALE) | IR (SEX) = | XXXXXXX | (MALE) | | | | | | | | | | | | | |
| | | | | | | | QT (ms) | | | Ö | QTcB (ms) | ( ) | | OTCF ( | (ms) | |
| ANALYSIS AN | ANALYSIS<br>VISIT | ECG | ECG DATETIME | USE<br>[1] | CSA I | TEST<br>RESIII.T ABN | CHG | ABN | TEST | ABN | CHG | ABN | TEST | ABN C | CHG | A<br>N<br>N |
| | | | | 7 | | | : | | | | | | | | ! | 1 |
| SCREENING SCREENING | CREENING | ECG 1 | ddMMMyyyy:hh:mm | ON | NO | H XX | | | XXX | н | | | XXX | н | | |
| | | ECG 2 | ddMMMyyyy:hh:mm | NO | NO | H XXX | | | XXX | Ή | | | XXX | H | | |
| | | ECG 3 | ddMMMyyyy:hh:mm | NO | NO | H XX | | | XXX | Ή | | | XXX | H | | |
| | | MEAN | ddMMMyyyy:hh:mm | | NO | H XX | | | XXX | Ή | | | XXX | H | | |
| CHALLENGE BASELINE | ASELINE | ECG 1 | ddMMMyyyy:hh:mm | NO | ~ | XX | | | XXX | | | | XXX | | | |
| | | ECG 2 | ddMMMyyyy:hh:mm | ON | ~ | XXX | | | XXX | | | | XXX | | | |
| | | ECG 3 | ddMMMyyyy:hh:mm | NO | ~ | XX | | | XXX | | | | XXX | | | |
| | | MEAN | ddMMMyyyy:hh:mm | | ~ | XX | | | XXX | | | | XXX | | | |
| T | TIME POINT 3 | BCG 1 | ddMMMyyyy:hh:mm | NO | | XX | XXX | 130,60 | | | XXX | [30,60] | | × | XX | |
| | | ECG 2 | ddMMMyyyy:hh:mm | NO | NO | XX | XXX | [30,60] | )] XXX | | XXX | [30,60] | XXX | × | XXX | |
| | | ECG 3 | ddMMMyyyy:hh:mm | NO | NO | XXX | XXX | [30,60] | )] XXX | | XXX | [30,60] | XXX | × | XX | |
| | | MEAN | ddMMMyyyy:hh:mm | | NO | XXX | XXX | [30,60] | )] XXX | | XXX | [30,60] | XXX | × | XX | |

<sup>[1]</sup> NO = NOT USED IN ANALYSIS TABLES AND FIGURES.
[2] CLINICALLY SIGNIFICANT ABNORMALITY (CRF DATA).
[3] CHANGE FROM BASELINE VALUE.
[4] ABNORMALITY: H = ABNORMALLY HIGH VALUE / L = ABNORMALLY LOW VALUE COMPARED TO THE NORMAL RANGE.

| SAS DATE AND TIME | 1 10 8 10 11 | <br> | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|---|---|---|---|
| | MORPHOLOGY FOR SUBJECTS WITH ANY ABNORMAL INTERPRETATION | <br> | | COMMENT | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | FOR SUBJECTS WITH AN | | | FINDING | ×××××××××××××××××××××××××××××××××××××× |
| NO | LOGY | <br> | | CSA [2] | YES<br>NO<br>NO |
| ANALYSIS VERSION | | | ALE) | USE CSA [1] INTERPRETATION [2] FINDING | ABNORMAL<br>ABNORMAL<br>ABNORMAL |
| 01 - | RETAT | <br> | M) XX | USE [1] | N N O N |
| MMV_PFSPZ-DVI BLOOD STAGE_19_01 - ANALYSI | LISTING 16.2.10.2: ECG INTERPRETATION AND | . SAFETY | COHORT 1<br>SUBJECT NUMBER (SEX) = XXXXXXXX (MALE) | ECG<br>DATETIME<br> | ddMMyyyy;hh:mm NO<br>ddMMyyyy;hh:mm NO<br>ddMMyyyy;hh:mm NO |
| MMV_PFSPZ-DV | LISTING 16.2 | ANALYSIS SET: SAFETY | COHORT 1<br>SUBJECT NUMB | ANALYSIS<br>VISIT | SCREENING<br>BASELINE<br>TIMEPOINT 3<br>ETC |

[1] NO = NOT USED IN ANALYSIS TABLES AND FIGURES. [2] CLINICALLY SIGNIFICANT ABNORMALITY (CRF DATA).

Page 100 or

SAS DATE AND TIME PAGE X OF Y

## Malaria clinical score

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.11.1: MALARIA SIGNS AND SYMPTOMS

ANALYSIS SET: SAFETY

COHORT 1

HYP TAC FEV HEA MYA ART FAT MAL CHI SWE ANO NAU VOM ABD \* X X X X X X X X X X X X X X\* \* CHG MCS ACT USE [2] ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMMyyyy:hh:mm ddMMMyyyy; hh: mm ddMMMyyyy:hh:mm ASSESSMENT DATETIME DAY [1] 88 99 111 112 113 114 21 21 BASELINE ANALYSIS UNSCHED UNSCHED DAY 12 DAY 13 DAY 14 DAY 10 DAY 21 DAY 11 VISIT DAY S DAY FIRST ANTIMALARIAL ddMMMyyyy:hh:mm TREATMENT DATETIME SUBJECT NUMBER XXXX


<sup>[1]</sup> DAY VS. INOCULATION, DAYS ON WHICH ANTIMALARIAL TREATMENT IS TAKEN ARE FLAGGED (\*). [2] NO = NOT USED IN ANALYSIS TABLES AND FIGURES.

MCS=MALARIA CLINICAL SCORE (/42); ACT=ACTUAL VALUE; CHG=CHANGE FROM BASELINE.

MALARIA SIGNS AND SYMPTOMS: HEADACHE, MYALGIA, ARTHRALGIA, FATIGUE/LETHARGY, MALAISE, CHILLS/SHIVERING/RIGORS, SWEATING/HOT SPELLS, ANOREXIA, NAUSEA, VOMITING, ABDOMINAL DISCOMFORT, FEVER, TACHYCARDIA, HYPOTENSION.

SAS DATE AND TIME PAGE X OF Y


MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

LISTING 16.2.11.2: MALARIA CLINICAL SCORES > 6 AND PARASITAEMIA

ANALYSIS SET: SAFETY

COHORT 1

\$ \$ \$ \$ \$ \$ \$ RESULT (p/mL) [3] ddMMMyyyy:hh:mm PARASITAEMIA ASSESSMENT DATETIME BASELINE ANALYSIS DAY 11 DAY 12 DAY 13 DAY 14 VISIT XX.X XXXX XX.X XXXX XX.X XXXX XX.X XXXX NO XX.X XXXX [2] ACT CHG MCS USE --1 ddMMMyyyy;hh:mm 11 ddMMMyyyy;hh:mm 12 ddMMMyyyy;hh:mm 13 ddMMMyyyy;hh:mm 14 \* ddMMMyyyy;hh:mm 15 \* ddMMMyyyy;hh:mm ASSESSMENT DATETIME DAY [1] BASELINE DAY 11 DAY 12 DAY 13 DAY 14 UNSCHED ANALYSIS VISIT FIRST ANTIMALARIAL ddMMMyyyy:hh:mm TREATMENT DATETIME SUBJECT NUMBER XXXX

ETC...

[1] DAY VS. INOCULATION, DAYS ON WHICH ANTIMALARIAL TREATMENT IS TAKEN ARE FLAGGED (\*). [2] NO = NOT USED IN ANALYSIS TABLES AND FIGURES. [3] POSITIVE QPCR RESULTS (2 250 PARASITES PER ML BLOOD) ARE FLAGGED (\$). MCS=MALARIA CLINICAL SCORE (/42); ACT=ACTUAL VALUE; CHG=CHANGE FROM BASELINE.

# 5. TEMPLATE FIGURES

## 5.1 PHARMACODYNAMICS

Programmer note: all PD figures shown in this section will be repeated for the m-PD set with adjusted numbering (e.g. 14.2.3.1.2).


SAS DATE AND TIME PAGE X OF Y

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

ANALYSIS SET: PD



Mean (95% CI)


FIGURE 14.2.3.1.1: BLOOD-STAGE PARASITE PROFILE: MEDIAN PARASITAEMIA ACTUAL VALUES OVER TIME

## Programmer notes:

One line per cohort and for all subjects.

Legend: Cohort 1, Cohort 2, All subjects.

X-axis 'Analysis Time Point' will show scheduled time points from Day 7 to Riamet Day 4, 72h.

Y-axis label: 'log10(Parasitaemia)'.

No CI interval will be shown.

• Jittering should be allowed to distinguish overlapping symbols.


SAS DATE AND TIME PAGE X OF Y

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

FIGURE 14.2.3.2.1: BLOOD-STAGE PARASITE PROFILE: INDIVIDUAL PARASITAEMIA ACTUAL VALUES OVER TIME




## Programmer notes:

- A separate plot per cohort and all subjects starting in a new page.
- One line per subject.
- Legend: Subject numbers.
- X-axis label: 'Time from first PCR positivity (days)'.
- Y-axis label: 'log10(Parasitaemia)'.
- For each subject, show the assessments from the subject's first PCR positivity to parasite clearance.
- Different plotting symbols will be used on the first assessment when antimalarial treatment was given and will be denoted by a footnote.


SAS DATE AND TIME PAGE X OF Y

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

FIGURE 14.2.3.3.1: TIME TO FIRST PCR POSITIVITY: KAPLAN MEIER PLOT

ANALYSIS SET: PD



POSITIVE PARASITAEMIA IS DEFINED AS QPCR OUTCOME 2 250 PARASITES PER ML BLOOD.


## Programmer notes:

- One line per cohort and all subjects.
- X-axis label: 'Time from PfSPZ inoculation (days)'.
  - Y-axis label: 'Probability (%)'.


# Programmer note: repeat Figure 14.2.3.3.1 for:

FIGURE 14.2.3.4.1: TIME TO PARASITAEMIA OF 25000 PARASITES PER ML BLOOD: KAPLAN MEIER PLOT FIGURE 14.2.3.5.1: TIME TO FIRST DOSE OF TREATMENT WITH RIAMET: KAPLAN MEIER PLOT FIGURE 14.2.3.6.1: TIME TO PARASITE CLEARANCE: KAPLAN MEIER PLOT

The footnotes and axes will be adapted accordingly.


## 5.2 SAFETY

# 7.2.1 Clinical laboratory evaluation

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

SAS DATE AND TIME PAGE X OF Y

FIGURE 14.3.2.1: INDIVIDUAL LABORATORY TEST ACTUAL VALUES OVER TIME

ANALYSIS SET: SAFETY




## Programmer notes:

- A separate plot per cohort and all subjects starting in a new page.
- One line per subject and one line for the median.
- X-axis 'Analysis Time Point' will show scheduled time points.
- Label Y-axis will be the laboratory test result.
- The following laboratory parameters will be shown in separate plots: liver biochemistry parameters (albumin, AST, ALT, ALP, GGT, total and direct bilirubin and total serum proteins), CRP and haemoglobin.


## 5.2.2 Vital signs

The analysis figures for vital signs parameters are largely identical to the laboratory figures.

FIGURE 14.3.3.1: INDIVIDUAL VITAL SIGNS ACTUAL VALUES OVER TIME

## Programmer notes:

- The following vital signs parameters will be shown in separate plots: heart rate and body temperature.
- The median time to first antimalarial treatment administration will be shown with a reference line.


## 5.2.3 ECG

The analysis figures for ECG parameters are largely identical to the laboratory figures.

FIGURE 14.3.4.1: INDIVIDUAL ECG ACTUAL VALUES OVER TIME

Programmer note: the following ECG parameters will be shown in separate plots: QTcF and QTcB.


SAS DATE AND TIME PAGE X OF Y

MMV\_PfSPZ-DVI Blood Stage\_19\_01

## Malaria clinical score

MMV\_PFSPZ-DVI BLOOD STAGE\_19\_01 - ANALYSIS VERSION

FIGURE 14.3.5.1: INDIVIDUAL MALARIA CLINICAL SCORE ACTUAL VALUES OVER TIME

ANALYSIS SET: SAFETY




## Programmer notes:

- A separate plot per cohort and all subjects starting in a new page.
- One line per subject and one line for the median.
- X-axis 'Analysis Time Point' will show scheduled time points.
- Label Y-axis will be 'Malaria clinical score'.
- Different symbols will be used for the time points where antimalarial treatment was taken for the first time and for the time point of peak parasitaemia. They will be specified in a footnote.
- The median time to first antimalarial treatment administration will be shown with a reference line.

# Programmer note: repeat Figure 14.3.5.1 for:

FIGURE 14.3.5.2: INDIVIDUAL MALARIA CLINICAL SCORE AND PARASITAEMIA ACTUAL VALUES OVER TIME

FIGURE 14.3.5.3: INDIVIDUAL MALARIA CLINICAL SCORE AND CRP ACTUAL VALUES OVER TIME

- Each figure will show a separate plot per cohort starting in a new page followed by a separate plot per individual subject starting in a new page.
- One line per subject and parameter. I.e. individual subjects plots will have 2 lines; cohort plots will have 2\*8 = 16 lines (if no missing
- X-axis 'Time from PfSPZ inoculation (days)' will show the relative time in days of the individual subject assessments.
- Label Y-axis will be 'Malaria clinical score' on the left Y-axis and 'log10(Parasitaemia)' / 'CRP (unit)' on the right Y-axis.
- The first antimalarial treatment administration will be shown with a reference line.




### **Certificate Of Completion**

Envelope Id: 7A8080D29B54469F91469E9C4688E6A0 Status: Completed Subject: Please DocuSign: MMV\_PfSPZ-DVI Blood Stage\_19\_01\_SAP\_v1.0.docx, MMV\_PfSPZ-DVI Blood Stage\_19\_01...

Source Envelope:

Document Pages: 167

Certificate Pages: 6

AutoNav: Enabled

Envelope Originator:

Daniel Izquierdo Juncas

Generaal de wittelaan 19a

Envelopeld Stamping: Disabled

MECHELEN, Antwerp 2800

Time Zone: (UTC+01:00) Brussels, Copenhagen, Madrid, Paris daniel.izquierdojuncas@sgs.com

IP Address: 165.225.93.35

Viewed: 2/11/2021 4:21:30 PM

Signed: 2/11/2021 4:23:23 PM

Sent: 2/11/2021 4:09:51 PM

Viewed: 2/11/2021 4:10:01 PM

Signed: 2/11/2021 4:11:35 PM

### **Record Tracking**

Status: Original Holder: Daniel Izquierdo Juncas Location: DocuSign

2/11/2021 4:03:36 PM daniel.izquierdojuncas@sgs.com

## Signer EventsSignatureTimestampbastiaan JansenSent: 2/11/2021 4:09:51 PM

bastiaan.jansen@sgs.com

Biostatistical Coordinator - Senior Statistician

GS BE

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

15ADFC6D-3E73-4686-B167-F978EA41202B

Using IP Address: 81.243.99.25

bastiaan Jansen

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document I approve this document

### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

Daniel Izquierdo Juncas daniel.izquierdojuncas@sgs.com

Biostatistician SGS LS

Security Level: Email. Account Authentication

(Required)

Daniel Izquierdo Juncas

Signature Adoption: Pre-selected Style

Signature ID:

690E6583-03D5-4613-A9EC-59ED7BAE2148

Using IP Address: 165.225.93.35

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):
I am the author of this document
I am the author of this document

## Electronic Record and Signature Disclosure:

Not Offered via DocuSign

**Signer Events** 

Farouk Chughlay chughlayf@mmv.org

Project and Medical Director

Farouk Chughlay

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Drawn on Device

Signature ID:

**Signature** 

6A2C1E23-2AEB-48DF-A6A5-44CF570BF27F

Using IP Address: 83.228.139.243

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 2/5/2021 11:52:45 AM

ID: cbc1c9da-6caf-461d-9c71-c22138d857b0

Myriam El Gaaloul elgaaloulm@mmv.org

Security Level: Email, Account Authentication

(Required)

Myriam El Gaaloul

Sent: 2/11/2021 4:23:28 PM Viewed: 2/13/2021 10:14:26 AM Signed: 2/13/2021 10:25:38 AM

**Timestamp** 

Sent: 2/11/2021 4:23:28 PM

Viewed: 2/11/2021 4:54:18 PM

Signed: 2/11/2021 4:55:13 PM

Signature Adoption: Pre-selected Style

Signature ID:

C2CA71F3-3AA8-43DA-B327-CC3B36DFB37C

Using IP Address: 213.55.244.6

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document I approve this document

COPIED

**Electronic Record and Signature Disclosure:** 

Accepted: 2/13/2021 10:14:26 AM

ID: 672a0588-36b7-450e-bb09-e42c22631e93

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------------------------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Ann Mallinus | COPTER | Sent: 2/13/2021 10:25:43 AM |

ann.mallinus@sgs.com

Management Assistant Biostatistics

SGS Belgium NV

Security Level: Email, Account Authentication

(Required)

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign

**Witness Events Signature Timestamp Notary Events Signature Timestamp** 

| Envelope Summary Events | Status | Timestamps |
|---------------------------------|------------------|-----------------------|
| Envelope Sent | Hashed/Encrypted | 2/11/2021 4:09:52 PM |
| Certified Delivered | Security Checked | 2/13/2021 10:14:26 AM |
| Signing Complete | Security Checked | 2/13/2021 10:25:38 AM |
| Completed | Security Checked | 2/13/2021 10:25:43 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature | Disclosure | |

## ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, SGS LS (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

## Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

## Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

## Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### How to contact SGS LS:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

## To advise SGS LS of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

## To request paper copies from SGS LS

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to Barbara.Buls@sgs.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

## To withdraw your consent with SGS LS

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to Arnaud.Luisier@sgs.com and in the body of such request you must state your email, full name, mailing address, and telephone number. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

## Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

## Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify SGS LS as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by SGS LS during the course of your relationship with SGS LS.